| Division | : | Worldwide Development |
|------------------|---|-----------------------------|
| Information Type | | Reporting and Analysis Plan |

| Title | : | Reporting and Analysis Plan for 450 Participant/6 Month<br>Strategic Interim and Final Analysis for Study 205724:<br>Randomized, Double-Blind (Sponsor Open), Placebo-<br>Controlled, Multi-centre, Dose Ranging Study to Evaluate<br>the Efficacy and Safety of Danirixin Tablets Administered<br>Twice Daily Compared with Placebo for 24 Weeks in Adult<br>Participants with Chronic Obstructive Pulmonary Disease |
|---|---|---|
| <b>Compound Number</b> | : | GSK1325756 |
| <b>Effective Date</b> | : | 30-OCT-2018 |

## **Description:**

• The purpose of this Reporting and Analysis Plan is to describe the planned 450 participant/6 month strategic interim and final analyses and output to be included in the Clinical Study Report for Protocol 205724.

## RAP Author(s):

| Approver | Date | Approval Method |
|----------------------------------------|-------------|-----------------|
| Statistics Leader, Clinical Statistics | 25-OCT-2018 | eTMF eSignature |
| Director Clinical Pharmacology | 29-OCT-2018 | eTMF eSignature |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|-------------------------------|-------------|-----------------|
| Programming Manager | 26-OCT-2018 | eTMF eSignature |
| Senior Scientific Director | 30-OCT-2018 | email |
| Clinical Development Manager | 26-OCT-2018 | eTMF eSignature |
| PPD Clinical Data Management | 26-OCT-2018 | eTMF eSignature |
| PPD Patient Reported Outcomes | 26-OCT-2018 | email |
| Global Regulatory Affairs | 25-OCT-2018 | eTMF eSignature |
| PPD Statistics Director | 26-OCT-2018 | eTMF eSignature |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Statistics Director (Respiratory Clinical Statistics) | 30-OCT-2018 | eTMF eSignature |
| Programming Manager (Respiratory Clinical Programming) | 26-OCT-2018 | eTMF eSignature |

## **TABLE OF CONTENTS**

| | | | PAGE |
|----|------|-----------------------------------------------------------|------|
| 1. | INTR | ODUCTION | 7 |
| • | 1.1. | RAP Amendment | |
| 2. | | MARY OF KEY PROTOCOL INFORMATION | |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objectives and Endpoints | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | 13 |
| 3. | PLAN | INED ANALYSES | 14 |
| | 3.1. | Interim Analyses | 14 |
| | | 3.1.1. Interim PK Analysis | |
| | | 3.1.2. Futility Analysis | |
| | | 3.1.3. Strategic Analysis | |
| | | 3.1.4. Administrative Interims | 14 |
| | 3.2. | Final Analyses | |
| 4. | ΔΝΔΙ | YSIS POPULATIONS | 16 |
| •• | 4.1. | Strategic Interim Analysis | |
| | 4.2. | Final Analysis | |
| | 4.3. | Protocol Deviations | |
| 5. | CONI | CIDEDATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| Э. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING VENTIONS | 18 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | 18 |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | | 5.4.1. Covariates and Other Strata | 19 |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | |
| | | Conventions | 20 |
| 6. | STUE | DY POPULATION ANALYSES | 21 |
| 0. | 6.1. | Overview of Planned Study Population Analyses | |
| | 0.1. | 6.1.1. Demographic and Baseline Characteristics | |
| | | 6.1.2. Prior and Concomitant Medications | 21 |
| | | 6.1.3. Exposure and Treatment Compliance | |
| 7. | EEE! | CACY ANALYSES | 22 |
| Ι. | 7.1. | Primary Efficacy Analyses | |
| | 1.1. | 7.1.1. Month 6 E-RS: COPD Total Score Dose-Response | |
| | | Analysis | |
| | | 7.1.1.1. Endpoint | |
| | | 7.1.1.2. Summary Measure | |
| | | 7.1.1.3. Population of Interest | |

| | | 7.1.1.4. | Strategy for Intercurrent (Post-Randomization) Events | 23 |
|---|---|---|---|---|
| | | 7.1.1.5. | Statistical Analyses / Methods | |
| | | | 7.1.1.5.1. Statistical Methodology | |
| | | | Specification | 23 |
| | 7.1.2. | F-RS: CO | OPD Subscale Scores Dose-Response Analysis | |
| | 7.1.2. | | OPD Total and Subscale Scores Longitudinal | 20 |
| | 7.1.5. | | | 25 |
| | | 7.1.3.1. | · | |
| | | 7.1.3.2. | • | |
| | | 7.1.3.3. | | 25 |
| | | 7.1.3.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.3.5. | | 26 |
| | | | 7.1.3.5.1. Bayesian MMRM Methodology | |
| | | | Specification | 26 |
| | | | 7.1.3.5.2. Frequentist MMRM Methodology | |
| | | | Specification | 2 <mark>7</mark> |
| 7.2. | Second | lary Efficacy | y Analyses | 28 |
| | 7.2.1. | | Rate of HCRU Exacerbations and Annual Rate of | |
| | | | Events | 29 |
| | | 7.2.1.1. | | |
| | | 7.2.1.2. | | |
| | | 7.2.1.3. | • | |
| | | 7.2.1.4. | | 20 |
| | | 7.2.1.7. | Events | 29 |
| | | 7.2.1.5. | Statistical Analyses / Methods | |
| | | | 7.2.1.5.1. Statistical Methodology | |
| | | | Specification | 29 |
| | 7.2.2. | Time to F | First HCRU Exacerbation and EXACT Event | |
| | | 7.2.2.1. | Endpoint | |
| | | 7.2.2.2. | Summary Measure | |
| | | 7.2.2.3. | • | |
| | | 7.2.2.3. | • | |
| | | 1.2.2.7. | Events | |
| | | 7.2.2.5. | Statistical Analyses / Methods | |
| | | 1.2.2.5. | | 32 |
| | | | 7.2.2.5.1. Statistical Methodology | 22 |
| | 700 | E DC: 00 | Specification | 32 |
| | 7.2.3. | | OPD Total and Subscale Scores Responder | 22 |
| | | | Foods sint | 33 |
| | | 7.2.3.1. | Endpoint | |
| | | 7.2.3.2. | Summary Measure | |
| | | 7.2.3.3. | Population of Interest | 33 |
| | | 7.2.3.4. | Strategy for Intercurrent (Post-Randomization) Events | 33 |
| | | 7.2.3.5. | Statistical Analyses / Methods | |
| | | 1.2.3.3. | | 33 |
| | | | 7.2.3.5.1. Statistical Methodology | 20 |
| | 704 | CODO T | Specification | |
| | 7.2.4. | | otal Score and CAT Score | |
| | 7.2.5. | | Jse | |
| <b>-</b> - | 7.2.6. | | Activity | |
| 7.3. | Explora | itory efficac | cy Analyses | 35 |

#### CONFIDENTIAL

| 7.3.3. Time to First Clinically Important Deterioration | | | 7.3.1. | E-RS: COPD Total Score | |
|---|---|---|---|---|---|
| 7.3.4. SGRQ Domain Scores 36 7.3.5. Participant Global Assessments 36 3. SAFETY ANALYSES 37 8.1. Adverse Events Analyses 37 8.2. Adverse Events of Special Interest Analyses 37 8.3. Clinical Laboratory Analyses 37 8.4. Spirometry 37 8.4. Spirometry 37 8.4.1. Endpoint 37 8.4.2. Summary Measure 37 8.4.3. Population of Intereurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses Methods 38 8.5. Other Safety Analyses 39 9.1. Primary Pharmacokinetic Analyses 39 9.1. Primary Pharmacokinetic Analyses 39 9.1. Derived Pharmacokinetic Parameters 39 9.1. Derived Pharmacokinetic Parameters 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 | | | 7.3.2. | | |
| 7.3.5. Participant Global Assessments 36 3. SAFETY ANALYSES 37 8.1. Adverse Events of Special Interest Analyses 37 8.2. Adverse Events of Special Interest Analyses 37 8.4. Spirometry 37 8.4. Spirometry 37 8.4.1. Endpoint 37 8.4.2. Summary Measure 37 8.4.3. Population of Interest 37 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9.1. Primary Pharmacokinetic Manalyses 39 9.1. Primary Pharmacokinetic Canalyses 39 9.1. Primary Pharmacokinetic Analyses 39 9.1. Primary Pharmacokinetic Analyses 40 9.2. Exploratory Pharmacokinetic Analyses 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 39 9.2. Statistical Methodology Specification 40 | | | | | |
| 8. SAFETY ANALYSES 37 8.1. Adverse Events Analyses 37 8.2. Adverse Events of Special Interest Analyses 37 8.3. Clinical Laboratory Analyses 37 8.4. Spirometry 37 8.4.1. Endpoint 37 8.4.2. Summary Measure 37 8.4.3. Population of Intercert 37 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9.1. Primary Pharmacokinetic Analyses 39 9.1. Primary Pharmacokinetic Parameters 39 9.1. Statistical Analyses / Methods 39 9.2. Exploratory Pharmacokinetic Parameters 39 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACOMYNAMIC ANALYSES 42 14. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population | | | | | |
| 8.1. Adverse Events of Special Interest Analyses 37 8.2. Adverse Events of Special Interest Analyses 37 8.3. Clinical Laboratory Analyses 37 8.4. Spirometry 37 8.4.1. Endpoint 37 8.4.2. Summary Measure 37 8.4.3. Population of Intercurrent (Post-Randomization) Events 38 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9. PHARMACOKINETIC ANALYSES 39 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Perived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Analyses / Methods 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACOMYNAMIC ANALYSES 42 13. REFERENCES 43 14. Appendix 1: Protocol Deviation Management and Definitions for P | | | 7.3.5. | Participant Giobai Assessments | 30 |
| 8.2. Adverse Events of Special Interest Analyses 37 8.3. Clinical Laboratory Analyses 37 8.4. Spirometry 37 8.4.1. Endpoint 37 8.4.2. Summary Measure 37 8.4.3. Population of Interest 37 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9.1. Primary Pharmacokinetic Analyses 39 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.2. Exploratory Pharmacokinetic Analyses 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1.1. Exclusions from | 8. | | | | |
| 8.3. Clinical Laboratory Analyses 37 8.4. Spirometry 37 8.4.1. Endpoint 37 8.4.2. Summary Measure 37 8.4.3. Population of Interest 37 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9. PHARMACOKINETIC ANALYSES 39 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methodos 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 | | _ | | | |
| 8.4. Spirometry 37 8.4.1. Endpoint 37 8.4.2. Summary Measure 37 8.4.3. Population of Interest 37 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.4.5. Other Safety Analyses 39 9. PHARMACOKINETIC ANALYSES 39 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2. Exploratory Pharmacokinetic Parameters 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12. Statistical Analyses / Methods 42 < | | _ | | | |
| 8.4.1. Endpoint 37 8.4.2. Summary Measure 37 8.4.3. Population of Interest 37 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14. 1. Appendix 1: Protocol Deviation Management and Defini | | | | | |
| 8.4.2. Summary Measure 37 8.4.3. Population of Interest 37 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9. PHARMACOKINETIC ANALYSES 39 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 43 14. APPENDICES 44 14. 2. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14. 2. Appendix 2: Schedule of Activities 45 14. 2. Appendix 3: Assessment Windows 5 | | 8.4. | | | |
| 8.4.3. Population of Interest. 37 8.4.4. Strategy for Intercurrent (Post-Randomization) Events. 38 8.4.5. Statistical Analyses / Methods. 38 8.5. Other Safety Analyses. 39 9. PHARMACOKINETIC ANALYSES. 39 9.1. Primary Pharmacokinetic Analyses. 39 9.1.1. Derived Pharmacokinetic Parameters. 39 9.1.2. Statistical Analyses / Methods. 39 9.2.1. Derived Pharmacokinetic Parameters. 40 9.2.1. Derived Pharmacokinetic Parameters. 40 9.2.2. Statistical Analyses / Methods. 40 9.2.2.1. Statistical Methodology Specification. 40 10. POPULATION PHARMACOKINETIC ANALYSES. 41 11. BIOMARKER ANALYSES. 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES. 42 13. REFERENCES. 43 14. APPENDICES. 43 14. APPENDICES. 44 14.1. Exclusions from Per Protocol Population. 44 14.2. Appendix 2: Schedule of Activi | | | | | |
| 8.4.4. Strategy for Intercurrent (Post-Randomization) Events 38 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9. PHARMACOKINETIC ANALYSES 39 9.1. Primary Pharmacokinetic Analyses 39 9.1. Derived Pharmacokinetic Parameters 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2. Exploratory Pharmacokinetic Parameters 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Exclusions from Per Protocol Population 44 14.2. Appendix 1: Protocol Defined Schedule of Events 45 14.2. Appendi | | | | | |
| 8.4.5. Statistical Analyses / Methods 38 8.5. Other Safety Analyses 39 9. PHARMACOKINETIC ANALYSES 39 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2. Exploratory Pharmacokinetic Parameters 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Analyses / Methods 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 13. REFERENCES 43 14. APPENDICES 44 14. APPENDICES 44 14. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.2.1 Protocol Defined S | | | | | |
| 8.4.5.1. Frequentist MMRM Methodology Specification | | | - | Statistical Analyses / Methods | 38 |
| 8.5. Other Safety Analyses 39 9. PHARMACOKINETIC ANALYSES 39 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2. Exploratory Pharmacokinetic Analyses 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.2. Appendix 2: Schedule of Activities 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases | | | 0.4.0. | | |
| 9. PHARMACOKINETIC ANALYSES | | 8.5. | Other Sa | | |
| 9.1. Primary Pharmacokinetic Analyses 39 9.1.1. Derived Pharmacokinetic Parameters 39 9.2. Exploratory Pharmacokinetic Analyses 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.2. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 | | | | • | |
| 9.1.1. Derived Pharmacokinetic Parameters 39 9.1.2. Statistical Analyses / Methods 39 9.2. Exploratory Pharmacokinetic Analyses 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1. Appendix 2: Schedule of Activities 44 14.2. Appendix 2: Schedule of Activities 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases 52 14.4.1. Study Phases for Diary Data 52 14.4.1. Study Phases for Event Data 53 <t< td=""><td>9.</td><td></td><td></td><td></td><td></td></t<> | 9. | | | | |
| 9.1.2. Statistical Analyses / Methods 39 9.2. Exploratory Pharmacokinetic Analyses 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases 52 14.4.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | 9.1. | | | |
| 9.2. Exploratory Pharmacokinetic Analyses 40 9.2.1. Derived Pharmacokinetic Parameters 40 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Event Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | | - | | |
| 9.2.1. Derived Pharmacokinetic Parameters | | 0.2 | | | |
| 9.2.2. Statistical Analyses / Methods 40 9.2.2.1. Statistical Methodology Specification 40 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.2.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | 9.2. | | | |
| 9.2.2.1. Statistical Methodology Specification | | | | | |
| 10. POPULATION PHARMACOKINETIC ANALYSES 41 11. BIOMARKER ANALYSES 42 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.4.1.4. Study Phases for Other Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | | 9.2.2. | | |
| 11. BIOMARKER ANALYSES 41 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1.1 Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.2.1 Protocol Defined Schedule of Events 45 14.3 Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1.1 Study Phases for Diary Data 52 14.4.1.2 Study Phases for Concomitant Medication 52 14.4.1.3 Study Phases for Event Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1 Reporting Process 54 | | | | • • | |
| 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES 42 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.2.1. Protocol Defined Schedule of Events 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | 10. | POPU | LATION F | PHARMACOKINETIC ANALYSES | 41 |
| 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.2.1. Protocol Defined Schedule of Events 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases for Diary Data 52 14.4.1.1. Study Phases for Concomitant Medication 52 14.4.1.2. Study Phases for Event Data 53 14.4.1.4. Study Phases for Other Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | 11. | BIOMA | ARKER AI | NALYSES | 41 |
| 12.1. Statistical Analyses / Methods 42 13. REFERENCES 43 14. APPENDICES 44 14.1.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.2.1. Protocol Defined Schedule of Events 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases for Diary Data 52 14.4.1.1. Study Phases for Concomitant Medication 52 14.4.1.2. Study Phases for Event Data 53 14.4.1.4. Study Phases for Other Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | | | | |
| 13. REFERENCES 43 14. APPENDICES 44 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population 44 14.1.1. Exclusions from Per Protocol Population 44 14.2. Appendix 2: Schedule of Activities 45 14.2.1. Protocol Defined Schedule of Events 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.4.1.4. Study Phases for Other Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | 12. | | | | |
| 14. APPENDICES | | 12.1. | Statistica | al Analyses / Methods | 42 |
| 14. APPENDICES | 13 | RFFFI | RENCES | | 43 |
| 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population | | | KENTOLO. | | |
| Protocol Population | 14. | | | | |
| 14.1.1. Exclusions from Per Protocol Population4414.2. Appendix 2: Schedule of Activities4514.2.1. Protocol Defined Schedule of Events4514.3. Appendix 3: Assessment Windows5114.4. Appendix 4: Study Phases5214.4.1. Study Phases5214.4.1.1. Study Phases for Diary Data5214.4.1.2. Study Phases for Concomitant Medication5214.4.1.3. Study Phases for Event Data5314.4.1.4. Study Phases for Other Data5314.5. Appendix 5: Data Display Standards & Handling Conventions5414.5.1. Reporting Process54 | | 14.1. | | | |
| 14.2. Appendix 2: Schedule of Activities 45 14.2.1. Protocol Defined Schedule of Events 45 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.4.1.4. Study Phases for Other Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | | Protocol | Population | 44 |
| 14.2.1.Protocol Defined Schedule of Events4514.3.Appendix 3: Assessment Windows5114.4.Appendix 4: Study Phases5214.4.1.Study Phases for Diary Data5214.4.1.1.Study Phases for Concomitant Medication5214.4.1.3.Study Phases for Event Data5314.4.1.4.Study Phases for Other Data5314.5.Appendix 5: Data Display Standards & Handling Conventions5414.5.1.Reporting Process54 | | | 14.1.1. | Exclusions from Per Protocol Population | 44 |
| 14.3. Appendix 3: Assessment Windows 51 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases for Diary Data 52 14.4.1.1. Study Phases for Concomitant Medication 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.4.1.4. Study Phases for Other Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | 14.2. | | | |
| 14.4. Appendix 4: Study Phases 52 14.4.1. Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.4.1.4. Study Phases for Other Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | 440 | | | |
| 14.4.1. Study Phases 52 14.4.1.1. Study Phases for Diary Data 52 14.4.1.2. Study Phases for Concomitant Medication 52 14.4.1.3. Study Phases for Event Data 53 14.4.1.4. Study Phases for Other Data 53 14.5. Appendix 5: Data Display Standards & Handling Conventions 54 14.5.1. Reporting Process 54 | | | | | |
| 14.4.1.1. Study Phases for Diary Data | | 14.4. | | | |
| 14.4.1.2. Study Phases for Concomitant Medication | | | 14.4.1. | | |
| 14.4.1.3. Study Phases for Event Data | | | | 14.4.1.2 Study Phases for Concomitant Medication | 52<br>52 |
| 14.4.1.4. Study Phases for Other Data | | | | | |
| 14.5. Appendix 5: Data Display Standards & Handling Conventions | | | | | |
| 14.5.1. Reporting Process54 | | 14.5. | Appendix | | |
| · | | - | 14.5.1. | Reporting Process | 54 |
| | | | 14.5.2. | . • | |

#### CONFIDENTIAL

| വ | 05 | 724 |
|---|-----|-----|
| | UU. | 124 |

| | 14.5.3. | Reporting | Standards for Pharmacokinetic Data | ! | 56 |
|---|---|---|---|---|---|
| 14.6. | Appendix | | I and Transformed Data | | |
| | 14.6.1. | General | | ! | 57 |
| | 14.6.2. | Study Pop | ulation | ! | 57 |
| | 14.6.3. | Efficacy | | ( | 61 |
| | 14.6.4. | | | | |
| 14.7. | Appendix | 7: Reporti | ng Standards for Missing Data | | 68 |
| | 14.7.1. | | Withdrawals | | |
| | 14.7.2. | | of Missing Data | | |
| | | | Handling of Missing and Partial Dates | | |
| 14.8. | | | of Potential Clinical Importance | | |
| | 14.8.1. | , | Values | | |
| | 14.8.2. | | | | |
| | 14.8.3. | | | | |
| 14.9. | | | ion Pharmacokinetic Analyses | | |
| | 14.9.1. | | Pharmacokinetic Dataset Specification | | 72 |
| | | 14.9.1.1. | Handling Missing Demographic and Covariate | | |
| | | | Data | | |
| | | 14.9.1.2. | Handling Missing Dose Times | | |
| | | | Handling Missing Times of PK Samples | | 72 |
| | | 14.9.1.4. | Handling of PK Data Below the Lower Limit of | | |
| | | 44045 | Quantification | | |
| 4440 | A | 14.9.1.5. | Dataset Specification | | |
| 14.10. | | | viations & Trade Marks | | |
| | | | ons | | |
| 1111 | | | (S | | |
| 14.11. | | | Data Displays | | |
| | | | ay Numbering | | |
| | | | esulation Tables | | |
| | | | ulation Figuresulation Figures | | |
| | | | ables | | |
| | | | gures | | |
| | | | ples | | |
| | | | ures | | |
| | 1 <del>4</del> .11.0. | Dharmaco | kinetic Tables | I | 14 |
| | | | kinetic Fableskinetic Figures | | |
| | 14.11.10 | Dharmaco | kinetic / Pharmacodynamic Figure | <u> </u> | 10 |
| | | | Tables | | |
| | | | Figures | | |
| | | | istings | | |
| 14 12 | | | ble Mock Shells for Data Displays | | |
| 17.14. | Whheling | \ ι∠. ∟λαιιι | ole intock offelið for þata þisplays | 15 | JU |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the 450 participant/6 month strategic interim. This RAP will also describe the final analyses to be included in the Clinical Study Report (CSR) for Protocol 205724.

| Revision Chronology | : | |
|---|---|---|
| 2016N293867_00 | 28-NOV-2016 | Original |
| 2016N293867_01 | 31-OCT-2017 | <ul> <li>Adds a second, optional, detailed pharmacokinetic profiling at Visit 10 in a subset of participants to allow for a better understanding of danirixin pharmacokinetics.</li> <li>Removes the Participant Exit Interview from the exploratory endpoints.</li> <li>Provides additional information and clarification for the following: spirometry assessments, exclusion for cancers other than lung cancer, permitted use of supplemental oxygen, permitted uses of chronic steroids, participant numbering requirement for rescreening, additional text to explain the timing of the planned interim analysis and updates to the analysis populations.</li> </ul> |

# 1.1. RAP Amendment

Revision chronology:

| RAP Section | Amendment Details |
|---|---|
| GSK1325756-205724 Statis 2018) | GSK1325756-205724 Statistical Analysis Plan Reporting and Analysis Plan Version 001 (31-Aug-2018) |
| GSK1325756-205724 Repor | ing and Analysis Plan Amendment1_Final [Insert Date] |
| Approvals | Removed PPD as she has left GSK. Added PPD replacement) as an additional approver |
| 2.2 Study Objectives and Endpoints | PK endpoints were not assessed in the strategic interim |
| 3.1.3 Strategic Analysis | Updated to past tense |
| 3.2 Final Analysis | Updated to reflect planned unblinding process |
| 4.1 Strategic Interim Analysis, 7.1.4.5.1 Bayesian MMRM Methodology Specification and 7.2.1.5.1 Statistical Methodology Specification | <ul> <li>ITT and Symptomatic populations not used for final analysis.</li> <li>(PP) added to Per Protocol population in the definition table.</li> </ul> |
| 6.1.2 Prior and Concomitant Medications | Additional concomitant medication table at Month 6 |
| 7.1.1 Month 6 E-RS: COPD<br>Total Score Dose-<br>Response Analysis | Clarification of posterior predictive probability of success calculation used at the Strategic Interim |

| RAP Section | Amendment Details |
|---|---|
| 7.1.2 Month 2-6 E-RS:<br>COPD Total Score Dose-<br>Response Analysis and<br>7.1.3.5.2 Frequentist<br>ANCOVA Methodology<br>Specification and 14.6.3<br>Efficacy | Month 2-6 E:RS: COPD Dose Response Analysis not required |
| 7.1.4.5.1 Bayesian MMRM Methodology Specification | Updates to Bayesian model specifications to improve convergence and mixing |
| 7.1.4.5.3 Frequentist<br>MMRM Methodology<br>Specification | Additional plots of LS Mean and daily mean E-RS: COPD scores. Plots of empirical distribution function for E-RS: COPD Total Scores. |
| 7.2.1.5.1 Statistical<br>Methodology Specification | Additional table for HCRU exacerbations treated with antibiotics. |
| 7.2.4 SGRQ Total Score and CAT Score | Additional plot of arithmetic mean and 90% CIs for SGRQ and CAT |
| 7.2.5 Rescue Medication | Additional plots daily rescue medication use |
| 7.3.1 E-RS: COPD Total<br>Score | Identify subgroups not required for final SAC |
| 7.3.3 Time to First<br>Clinically Important<br>Deterioration | • |
| 8.3 Clinical Laboratory<br>Analysis | Remove urinalysis outputs because no PCI ranges are defined for urinalysis |
| 8.4.5.1 Frequentist MMRM Methodology Specification | Additional summaries of FEV1/FVC ratio and plots of arithmetic mean and 90% CIs for all spirometry endpoints. |
| 11 Biomarker Analysis | Additional tables and boxplots in subjects with pneumonia |
| 14.4.1.1 Study Phases for Diary Data | Clarify that Diary data phases applies to EXACT events |
| 14.6.2 Study Population | Additional COPD medication combinations table at Month 6 |
| 14.6.3 Efficacy | Clarify definitions for Season, time to first, raw annual rate and offset. Remove definition of CID as not reporting this exploratory endpoint. |
| 14.6.4 Safety | Clarify definition for character laboratory parameters. Add definition of ICS use for pneumonia table. |
| 14.11 Appendix 11: List of Data Displays | <ul> <li>Updates to tables and figures.</li> <li>Remove urinalysis outputs</li> <li>Remove CID tables</li> </ul> |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| All Participants population | All Subjects population | R&D Clinical Data Standards Board<br>(CDSB) recommendation to use the<br>term 'Subjects' in all displays (Tables,<br>Figures & Listings) |
| No Intent-to-treat (ITT) population | ITT population defined<br>to be used for selected<br>efficacy displays | Used for key efficacy displays to<br>enable phase III planning |
| No Per Protocol (PP) population | PP population defined<br>and used for efficacy<br>displays | Remove data from participants who had a protocol deviation considered to impact efficacy during the treatment period. |
| No Symptomatic population | Symptomatic<br>population defined and<br>used for selected study<br>population and efficacy<br>displays | Used to explore the subgroup of symptomatic participants. |
| No PK2 population | PK2 population defined<br>and used for PK dry<br>blood spot vs wet<br>whole blood | Used to compare dry blood spot with wet whole blood |
| mITT population used for efficacy endpoints | PP population used for efficacy endpoints | Remove data from participants who had a protocol deviation considered to impact efficacy during the treatment period. |
| The final Emax model will<br>be repeated using months<br>1-6 and months 3-6. | The final Emax model will be repeated using months 2-6. | Team decision to include most informative time period. |
| The protocol states that exacerbation rates for the danirixin and placebo groups, along with the ratio in exacerbation rates danirixin/placebo, will be estimated and corresponding 95% credible intervals will be produced. | 90% credible intervals<br>will be produced for all<br>Bayesian efficacy<br>analyses including<br>exacerbation rates. | Inconsistency in protocol. |

# 2.2. Study Objectives and Endpoints

| Ob | jectives | End | dpoints | Assessed in<br>Strategic<br>Interim |
|---|---|---|---|---|
| Pri | mary Objectives | Pri | mary Endpoints | |
| • | To characterize the dose response of danirixin compared with placebo on the incidence and severity of respiratory symptoms in participants with chronic obstructive pulmonary disease (COPD) | • | Change from baseline in respiratory symptoms measured by the Evaluating Respiratory Symptoms in COPD (E-RS: COPD) daily diary: total score and subscales (i.e. breathlessness, cough and sputum, and chest symptoms) | Yes |
| • | To compare the safety of danirixin with placebo in participants with COPD | • | Adverse events (AE), clinical laboratory values, vital signs, electrocardiogram (ECG) | Yes <sup>[1]</sup> |
| Ser | condary Objectives | Sec | condary Endpoints | |
| • | To characterize the dose response of danirixin compared with placebo on the annual rate of moderate/severe COPD exacerbations in participants with COPD | • | Healthcare Resource Utilization (HCRU)-defined COPD exacerbations | Yes |
| • | To further characterize the clinical activity of | • | E-RS: COPD Responder Analysis (including subscales) | Yes |
| | danirixin compared to placebo in participants with COPD | • | Number of Exacerbations of Chronic<br>Pulmonary Disease (EXACT) tool<br>defined events | No |
| | | • | Time to first EXACT event | No |
| | | • | EXACT event severity | No |
| | | • | EXACT event duration for all events Time to first HCRU-defined COPD exacerbation | No<br>Yes |
| | | • | Time to first severe HCRU-defined COPD exacerbation | Yes |
| | | • | HCRU-defined COPD exacerbation duration | Yes |
| | | • | Change from baseline for the St.<br>George's Respiratory Questionnaire<br>(SGRQ) total score (derived from | Yes |

| Objectives | Endpoints | Assessed in Strategic Interim |
|---|---|---|
| | SGRQ-C) | |
| | SGRQ responder analysis | Yes |
| | Change from baseline for the COPD Assessment Test (CAT) total score | Yes |
| | CAT responder analysis | Yes |
| | Lung function (forced expiratory volume in 1 second [FEV1], FEV1 % predicted, forced vital capacity [FVC], FEV1/FVC ratio) | Yes |
| | Rescue medication use | Yes |
| | Participant experience of physical activity (subset of approximately 50% of participants) measured using Clinical Visit PROactive Physical Activity in COPD Tool (C-PPAC) | Yes <sup>[2]</sup> |
| To characterize the pharmacokinetics of danirixin in participants with COPD | Danirixin concentration and standard<br>pharmacokinetic (PK) parameters for<br>danirixin (e.g. AUC, Cmax, Tmax),<br>using dried blood spot data | No |
| Exploratory Objectives | Exploratory Endpoints | |
| To further explore study participants' experience | Time to first Clinically Important<br>Deterioration (CID) | No |
| with study treatment and overall experience with the study | SGRQ domains | Yes |
| To characterize the effect<br>of danirixin on lung<br>matrix<br>destruction/remodelling | Blood/serum/plasma biomarkers that<br>are indicative of extracellular matrix<br>turnover/remodelling (e.g. elastin and<br>collagen neo-epitopes) | No |
| Comparison between<br>dried blood spot and wet<br>whole blood analysis of<br>danirixin concentrations<br>in partipants with COPD | Danirixin concentration and standard<br>pharmacokinetic parameters for<br>danirixin (e.g. AUC, Cmax, Tmax) | No |

| Objectives | Endpoints | Assessed in Strategic Interim |
|---|---|---|
| To characterise danirixin exposure-response relationships for various safety parameters, if appropriate | Danirixin systemic exposure and<br>various efficacy/pharmacodynamic<br>(PD)/safety parameters, if appropriate | No |

- [1] AEs, serious AEs (SAEs), drug-related AEs, AEs leading to withdrawal, AEs of special interest (AESI), laboratory data, ECG
- [2] Summary of C-PPAC questionnaire responses only

## 2.3. Study Design



#### **Overview of Study Design and Key Features**

(Day 1). This analysis was performed in December 2017.

A protocol specified futility interim analysis based on the E-RS: COPD endpoint was conducted after approximately 150 participants had completed 3 months of study treatment. This analysis was performed in February 2018.

A further protocol specified strategic interim analysis will be conducted when approximately 450 participants have completed 6 months of treatment. This strategic interim will be used to support GlaxoSmithKline (GSK) decisions regarding additional investment and further development of danirixin. It will include endpoints as specified in Section 2.2 and in the list of data displays in Appendix 11. No changes will be made to the study based on the results of this strategic interim analysis unless a safety concern is identified.

Outputs containing unblinded treatment assignments will be created for all interim analyses and will only be made available to a limited number of GSK staff. Full details will be included in the study results dissemination plan (SRDP).

## 2.4. Statistical Hypotheses

The primary efficacy endpoint is the change from baseline of E-RS: COPD total score at Month 6. The primary objective of the study is to characterize the dose response of danirixin and select appropriate dose(s) for future drug development.

A model based probability inference approach in Bayesian framework will be used to guide decision-making around dose selection. The posterior probability that the change from baseline of E-RS: COPD total score for each active dose is less than placebo will be derived.

No formal statistical hypothesis will be tested in the primary efficacy analysis.

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

#### 3.1.1. Interim PK Analysis

After approximately 10 participants in the PK subset for each treatment group had completed Visit 3 (Day 1), an interim evaluation of danirixin PK parameters was undertaken. The purpose of the interim PK analysis was to determine if danirixin exposures were within the expected range. No formal HARP outputs were produced.

## 3.1.2. Futility Analysis

An interim analysis was conducted to allow for the possibility of stopping early for futility after approximately 150 participants had completed 3 months of treatment. This is described in a separate RAP. Outputs featuring unblinded treatment assignments were created and shared with the study team and those listed in the Study Results Dissemination Plan (SRDP).

#### 3.1.3. Strategic Analysis

When approximately 450 participants had completed 6 months of treatment, a further interim analysis was performed for strategic planning purposes, as described in this RAP. This analysis was planned to be used to aid in the planning of future studies and for a better understanding of benefit/risk profile of danirixin. No changes were made to the study based on the results of this strategic interim analysis.

The analyses were performed after the completion of the following sequential steps:

- 1. The date of the planned Visit 10 for the 450th completed participant (01AUG2018) had been met.
- 2. All required database cleaning activities had been completed by Data Management (DM) on data collected up until 01AUG18. Data collected between 02AUG2018 and 5SEP2018 (DBR) for ongoing subjects was not cleaned.
- 3. Unblinded randomization schedules were released by Randomization coordinator.

Data was reported in System Independent (SI) format. Outputs featuring unblinded treatment assignments were created for this strategic interim analysis, reviewed by the study team and shared with selective GSK personnel (to be included in the SRDP).

#### 3.1.4. Administrative Interims

Administrative assessments of danirixin exposure, efficacy and spirometry data may be undertaken during the conduct of the study as data becomes available. No decisions regarding study conduct will be made based on these assessments. The reporting team will have access to the unblinded participant treatment assignments. The unblinded study team (as defined in the 205724 Study Charter) will have access to unblinded aggregate data grouped by study treatment assignment.

An administrative interim was performed in October 2017 and included plots of E-RS: COPD total score (and the subgroups) over time by treatment, to aid internal decision-making on the project.

## 3.2. Final Analyses

The final planned analyses for this Clinical Data Interchange Standards Consortium (CDISC) study will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. SI data to Study Data Tabulation Model (SDTM) data conversion has been completed by Accenture and quality control (QC) of blinded SDTM has been completed by CDAD and DM. DM will provide the blinded SI PC dataset to Accenture.
- 3. All required database cleaning activities have been completed and final SI Source Data Lock (SDL) has been declared by DM.
- 4. Study is unblinded
  - Randomization schedules and container data are released in RANDALL NG.
  - SMS2000 data is released in HARP
- 5. The SDTMs (including the PK) are unblinded by clinical programming (or representative) using the interim unblinding process.
- 6. Database freeze (DBF) on unblinded SDTM datasets is declared by DM.

# 4. ANALYSIS POPULATIONS

# 4.1. Strategic Interim Analysis

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>(ALLSUB) | All participants screened and for whom a record exists on the study database. | <ul> <li>Participant disposition</li> <li>Reasons for withdrawal prior to randomization</li> <li>Inclusion/exclusion/randomization criteria deviations for non-randomized participants</li> <li>AEs and SAEs for non-randomized participants</li> </ul> |
| Intent-to-treat<br>(ITT) | <ul> <li>All randomized participants apart from those who were randomized in error (i.e. were also recorded as screen or run-in failures and did not receive a dose of study treatment).</li> <li>Any participant who receives a treatment randomization number will be considered to have been randomized.</li> <li>Randomized participants will be assumed to have received study medication unless definitive evidence to the contrary exists.</li> <li>Data will be reported according to the randomized treatment.</li> </ul> | <ul> <li>Selected efficacy displays as described in Section 7</li> <li>Strategic Interim only</li> </ul> |
| Modified<br>Intent-To-<br>Treat (mITT) | <ul> <li>Same as the Intent-to-treat population, but this population will be 'modified' in that all data summaries and analyses for this population will be based on the actual treatment received, if it is different to the randomized treatment.</li> <li>If any participant received more than one treatment during a treatment period, their data will be reported according to the treatment they received for the longest period of time.</li> </ul> | <ul><li>Study Population</li><li>Safety</li></ul> |
| Per Protocol<br>(PP) | All participants from the mITT population who<br>did not have a protocol deviation considered<br>to impact efficacy | Efficacy |
| Symptomatic | All participants in the PP population who have Chronic Mucus Hypersecretion (CMH) according to baseline SGRQ (see Section 14.6.2) and baseline E-RS: COPD total score (see Section 5.2) >=10. | <ul> <li>Study Population</li> <li>Selected efficacy displays as described in Section 7</li> <li>Strategic Interim only</li> </ul> |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

## 4.2. Final Analysis

The final analysis will use the same populations as above, plus additional populations as defined below.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| PK | All participants in the mITT population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values) obtained and analysed whilst on treatment with danirixin. | • PK |
| PK2 | All participants in the PK population who had at least 1 non-missing PK assessment (NQ values will be considered as non-missing values) obtained and analysed whilst on treatment with danirixin from a dry blood spot sample and corresponding wet whole blood sample. | PK Dry Blood Spot<br>vs Wet Whole<br>Blood |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

In the event one or more investigators are withdrawn from the study due to concerns over protocol deviation then a further population will be defined which will consist of all participants in the PP population excluding participants from those investigative sites. This population will be used to perform additional sensitivity analysis for the primary efficacy endpoint only and will only be defined if the combined enrolment at these sites exceeds  $\geq 2\%$  of the overall PP study enrolment. No other analyses will be repeated.

#### 4.3. Protocol Deviations

Protocol Deviations (PDs) will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (6JUL2018, V2.0):

- Data will be reviewed prior to SDL to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- Participants who received an incorrect treatment container will be captured as an important protocol deviation. Whether or not the incorrect container contained incorrect treatment will be identified following DBF in the analysis dataset and the PD will be flagged accordingly.
- This dataset will be the basis for the summaries and listings of protocol deviations.
- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarised and listed.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|------|----------------------------------------|-------------|--------------|
| | RandAll NG Data Displays for Reporting | | Reporting |
| Code | Description | Description | Order in TLF |
| D5 | Danirixin 5mg | DNX 5mg | 2 |
| D10 | Danirixin 10mg | DNX 10mg | 3 |
| D25 | Danirixin 25mg | DNX 25mg | 4 |
| D35 | Danirixin 35mg | DNX 35mg | 5 |
| D50 | Danirixin 50mg | DNX 50mg | 6 |
| PO | Placebo oval | Placebo | 1 |
| PR | Placebo round | Placebo | 1 |

Treatment comparisons will be displayed as in the danirixin dose column with the descriptor: Column vs Placebo.

## 5.2. Baseline Definitions

Any assessments made after the start of study treatment will not be included in the derivation of baseline. Assessments made on the same day as the start of treatment are assumed to be taken prior to first dose.

If baseline data are missing, no derivation will be performed and baseline will be set to missing.

| Parameter | Baseline Used in Data Display |
|---|---|
| E-RS: COPD total and subscale scores | Mean score during a stable period between (Latest of (7 days before Study treatment start date (Day 1) and day of Visit 1 (Screening)) and day before Day 1 of study treatment. Data must be present on at least 4 days |
| EXACT (for determining EXACT events) | Defined according to the EXACT User Manual v8.0 (Evidera, 2016a) |
| SGRQ total and domain scores | Day 1 |
| CAT score | Day 1 |
| Rescue use (diary card and sensor data, mean number of puffs/occasions per day and percentage of rescue-free days) | Mean score during a stable period between (Latest of (7 days before Study treatment start date (Day 1) and day of Visit 1 (Screening)) and day before Day 1 of study treatment. Data must be present on at least 4 days. |
| PROactive score | A PROactive Total Score and two domain scores (amount and difficulty) will be derived using data from the C-PPAC questionnaire on Day 1 and physical activity |

| Parameter | Baseline Used in Data Display |
|---|---|
| | monitor worn between Visit 2 and Visit 3 (7 days). The activity monitor must have been worn for at least 3 days with >=8 hours wearing (the 3 days do not need to be consecutive). Further details of the derivation are described in Section 14.6.3 and in the IMI PROactive user manual (14JUN16). |
| Blood pressure (BP) | Latest pre-dose assessment with a non-missing value for both systolic and diastolic BP, including those from unscheduled visits |
| Pulse rate, laboratory data, ECG | Latest pre-dose assessment with a non-missing value for the individual assessment, including those from unscheduled visits |
| Post-bronchodilator<br>(BD) FEV1, post-BD<br>FVC | Day 1 |

#### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be summarized by country and investigative site. Country will be included as a fixed effect in statistical models and treatment by country interaction investigated as described in Section 7 and Section 8. Results will be presented for all countries combined except as specified in Section 7.

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The covariates and other strata listed below will be used in statistical models and treatment by covariate/stratum investigated as defined in Section 7, Section 14.6.2 and Section 14.6.3.

| Category | Details |
|---|---|
| Strata | Smoking status |
| Covariates | Treatment, visit/Month, baseline, smoking status at screening, country, gender, exacerbation history (≤1, ≥2 moderate/severe), post-bronchodilator % predicted FEV1, CMH status at baseline, season of data collection. |

## 5.4.2. Examination of Subgroups

The subgroups listed below will be used in statistical analyses as described in Section 7.

| Subgroup | Categories |
|---|---|
| Season | Spring, Summer, Fall, Winter (see Section 14.6.3) |
| Country | Australia, Canada, Germany, Korea, Netherlands, Poland, Romania, Spain, US |
| Exacerbation history | History of ≥2 moderate/severe exacerbations vs <2 moderate/severe exacerbation |
| COPD medication at Baseline | ICS+LABA+LAMA vs. ICS+LABA vs. LABA+LAMA vs. Other COPD medication |
| ERS10 | Baseline E-RS: COPD Total Score <10, ≥10 |
| CAT10 | Baseline CAT Score <10, ≥10 |
| Smoking status at Screening | Current, Former |
| % predicted FEV1 at Screening | <50%, ≥50% |
| CMH status at baseline | CMH+, CMH- (see Section 14.6.2) |

## 5.5. Multiple Comparisons and Multiplicity

No multiplicity adjustment will be made for this study, as the primary objective of the study is to model the danirixin dose response and use it to select Phase III dose(s).

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|-----------------------------------------------------------|
| 14.3 | Appendix 3: Assessment Windows |
| 14.4 | Appendix 4: Study Phases |
| 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 14.6 | Appendix 6: Derived and Transformed Data |
| 14.7 | Appendix 7: Reporting Standards for Missing Data |
| 14.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

Study population displays including analyses of participant disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Results will be presented for each treatment and overall.

Details of the planned displays including the population to be used for each display and which displays are produced for the strategic interim are presented in Appendix 11. Additional details are provided below.

#### 6.1.1. Demographic and Baseline Characteristics

The summary of exacerbation history at Screening will include the number and percentage of participants reporting mild, moderate, severe and moderate/severe exacerbations  $(0, 1, \ge 2)$ ; see Section 14.6.2) in the 12 months prior to screening.

#### 6.1.2. Prior and Concomitant Medications

Non-COPD medication tables will report by Anatomical Therapeutic Chemical (ATC) level 1 classification and ingredient. Multi-ingredient non-COPD medications will be presented according to their combination ATC classification rather than the classifications of the ingredients.

COPD medication tables will report by respiratory medication class (RMC) and ingredient (See Section 14.6.2). The number and percentage of participants taking each medication in the RMC categories (defined in Section 14.6.2) will be presented.

The number and percentage of subjects taking each medication in the RMC categories ICS, LABA, LAMA, PDE4 inhibitors, Xanthines, Anti-IgE, Anti-IL5 and combinations of these RMCs on the day of the Screening visit, at Baseline (Day 1) and at Month 6 will be presented.

### 6.1.3. Exposure and Treatment Compliance

Calculation of treatment compliance will be based on the number of tablets dispensed and returned as described in Section 14.6.2. Calculation of diary compliance will be based on the number of days with non-missing E-RS: COPD total score as described in Section 14.6.2. Percentage treatment and diary compliance will be summarized categorically and with descriptive statistics.

#### 7. EFFICACY ANALYSES

Details of the planned displays including the population to be used for each display and which displays are produced for the strategic interim are presented in Appendix 11. Additional details are provided below.

For this study, no data were scheduled to be collected after discontinuation of study treatment, therefore accounting for non-recorded missing data following study withdrawal is addressed by the strategy for the intercurrent event of treatment discontinuation

## 7.1. Primary Efficacy Analyses

#### 7.1.1. Month 6 E-RS: COPD Total Score Dose-Response Analysis

The estimand is the effect of actual treatment in the population of participants who did not experience a protocol deviation considered to impact efficacy and completed six months of treatment.

A Bayesian dose response model will be applied to the change from baseline to Month 6 and used to estimate the treatment difference between placebo and each dose.

The dose-response model will be fitted using Bayesian techniques with non-informative priors for E0 and Emax and a functional uniform prior (FUP) for ED50 and the slope parameter, m (Bornkamp, 2014). The rationale for this choice of inference is that the FUP shrinks the dose-response towards a flat line throughout the dose range, therefore providing more conservative estimates of the dose-response relationship compared to maximum likelihood.

For the strategic interim, the posterior predictive probability of success (PPS) at the end of the study will be calculated for each dose using the formula suggested by Spiegelhalter et al. (Spiegelhalter, 2004) as follows:

$$PPS = \Phi \left[ \frac{\sqrt{(m+n)}}{\sqrt{mn}} \frac{(-my_m)}{\sigma_{trt \ diff}} + \sqrt{\frac{m}{n}} z_{0.9} \right]$$

Where m is the average number of participants with Month 6 data in the placebo and comparative dose arm, n is the average number of participants yet to be observed (assuming 90% of participants, rounded to the nearest integer, in each treatment group will provide month 6 data at end of study. If the actual number of participants at month 6 exceeds this, the actual number will be used),  $V_m$  is the posterior mean difference from the fitted model, and  $\sigma_{trt\ diff}$  is the standard deviation (SD) of the posterior mean difference.

#### 7.1.1.1. **Endpoint**

Change from baseline in Month 6 E-RS: COPD total score as defined in Section 14.6.3.

#### 7.1.1.2. Summary Measure

For the strategic interim, the summary measure is the posterior predictive probability of success for each danirixin dose, where success is the probability that a true difference from placebo is less than 0 is >95% at Month 6.

For the final analysis, the summary measure is the posterior probability that a true difference from placebo is less than 0 at Month 6 for each danirixin dose.

#### 7.1.1.3. Population of Interest

PP population.

## 7.1.1.4. Strategy for Intercurrent (Post-Randomization) Events

For the primary efficacy analysis, the intercurrent event of interest is occurrence of a protocol deviation considered to impact efficacy during the treatment period (see Appendix 1). An 'as treated' strategy will be used to account for this event - only Month 6 E-RS: COPD data (see Section 14.6.3) collected prior to the occurrence of a protocol deviation considered to impact efficacy will be used in the analysis.

The intercurrent event of treatment discontinuation is accounted for in the endpoint definition as only data at Month 6 will be used.

#### 7.1.1.5. Statistical Analyses / Methods

#### 7.1.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Change from baseline in Month 6 E-RS: COPD total score

#### **Model Specification**

#### Bayesian dose response model:

- Models of the following form will be considered:
  - Response=E0+ Emax\* f(dose)
    - Log-linear model: f(dose)=log(dose+0.01), where 0.01 is an offset to allow the model to fit for zero dose (placebo).
    - 3-parameter emax model: f(dose)=dose/(dose+ed50)
    - 4-parameter emax model: f(dose)=dose^m/(dose^m+ED50^m)

#### Where:

- E0 = the response at dose = 0 (placebo).
- Emax = the maximal response over placebo,
- o ED50= the dose that yields 50% of the maximal response,
- m= dose-response slope parameter.
- The log-linear, 3-parameter emax and 4-parameter emax model will be fitted without adjusting
  for covariates. If possible, covariates (i.e., baseline, smoking status, country) will be included in
  the E0 and Emax terms of the model for the final analysis
- Normal non-informative priors will be used for the E0 and Emax parameters with mean 0 and SD 100. A FUP will be used for the ED50 and m parameters (Bornkamp, 2014), where the

- prior density for the FUP is based on all the parameters in the model. An inverse -gamma prior with shape of 0.001 and scale of 0.001 will be used for the residual variance.
- Parameters will be blocked such that the MCMC procedure samples from E0 and Emax first, then the ED50 and m parameters and then finally the residual variance parameter.
- For the functional uniform priors, the density will be calculated for values of dose from 0.0001 to 50 in steps of 5 (i.e. 0.0001, 5.0001, 10.0001,..., 50.0001).
- 3 MCMC chains will be fitted using the following starting values (as required for the parameters in each particular model):

| Parameter | Chain 1 | Chain 2 | Chain 3 |
|-------------------|-------------------------------------|---------|---------|
| E0 | Posterior mean for placebo from | -15 | 15 |
| | MMRM at Month 6 (See Section 7.1.3) | | |
| Emax | Posterior mean for 50mg dose from | 15 | -15 |
| | MMRM at Month 6 (See Section 7.1.3) | | |
| ED50 | 25 | 10 | 50 |
| М | 1 | 2 | 4 |
| Residual variance | 6 | 8 | 10 |

- 100,000 MCMC samples will be generated using a thin of 50 to leave 2000 retained samples, and after a burn-in of 10,000 samples for each of the three sets of starting values. All postburn-in samples from the 3 chains will be used for inference. The number of samples generated and the thin may be increased to reduce the ratio of the MCSE to the posterior SD, as deemed necessary.
- The seeds used to for the three chains were generated using the ranuni function in SAS and are listed in Section 14.5.2.
- The best fitting model will be the model with the smallest average DIC over the 3 chains where
  convergence is deemed to have been achieved. If the best fitting model is one that adjusts for
  covariates, all outputs will be presented adjusting for the mean in the observed covariate.
- Production and QC will be deemed to have agreement if the QC value is the following range:
  - if a number is reported to 0dp and there is a difference of  $\pm$  1 (number of participants must agree)
  - if a number is reported to 1dp and there is a difference of  $\pm$  0.1
  - if a number is reported to 2dp and there is a difference of  $\pm$  0.01
  - if a number is reported to 3dp and there is a difference of  $\pm$  0.001
  - if a number is reported to 4dp and there is a difference of ± 0.0001

#### **Model Checking & Diagnostics**

- Posterior density plots and plots of the posterior samples (chains) will be produced for all the parameters in the model.
- The posterior density for the adjusted mean change from baseline in E-RS: COPD total score in each treatment group and differences versus placebo for each danirixin dose will be plotted.
- The Gelman-Rubin R estimate from the three chains will be calculated for all parameters in the model and the differences from placebo for each danirixin dose.

#### **Model Results Presentation**

The following will be presented for each analysis based on the best fitting model using all post-burn in samples available.

- The posterior mean, median, SD and 90% credible interval (CrI) for the change from baseline in E-RS: COPD total score for each treatment group.
- The posterior mean and 90% CrI for the difference from placebo for each danirixin dose.

- The posterior probability that difference from placebo is less than 0, -0.5, -1, -1.5 and -2 for each danirixin dose.
- For the strategic interim, the posterior predictive probability of success for each danirixin dose, where success is the probability that the difference from placebo is less than 0 is >95%.
- A figure of the fitted mean dose response model with the 90% Crl for all possible doses in the
  dose range, overlaid with the Month 6 adjusted posterior means and 90% Crl from the
  longitudinal model in Section 7.1.3.

## **Sensitivity and Supportive Analyses**

At the strategic interim, a supportive analysis will be conducted to estimate the effect of actual
treatment in the population of participants who were confirmed as having CMH according to
SGRQ, were symptomatic at baseline, did not experience a protocol deviation considered to
impact efficacy, and completed six months of treatment. The population used will be the
Symptomatic population; all other details will be the same as for the primary analysis.

#### 7.1.2. E-RS: COPD Subscale Scores Dose-Response Analysis

The primary analysis described in Section 7.1.1 will be repeated for the three E-RS: COPD subscale scores of breathlessness, cough and sputum and chest symptoms.

## 7.1.3. E-RS: COPD Total and Subscale Scores Longitudinal Analysis

The estimand is the effect of actual treatment in the population of participants who did not experience a protocol deviation considered to impact efficacy. A supportive analysis will be performed to assess the effect of randomized treatment in all randomized and dosed participants.

A Bayesian mixed effects analysis with repeated measures (MMRM) will be performed on the monthly E-RS: COPD total and subscale scores.

A frequentist MMRM analysis will be performed on the monthly E-RS: COPD total scores and repeated to assess the impact of various covariates.

#### **7.1.3.1.** Endpoint

Change from baseline in monthly mean E-RS: COPD total and subscale scores as defined in Section 14.6.3.

#### 7.1.3.2. Summary Measure

For the Bayesian MMRM the summary measure is the adjusted posterior mean difference from placebo for each danirixin dose.

For the frequentist MMRM the summary measure is the adjusted mean difference from placebo for each danirixin dose.

#### 7.1.3.3. Population of Interest

PP population.

#### 7.1.3.4. Strategy for Intercurrent (Post-Randomization) Events

A 'hypothetical' strategy will be used to account for the intercurrent events of occurrence of a protocol deviation considered to impact efficacy during the treatment period (see Appendix 1) and treatment discontinuation, to estimate the effect if participants had not deviated from the protocol and remained on treatment. Only E-RS: COPD data prior to the occurrence of a protocol deviation considered to impact efficacy or treatment discontinuation will be used in the analysis. Subsequent data up to Month 6 will be assumed to be missing at random (MAR).

#### 7.1.3.5. Statistical Analyses / Methods

#### 7.1.3.5.1. Bayesian MMRM Methodology Specification

#### **Endpoint / Variables**

Change from baseline in monthly E-RS: COPD total and subscale scores

#### **Model Specification**

- Bayesian mixed models repeated measures approach.
- The model will include treatment\*visit, baseline\*visit, country and smoking status parameters.
   Note that the model will not include an intercept. Visit will consist of six levels (Month 1-Month 6), and Treatment will consist of six levels (placebo and 5 active doses). If the model does not run, the country covariate will be removed.
- The priors for the mean vector for each of the parameters (i.e covariates) will each follow a normal distribution with mean 0 and SD 1000. The prior for the variance-covariance will follow an inverse Wishart distribution with degrees of freedom equal to the number of visits and an identity scale array. 150,000 samples will be generated with a thin of 75 after a burn-in of 10,000 samples. The number of samples or thin may be increased as needed to reduce the MCSE/SD<0.01 as deemed necessary.</p>
- Three chains will be used to calculate the gelman-rubin R statistic:
  - Chain 1: The starting value for all covariates in the model will be 0.
  - Chain 2: The starting value for all covariates in the model will be 2.
  - Chain 3: The starting value for all covariates in the model will be -2.
- The seeds used to for the three chains were generated using the ranuni function in SAS and are listed in Section 14.5.2.
- All post-burn-in samples will be used when creating outputs.

#### **Model Checking & Diagnostics**

- Posterior density plots and plots of the posterior samples (chains) will be produced for all the parameters in the model.
- The posterior density for the adjusted mean change from baseline in E-RS: COPD score in each treatment group and differences versus placebo for each danirixin dose will be plotted.
- The Gelman-Rubin R estimate from the three chains will be calculated for all parameters in the model and the differences from placebo for each danirixin dose.
- Distributional assumptions underlying the model used for analyses using MMRM will be
  examined by obtaining a normal probability plot of the residuals and a plot of the residuals
  versus the fitted values (i.e. checking the normality assumption and constant variance
  assumption of the model respectively) to gain confidence that the model assumptions are

reasonable. Plots of residuals versus covariates and baseline versus response will also be examined.

#### **Model Results Presentation**

- The adjusted posterior mean change from baseline and the associated 90% equi-tailed CrI for each Month for each treatment.
- The adjusted mean difference from placebo and the associated 90% equi-tailed CrI for each Month for each danirixin dose.
- The probability that each treatment difference is less than 0, -0.5, -1, -1.5 and -2 for each month for each danirixin dose.
- A figure of the posterior mean and 90% equi-tail Crl for each Month for each treatment.

#### **Sensitivity and Supportive Analyses**

- At the strategic interim a supportive analysis of monthly E-RS: COPD total score will be
  conducted to estimate the effect of actual treatment in the population of participants who were
  confirmed as having CMH according to SGRQ, were symptomatic at baseline, and did not
  experience a protocol deviation considered to impact efficacy. The population used will be the
  Symptomatic population; all other details will be the same as for the primary analysis.
- At the strategic interim a further supportive analysis will be conducted to estimate the effect of the randomized treatment. The population used will be the ITT (according to randomized treatment). A 'treatment policy' strategy will be used to account for the intercurrent event of occurrence of a protocol deviation considered to impact efficacy during the treatment period (see Appendix 1). All E-RS: COPD data up the time of treatment discontinuation or Month 6 (see Section 14.6.3) will be used in the analysis, regardless of any protocol deviation. A 'hypothetical' strategy will be used to account for the intercurrent event of treatment discontinuation. Data after treatment discontinuation will be considered MAR.

#### 7.1.3.5.2. Frequentist MMRM Methodology Specification

#### **Endpoint / Variables**

Change from baseline in monthly E-RS: COPD total score

#### Model Specification

- The following covariates will be included in the model: baseline, country, smoking status at screening, treatment, Month, Month\*baseline and Month\*treatment interactions, where Month is nominal. Month will consist of six levels (Month 1-Month 6), and treatment will consist of six levels (placebo and 5 active doses)
- Two models will be fitted; one with a response variable of E-RS: COPD Total Score, and one
  with a response variable of change from baseline in E-RS: COPD Total Score.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used. If this method does not run, the residual method will be used instead
- The OM option will be used to derive the least square (LS) means using coefficients which are based on the participants used in the analysis. The OM option requires an OM dataset which has a row for every participant-visit combination that contains all of the covariates used in the model and a macro variable containing the mean baseline for the participants used in the

analysis.

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analyses using MMRM will be
examined by obtaining a normal probability plot of the residuals and a plot of the residuals
versus the fitted values (i.e. checking the normality assumption and constant variance
assumption of the model respectively) to gain confidence that the model assumptions are
reasonable. Plots of residuals versus covariates and baseline versus response will also be
examined.

#### **Model Results Presentation**

- LS mean and LS mean changes from baseline with their corresponding standard errors (SEs) for each Month and each treatment
- Estimated treatment differences from placebo and corresponding 90% confidence intervals (CIs) and p-values for each Month and each danirixin dose.
- A figure of LS mean changes from baseline and 90% CIs for each treatment by Month will be generated.
- A figure of LS mean and 90% Cls for each treatment by Month will be generated.
- The type III tests of fixed effects from the model will be presented.

## **Summary Results Presentation**

- A figure of daily mean E-RS: COPD total and subscale scores over time (Days -7 to 168) for the PP population.
- A figure of daily mean E-RS: COPD total and subscale scores over time by completer status (Days -7 to 168) for the PP population.
- A figure of daily mean change from baseline E-RS: COPD total and subscale scores over time for the PP population.
- A figure of daily mean (± SE) change from baseline E-RS: COPD total and subscale scores
  over time for each dose and placebo in a separate panel. This figure will be produced for the
  PP and Symptomatic populations (Strategic interim only).
- A figure of daily mean (± SE) E-RS: COPD total and subscale scores over time (Days -7 to 168) for each dose and placebo in a separate panel. This figure will be produced for the PP population.
- Summary statistics for baseline E-RS: COPD total and subscale scores for each treatment and overall for participants with non-missing score for each Month, for the PP and Symptomatic (Strategic interim only) population.
- Summary statistics for raw and change from baseline monthly mean E-RS: COPD total and subscale scores for each month for each treatment, for the PP and Symptomatic population (Strategic interim only).
- Empirical distribution function plot of E-RS: COPD Total Scores at Baseline and at Month 6.

## 7.2. Secondary Efficacy Analyses

The estimand is the effect of actual treatment in the population of participants who did not experience a protocol deviation considered to impact efficacy.

A supportive analysis will be conducted to estimate the treatment policy effect of the randomized treatment on the annual rate of HCRU exacerbations in all randomized and dosed participants.

# 7.2.1. Annual Rate of HCRU Exacerbations and Annual Rate of EXACT Events

#### 7.2.1.1. **Endpoint**

Annual rate of moderate/severe HCRU exacerbations as defined in Section 14.6.3.

Annual rate of EXACT events as defined in Section 14.6.3.

#### 7.2.1.2. Summary Measure

Rate ratio (also expressed as percentage rate reduction) for each danirixin dose vs. placebo

#### 7.2.1.3. Population of Interest

PP population

#### 7.2.1.4. Strategy for Intercurrent (Post-Randomization) Events

The intercurrent events of interest are occurrence of a protocol deviation considered to impact efficacy during the treatment period (see Appendix 1) and treatment discontinuation. An 'as treated' strategy will be used to account for these events to estimate the effect if participants had not deviated from the protocol and remained on treatment. Only HCRU exacerbations/EXACT events prior to the occurrence of a protocol deviation considered to impact efficacy will be used in the analysis.

#### 7.2.1.5. Statistical Analyses / Methods

#### 7.2.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- Annual rate of On-treatment moderate/severe HCRU exacerbations
- Annual rate of On-treatment EXACT events

#### **Model Specification**

- Bayesian generalized linear model assuming a negative binomial distribution for the underlying exacerbation rate with a log link function
- Terms in the model:
  - Response: number of on-treatment, moderate/severe HCRU exacerbations or EXACT events per participant.
  - Categorical: treatment group, gender, exacerbation history (≤1, ≥2 moderate/severe), smoking status (screening), country
  - Continuous: post-bronchodilator % predicted FEV1 (Screening)
  - An offset to account for the length of time on treatment for each participant will be

- included in the model as log<sub>e</sub> (length of time) as defined in Section 14.6.3.
- Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.
- All the terms in the model will follow a normal distribution with a mean of 0 and a SD of 100, except for dispersion which follows a gamma distribution with shape and inverse scale of 0.001.
- Three chains will be used to calculate the gelman-rubin R statistic:
  - Chain 1: The starting value for all covariates in the model will be the maximum likelihood estimation (MLE), except dispersion which will be 0.1.
  - Chain 2: The starting value for all covariates in the model will be 130% of the MLE, except for dispersion which will be 0.2.
  - Chain 3: The starting value for all covariates in the model will be 70% of the MLE, except for dispersion which will be 0.4.
- The seeds used to for the three chains were generated using the ranuni function in SAS and are listed in Section 14.5.2.
- Burn-in 2000, thin 5, and 10,000 MCMC samples will be generated for 2000 retained samples

#### **Model Checking & Diagnostics**

- The fit of the regression models will be examined using "Q-Q" plots of the standardized residuals. Interpretation of these plots will be aided by the addition of simulated envelopes as proposed by Atkinson (Atkinson, 1985).
- The Gelman-Rubin R estimate will be calculated for all parameters in the model and the rate ratios vs. placebo for each danirixin dose.
- Autocorrelation plots will be visually inspected to assess degree of autocorrelation (should decline rapidly and show no oscillation patterns).

#### Model Results Presentation

- Model estimated median exacerbation/event rate and associated 90% Crl for each treatment group
- Median rate ratio and associated 90% Crl, percent reduction in annual exacerbation/event rate and associated 90% Cl for each danirixin dose vs. placebo
- The probability that the true exacerbation rate ratio is less than 1, 0.9 and 0.8 for each danirixin dose will be presented
- A figure of the rate ratios and associated 90% Crls for each danirixin dose vs. placebo

#### **Summary Results Presentation**

#### For HCRU exacerbations:

- Number and percent of participants reporting an exacerbation (mild, moderate, severe and moderate/severe), number and percent of participants with each number of moderate/severe exacerbations (0, 1, ≥2), the total number of exacerbations per treatment and annual raw exacerbation rate (as defined in Section 14.6.3). This table will be repeated for HCRU exacerbations that were treated with Antibiotics and will include the number and percentage of participants who were receiving ICS treatment at the time of the exacerbation.
- For each moderate/severe exacerbation, the outcome, severity, duration, whether the
  exacerbation led to hospitalization, systemic/oral corticosteroids being taken, antibiotics being
  taken, or emergency room visit.

#### For EXACT events:

• Number and percent of participants reporting an EXACT-defined event, number and percent of

participants with each number of EXACT-defined events (0, 1, ≥2), the number of EXACT-defined events and annual raw event rate (as defined in Section 14.6.3) will be summarized for all events and for recovered, censored and persistent worsening events separately for each treatment group. The duration and severity (indicated by the maximum observed value and duration) will be reported for all events.

## Sensitivity and Supportive Analyses

At the strategic interim a supportive analysis of HCRU exacerbations will be conducted to
estimate the effect of the randomized treatment. The population used will be the ITT
(according to randomized treatment). A 'treatment policy' strategy will be used to account for
the intercurrent event of occurrence of a protocol deviation considered to impact efficacy during
the treatment period (see Appendix 1). All on-treatment exacerbations up the time of treatment
discontinuation will be used in the analysis, regardless of any protocol deviation. An 'as treated'
strategy will be used to account for the intercurrent event of treatment discontinuation – no
exacerbations will be recorded after treatment discontinuation/study withdrawal.

#### 7.2.2. Time to First HCRU Exacerbation and EXACT Event

#### **7.2.2.1.** Endpoint

Time to first moderate/severe HCRU exacerbation as defined in Section 14.6.3.

Time to first severe HCRU exacerbation as defined in Section 14.6.3.

Time to first EXACT event as defined in Section 14.6.3.

#### 7.2.2.2. Summary Measure

Hazard ratio (also expressed as percentage risk reduction) for each danirixin dose vs. placebo)

#### 7.2.2.3. Population of Interest

PP population

#### 7.2.2.4. Strategy for Intercurrent (Post-Randomization) Events

The intercurrent events of interest are occurrence of a protocol deviation considered to impact efficacy during the treatment period (see Appendix 1) and treatment discontinuation. An 'as treated' strategy will be used to account for these events to estimate the effect if participants had not deviated from the protocol and remained on treatment. Only first exacerbations/EXACT events prior to the occurrence of a protocol deviation considered to impact efficacy will be used in the analysis.

#### 7.2.2.5. Statistical Analyses / Methods

#### 7.2.2.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- Time to first On-treatment moderate/severe HCRU exacerbation
- Time to first On-treatment severe HCRU exacerbation
- Time to first On-treatment EXACT event

#### **Model Specification**

- Bayesian proportional hazards model
- Terms in the model:
  - Response: time to first on-treatment, moderate/severe HCRU exacerbation or EXACT event
  - Categorical: treatment group, gender, exacerbation history (≤1, ≥2 moderate/severe), smoking status (screening), country
  - Continuous: post-bronchodilator % predicted FEV1 (Screening)
  - Non-informative priors will be used for all modelling parameters. Wherever possible conjugate priors will be utilised.
  - All the terms in the model will follow a normal distribution with a mean of 0 and a SD of 100
- The 'exact' method will be used for handling ties. If the analysis will not run using the 'exact' method, then the 'Efron' method for handling ties will be used instead.
- Three chains will be used to calculate the gelman-rubin R statistic:
  - Chain 1: The starting value for all covariates in the model will be the MLE, except dispersion which will be 0.1.
  - Chain 2: The starting value for all covariates in the model will be 130% of the MLE, except for dispersion which will be 0.2.
  - Chain 3: The starting value for all covariates in the model will be 70% of the MLE, except for dispersion which will be 0.4.
- The seeds used to for the three chains were generated using the ranuni function in SAS and are listed in Section 14.5.2.
- Burn-in 2000, thin 5, and 10,000 MCMC samples will be generated for 2000 retained samples
- Kaplan-Meier survivor functions will be obtained for each treatment group using PROC LIFETEST with a TIME statement.

## **Model Checking & Diagnostics**

 The proportional hazards assumption will be examined by obtaining the Kaplan-Meier estimates of the survival function S(t) over time separately for each treatment group. In addition, the In {-ln[S(t)]} plot will be produced.

#### **Model Results Presentation**

- Hazard ratio and the percent reduction in risk for each danirixin dose compared with placebo with associated 90% Crl.
- The probability of having an event, 90% Crl and first quartile and median time to event for each treatment group will be presented.
- The probability that the true hazard ratio is less than 1 for each danirixin dose will be presented.

 Kaplan-Meier curves showing the probability of having an event over time for each treatment group separately plotted on the same figure

#### 7.2.3. E-RS: COPD Total and Subscale Scores Responder Analysis

#### **7.2.3.1.** Endpoint

Response according to E-RS: COPD total score, subscale scores, SGRQ total score or CAT score as defined in Section 14.6.3.

#### 7.2.3.2. Summary Measure

Ratio of odds of being a responder vs. not for each danirixin dose vs. placebo

#### 7.2.3.3. Population of Interest

PP population

#### 7.2.3.4. Strategy for Intercurrent (Post-Randomization) Events

A 'hypothetical' strategy will be used to account for the intercurrent events of occurrence of a protocol deviation considered to impact efficacy during the treatment period (see Appendix 1) and treatment discontinuation, to estimate the effect if participants had not deviated from the protocol and remained on treatment. Only response data prior to the occurrence of a protocol deviation considered to impact efficacy or treatment discontinuation will be used in the analysis. Subsequent data up to Month 6 will be assumed to be missing at random (MAR).

#### 7.2.3.5. Statistical Analyses / Methods

#### 7.2.3.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

 Response according to E-RS: COPD total score, subscale scores, SGRQ total score or CAT score

#### **Model Specification**

- Generalized linear mixed model
- Terms in the model:
  - Dependent : response (yes/no)
  - o Categorical: treatment group, smoking status (screening), country, visit/month
  - Continuous : baseline
  - Interaction: baseline\*visit/month, treatment group\*visit/month
- The model will be fit with an unstructured variance-covariance matrix with one single model to include all visits/months where the assessment in question is scheduled to be performed.
- Computation of confidence intervals for the odds ratios is based on the individual Wald tests.

#### **Model Checking & Diagnostics**

 Pearson residuals will be plotted by using PLOTS=PEARSONPANEL option for the model statement in SAS.

#### **Model Results Presentation**

- Number and percentage of responders and non-responders for each treatment at each visit/month
- Odds ratio for comparison of each danrixin dose with placebo, with associated 90% CI and p-value

#### 7.2.4. SGRQ Total Score and CAT Score

SGRQ total score and CAT score at each visit will be analysed using the same methodology as for E-RS: COPD total and subscale scores longitudinal analysis (as described in Section 7.1.3.5.1). Visit will be substituted for Month. A figure of mean and 90% CIs for each treatment over time will be generated for SGRQ Total Score and CAT Score.

#### 7.2.5. Rescue Use

The monthly mean number of puffs of rescue use per day according to diary card data and the monthly mean number of occasions of rescue use per day according to sensor data and the monthly percentage of rescue-free days according to diary card data and according to sensor data will be analysed using the same methodology as for E-RS: COPD total and subscale scores longitudinal analysis (as described in Section 7.1.3.5.2). A figure of daily mean number of puffs of rescue medication per day using diary data over time and daily mean number of occasions of rescue medication per day using sensor data over time will be generated for the PP population.

Additional analysis of rescue use according to sensor data may be performed and will be defined in a separate RAP.

#### 7.2.6. Physical Activity

Assessment of physical activity during clinical visits (C-PPAC) has been developed to capture experience of physical activity in participants with COPD. This physical activity data will be combined with activity monitor data to assess physical activity experience according to the IMI PROactive User Guide (14JUN16). A PROactive Total Score and two domain scores (amount and difficulty) will be derived.

Raw and change from baseline PROactive Total Score and Domain scores (Amount and Difficulty) will be summarized.

For the strategic interim, the responses to the C-PPAC questions at each visit will be summarized.

Additional analysis of activity monitor data may be performed and will be defined in a separate RAP.

## 7.3. Exploratory Efficacy Analyses

#### 7.3.1. E-RS: COPD Total Score

For the final analysis the list of subgroups may be amended.

#### **Exploratory Statistical Analyses**

#### **Model Specification**

For the PP population, an assessment of whether the effect of treatment on E-RS: COPD Total Score is modified by:

- Baseline E-RS: COPD Total Score (continuous) (Strategic Interim only)
- Smoking Status at Screening
- Country (Strategic Interim only)

will be made by fitting separate repeated measures models, identical to the MMRM model described in Section 7.1.3.5.2 but also including additional terms for the treatment by factor interaction.

An assessment will be made of whether the effect of treatment on E-RS: COPD Total Score is modified by the following factors (as defined in Section 5.4.2):

- Percent Predicted FEV1 at Screening (continuous)
- Baseline CAT Score (continuous)
- Exacerbation history (Strategic Interim only)
- COPD Medication at Baseline (Strategic Interim only)
- CMH status at baseline (Strategic Interim only)
- Season (Strategic Interim only)

This will be made by fitting separate repeated measures models, identical to the model described above but also including additional terms for the factor and the treatment by factor interaction.

If an interaction from these analyses is significant at the 10% level it implies that the effect of treatment on E-RS: COPD Total Score is modified by the factor. The analysis will be run by each level of the factors as listed below regardless of significance level (excluding any groups with sparse data):

- Baseline E-RS: COPD Total Score <10, ≥10 (Strategic Interim only)</li>
- Smoking Status at Screening Former, Current
- Country (Strategic Interim only)
- Percent Predicted FEV1 at Screening <50, ≥50</li>
- Baseline CAT Score <10, ≥10</li>
- Exacerbation history (history of ≥2 moderate/severe exacerbations, <2 moderate/severe exacerbation) (Strategic Interim only)
- COPD Medication at Baseline (ICS+LABA+LAMA vs. ICS+LABA vs. LABA+LAMA vs. Other COPD medication) (Strategic Interim only)
- CMH +, (Strategic Interim only)
- Season (The estimates from this model will be presented for each season.) (Strategic Interim only)

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analyses using MMRM will be examined by
obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values
(i.e. checking the normality assumption and constant variance assumption of the model respectively)
to gain confidence that the model assumptions are reasonable. Plots of residuals versus covariates
and baseline versus response will also be examined.

#### **Exploratory Statistical Analyses**

#### **Model Results Presentation**

- The interaction p-values from the interactions of treatment with the factors above will be presented.
- Comparisons of each danirixin dose with placebo for each level of each categorical subgroup.
- LS Mean changes from baseline estimates for each treatment by visit (except for season) along with 90% CIs will be obtained for each level of the subgroup.
- LS Mean changes from baseline estimates for each treatment along with 90% CIs will be obtained for each level of the season subgroup.
- LS Mean changes from baseline estimates and 90% CIs will be plotted against treatment in separate panels for each level of the factor for Month 6 (except for season).LS Mean changes from baseline estimates and 90% CIs will be plotted by treatment for each level of the season subgroup.
- If an interaction between treatment and factor is significant at the 10% level an additional plot of LS
  Mean changes from baseline and 90% CIs against treatment by Month will be produced with a
  separate plot for each level of the factor (except for season).

#### **7.3.2. CAT Score**

CAT score will be analysed using the same methodology as for E-RS: COPD total scores exploratory statistical analysis (as described in Section 7.3.1).

#### 7.3.3. Time to First Clinically Important Deterioration

Following the Strategic Interim, the study team decided not to report this exploratory endpoint.

#### 7.3.4. SGRQ Domain Scores

Raw and change from baseline SGRQ domain scores will be summarized.

#### 7.3.5. Participant Global Assessments

Participant global assessments of severity, change in severity, activity limitation and change in activity limitation will be summarized.
#### 8. SAFETY ANALYSES

Details of the planned displays including the population to be used for each display and which displays are produced for the strategic interim are presented in Appendix 11. Additional details are provided below.

The estimand is the effect of actual treatment in the population of participants who were randomized and dosed. All collected data will be included in reporting as described below. Non-recorded missing data following study withdrawal will not be imputed.

# 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of AEs, SAEs and other significant AEs will be based on GSK Core Data Standards.

# 8.2. Adverse Events of Special Interest Analyses

AESI have been defined as AEs which have specified areas of interest for the COPD population. A list of Standardized Medical Dictionary for Regulatory Activities (MedDRA) Queries (SMQs) and other groupings for AESI is provided in Section 14.6.4

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests and liver function tests will be based on GSK Core Data Standards.

# 8.4. Spirometry

The estimand is the effect of actual treatment in the population of participants who were randomised and dosed.

A frequentist MMRM analysis will be performed on spirometry data.

# 8.4.1. Endpoint

Change from baseline in post-BD FEV1

Change from baseline in post-BD FVC

# 8.4.2. Summary Measure

The summary measure is the adjusted mean difference from placebo for each danirixin dose.

#### 8.4.3. Population of Interest

mITT population.

#### 8.4.4. Strategy for Intercurrent (Post-Randomization) Events

The intercurrent event of interest is treatment discontinuation. A 'hypothetical' strategy will be used to account for this event. All recorded data up to the time of treatment discontinuation will be included in the analysis. Subsequent data up to Day 168 will be assumed to be missing at random (MAR).

#### 8.4.5. Statistical Analyses / Methods

# 8.4.5.1. Frequentist MMRM Methodology Specification

# **Endpoint / Variables**

- Change from baseline in post-BD FEV1
- Change from baseline in post-BD FVC

#### **Model Specification**

- The following covariates will be included in the model: baseline, country, smoking status at screening, treatment, Visit, Visit \*baseline and Visit \*treatment interactions, where Visit is nominal. Visit will consist of two levels (Day 84 and 168), and treatment will consist of six levels (placebo and 5 active doses)
- Two models will be fitted; one with a response variable (FEV1 or FVC), and one with a response variable of change from baseline (FEV1 or FVC).
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used. If this method does not run, the residual method will be used instead
- The OM option will be used to derive the least square (LS) means using coefficients which are based on the participants used in the analysis. The OM option requires an OM dataset which has a row for every participant-visit combination that contains all of the covariates used in the model and a macro variable containing the mean baseline for the participants used in the analysis.

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the model used for analyses using MMRM will be
examined by obtaining a normal probability plot of the residuals and a plot of the residuals
versus the fitted values (i.e. checking the normality assumption and constant variance
assumption of the model respectively) to gain confidence that the model assumptions are
reasonable. Plots of residuals versus covariates and baseline versus response will also be
examined.

#### **Model Results Presentation**

- LS mean and LS mean changes from baseline with their corresponding standard errors (SEs) for each visit and each treatment
- Estimated treatment differences from placebo and corresponding 90% confidence intervals (CIs) and p-values for each visit and each danirixin dose.
- A figure of LS mean changes from baseline and 90% CIs for each treatment by visit will be generated.
- The type III tests of fixed effects from the model will be presented.

#### **Summary Results Presentation**

- Summary statistics for baseline post-BD FEV1, FVC and FEV1/FVC for each treatment and
  overall for participants with non-missing assessments for each Visit, for the mITT population.
- Summary statistics for raw and change from baseline post-BD FEV1, FVC and FEV1/FVC for each visit for each treatment, for the mITT population.
- A figure of mean and 90% CIs for each treatment by visit (including baseline, Day 84 and Day 168) will be generated for post-BD FEV1, FVC and FEV1/FVC.

# 8.5. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified.

#### 9. PHARMACOKINETIC ANALYSES

# 9.1. Primary Pharmacokinetic Analyses

#### 9.1.1. Derived Pharmacokinetic Parameters

PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. PK parameters listed will be determined from the blood concentration-time (dry blood spot) data at Visit 3 and 10, as data permits for participants in the PK sub-set collecting PK samples at pre-dose, 0.5. 1. 2. 4. 6, 8, 10, 12 hours post-dose.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Tlast | Time of last quantifiable concentration |

#### NOTES:

Additional parameters may be included as required.

#### 9.1.2. Statistical Analyses / Methods

No formal statistical analysis of the dry blood spot PK concentrations or PK parameters will be performed. Details of the planned displays are provided in Appendix 11 and will be based on GSK Data Standards and statistical principles.

# 9.2. Exploratory Pharmacokinetic Analyses

#### 9.2.1. Derived Pharmacokinetic Parameters

Note: Approximately 20% of the wet whole blood samples collected at Visit 3 will be analysed for danirixin concentrations to provide an analytical comparison between dried blood spot and wet whole blood sample results. The expectation is that samples selected will mainly come from those samples provided by participants in the PK sub-set (i.e. collecting samples over 12 hours) and be distributed across danirixin treatment groups.

PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. PK parameters listed will be determined from the blood concentration-time (wet whole blood) data at Visit 3, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Tlast | Time of last quantifiable concentration |

#### NOTES:

Additional parameters may be included as required.

# 9.2.2. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11 and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 9.2.2.1. Statistical Methodology Specification

An extension of the Bland and Altman approach [Bland, 1986; Bland, 1999] will be used to quantify the agreement between the assay methods using log-transformed data, including hematocrit in the model. Age and weight will also be added one at a time in a model building approach and their significance in the model will be assessed. Limits of agreement and the coefficient of variation will be assessed to determine the agreement of the assay methods and whether wet whole blood assay is comparable to dry blood spot assay.

A sensitivity analysis will be performed excluding dry blood spot concentrations above the assay higher level of quantification of 1000 ng/mL.

#### **Endpoint / Variables**

 Log-transformed Danirixin blood concentration and pharmacokinetic parameter (Cmax and AUC(0-t)) data

#### **Model Specification**

- The Bland and Altman method will be used.
- The following covariates will be included in the model: haematocrit, age and weight.

#### **Model Results Presentation**

- Separate outputs will be produced for Danirixin concentration and pharmacokinetic parameters (although both will be analyzed using the same model)
- Estimates of intercept and slope on log-scale for Danirixin concentration and pharmacokinetic parameters, bias at concentration is 0, %CVw, geometric means and limit of agreement at concentration is 0.
- Comparative plots of individual blood concentration and pharmacokinetic parameter data.
- Supportive SAS output from statistical analysis.

#### **Sensitivity and Supportive Analyses**

 A sensitivity analysis excluding dry blood spot concentrations above the assay HLOQ of 1000 ng/mL will be performed.

#### 10. POPULATION PHARMACOKINETIC ANALYSES

PK data from this study may be combined with historic data for the purposes of population PK (PopPK) modelling which would be the subject of a separate analysis plan and would be presented separately from the main CSR.

To support this analysis a PopPK dataset will be generated. The details for the dataset specifications are provided in Appendix 9.

# 11. BIOMARKER ANALYSES

C-reactive protein and fibrinogen data will be summarized in the same way as laboratory data. Summary tables and boxplots for each treatment by visit (including screening, baseline, Day 84 and Day 168) will be generated for the mITT populations and also for the subset of subjects who have an event in the 'Infective pneumonia' SMQ.

Exploratory biomarker analysis will be the subject of a separate RAP.

# 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

Graphical assessment of the relationship between individual danirixin exposure and PD endpoints will be conducted.

Contingent on any PK/PD relationship(s) being identified from the graphical assessment a PK/PD dataset will be generated. The details for the methodology and dataset specifications will be provided in a separate document after review of the graphical assessment of the relationship between PK and PD endpoints.

# 12.1. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11 and will be based on GSK Data Standards and statistical principles.

# 13. REFERENCES

Atkinson, AC. (1985) Plots, Transformations and Regression. Clarendon Press.

Bland JM, Altman DG. (1986). Statistical methods for assessing agreement between two methods of clinical measurement. Lancet, i, 307-310

Bland JM, Altman DG. (1999). Measuring agreement in method comparison studies. Statistical Methods in Medical Research 1999; 8: 135-160.

Bornkamp, B. (2014). Practical considerations for using functional uniform prior distributions for dose-response estimation in clinical trials. Biometrical Journal, 947–962.

Chong J, Leung, B and Poole P. Phosphodiesterase 4 inhibitors for chronic obstructive pulmonary disease. Cochrane Database Syst. Rev. 2013; Issue 11

Crim C, Dransfield MT, Bourbeau J, et al. Pneumonia risk with inhaled fluticasone furoate and vilanterol compared with vilanterol alone in patients with COPD. Ann. Am. Thorac. Soc. 2015; 12(1): 27-34

Drummond MB, et al. Inhaled corticosteroids in patients with stable chronic obstructive pulmonary disease: a systemic review and meta-analysis. JAMA. 2008; 300(20): 2407 - 16

EMA press release. PRAC reviews known risk of pneumonia with inhaled corticosteroids for chronic obstructive pulmonary disease. 2016

Evidera (2016a) The Exacerbations of Chronic Pulmonary Disease Tool (EXACT) Patient-Reported Outcomes (PRO), User Manual (Version 8.0).

Evidera (2016b) Evaluating Respiratory Symptoms (E-RS<sup>™</sup>) in COPD (E-RS<sup>™</sup>: COPD), User Manual (Version 5.0)

IMI PROactive in COPD Daily and Clinical Instruments D-PPAC and C-PPAC User Guide (14JUN16)

Jones PW and Forde Y. (2016) St. Georges Respiratory Questionnaire for COPD Patients Manual, version 1.3

Spencer S, Karner C, Cates CJ, Evans DJ. Inhaled corticosteroids versus long-acting beta2-agonists for chronic obstructive pulmonary disease. Cochrane Database of Systematic Reviews 2011, Issue 12.

Spiegelhalter, D. J., Abrams, K. R., & Myles, J. P. (2004). Bayesian approaches to clinical trials and health-care evaluation. John Wiley & Sons.

# 14. APPENDICES

# 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 14.1.1. Exclusions from Per Protocol Population

A participant meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|---|---|
| 01 | Inclusion #2 – FEV1/FVC ratio >=0.70 or % predicted FEV1<40% at Screening |
| 02 | Inclusion #4 – <2 historical exacerbations or one historical exacerbation with screening fibrinogen <3 g/L |
| 03 | Inclusion #5 - Smoking history of <10 pack years at Screening |
| 04 | Exclusion #4 - Screening visit is less than 14 days since the completion of a course of antibiotics or oral steroids for a COPD exacerbation |
| 05 | Exclusion #14 - Use of PDE4 inhibitors within 30 days of Screening |
| 06 | Exclusion #26 - Oxygen use that is not PRN at Screening |

At the strategic interim a participant meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|---|---|
| 07 | Xanthines at any time between the day after screening and end of treatment |
| 08 | PDE4 inhibitors at any time between screening and end of treatment |
| 09 | Chronic use (more than 3 months) of erythromycin or azithromycin for between screening and end of treatment |
| 10 | Participants who stopped study medication for more than 14 days |
| 11 | Blind broken |

For the final analysis a participant meeting any of the following criteria will have data excluded from the time of the deviation. If a prohibited medication is taken prior to randomisation the participant will be excluded from the Per Protocol population.

| Number | Exclusion Description |
|---|---|
| 07 | Xanthines at any time between the day after screening and end of treatment |
| 08 | PDE4 inhibitors at any time between screening and end of treatment |
| 09 | Chronic use (more than 3 months) of erythromycin or azithromycin between screening and end of treatment |
| 10 | Participants who stopped study medication for more than 14 days will be excluded from the PP analyses from the time they stopped taking study medication. |
| 11 | Data excluded from date of breaking of blind. |

# 14.2. Appendix 2: Schedule of Activities

# 14.2.1. Protocol Defined Schedule of Events

| | | | | | | | Study V | isits | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre-<br>Screening <sup>a</sup><br>(Visit 0) | Screening <sup>a</sup> (Visit 1) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Early<br>Withdrawal | Follow Up |
| Study Day | | | -7 | 1 | 14 | 28 | 56 | 84 | 112 | 140 | 168 | | (up to 28 days post last dose) |
| Assessment Window | -30 | d | ±<br>0d | +<br>3d | ± 3d | ±<br>3d | ± 3d | ± 3d | ± 3d | ± 3d | ±<br>3d | | |
| Eligibility | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | |
| Genetic Sample<br>Informed Consent <sup>b</sup> | X | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | |
| COPD Exacerbation<br>History | X | | | | | | | | | | | | |
| Pre-Screening<br>Fibrinogenc | X | | | | | | | | | | | | |
| Smoking History <sup>d</sup> | | X | | | | | | | | | | | |
| Smoking Status <sup>d</sup> | | X | X | | | | | | | | | | |
| Inclusion and Exclusion criteria | | X | | | | | | | | | | | |
| Medical history <sup>e</sup> | | X | | | | | | | | | | | |
| Full physical examination including height and weight | | X | | | | | | | | | | | |

| | | | | | | S | Study V | isits | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre-<br>Screening <sup>a</sup><br>(Visit 0) | Screening <sup>a</sup> (Visit 1) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Early<br>Withdrawal | Follow Up |
| Study Day | | | -7 | 1 | 14 | 28 | 56 | 84 | 112 | 140 | 168 | | (up to 28 days post last dose) |
| Assessment Window | -30 | d | ±<br>0d | +<br>3d | ±<br>3d | ±<br>3d | ± 3d | ±<br>3d | ± 3d | ±<br>3d | ± 3d | | |
| Chest x-ray (CXR)f | | X | | | | | | | | | | | |
| HIV, Hepatitis B and C screening <sup>g</sup> | | X | | | | | | | | | | | |
| Pulse Oximetry | | X | | | | | | | | | | | |
| Additional Eligibility an | nd In Study Ass | essments | | | | | | | | | | | |
| Verify Eligibility <sup>h</sup> | | | X | X | | | | | | | | | |
| Brief Physical | | | | X | | | | X | | | X | X | X |
| Urine or serum pregnancy test <sup>i</sup> | | X | | X | | X | X | X | X | X | X | X | |
| Laboratory<br>assessments (clinical<br>chemistry (includes<br>liver chemistries),<br>hematology,<br>urinalysis) | | X | | X | | X | | | | | X | X | Х |
| Additional Liver chemistries only | | | | | X | | X | X | | | | | |
| 12-lead ECG | | X | | X | | X | | X | | | X | X | |
| Vital signs | X | X | | X | | X | | X | | | X | X | |
| Spirometry | | X | | X | | | | X | | | X | X | |
| Randomization | | | | X | | | | | | | | | |

| | | | | | | S | Study V | isits | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre-<br>Screening <sup>a</sup><br>(Visit 0) | Screening <sup>a</sup> (Visit 1) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Early<br>Withdrawal | Follow Up |
| Study Day | | | -7 | 1 | 14 | 28 | 56 | 84 | 112 | 140 | 168 | | (up to 28 days post last dose) |
| Assessment Window | -30 | d | ±<br>0d | +<br>3d | ±<br>3d | ±<br>3d | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | | |
| Dispense Study<br>Medication | | | | X | | X | X | X | X | X | | | |
| Dispense log pad and provide training | | | X | | | | | | | | | | |
| Dispense MDI sensors and provide training | | | X | | | | | | | | | | |
| Dispense physical activity monitor and provide training | | | X | | | | | | | | | | |
| Study treatment | | | | <del>(</del> = | | | | | | | ==> | | |
| Study treatment compliance (ediary) | | | | <b>←</b> = | | | | | | | <b>==</b> → | | |
| Collect IP | | | | | | <b>←==</b> | | | | | <del>-</del> | X | X |
| Collect MDI sensors | | | | | | | | | | | | X | X |
| Collect physical activity monitor | | | | | | | | | | | | X | X |
| Collect log pad | | | | | | | | | | | | X | X |
| Adverse Event (AE) review | | | | <del>-</del> = | | | | | | | == <del>→</del> | X | X |
| Serious Adverse<br>Event (SAE) review | <del></del> | | | | ==== | | | | | | <b>==→</b> | X | X |

| | | | | | | 5 | Study V | isits | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre-<br>Screening <sup>a</sup><br>(Visit 0) | Screening <sup>a</sup> (Visit 1) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Early<br>Withdrawal | Follow Up |
| Study Day | | | -7 | 1 | 14 | 28 | 56 | 84 | 112 | 140 | 168 | | (up to 28 days post last dose) |
| Assessment Window | -30 | d | ±<br>0d | +<br>3d | ± 3d | ± 3d | ± 3d | ±<br>3d | ± 3d | ±<br>3d | ± 3d | | |
| Concomitant medication review | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Clinical Outcomes Asse | essments | | | | | | | | | | | | |
| COPD Exacerbations | | | <del></del> | | | | | | | | ==> | X | X |
| EXACT-PRO <sup>j</sup> | | | <del></del> | | | | | | | | ==> | | |
| Rescue Medication<br>Use <sup>k</sup> | | | <del></del> | | | | | | | | <del>-</del> | | |
| SGRQ-C | | | | X | | | | X | | | X | X | |
| COPD Assessment<br>Test | | | | X | | | | X | | | X | X | |
| PROactive<br>Questionnaire <sup>1</sup> | | | | X | | | | X | | | X | | |
| Physical Activity<br>Monitor <sup>l</sup> | | | X | | | | | X | | | X | | |
| Participant Global<br>Impression of COPD<br>Severity | | | X | | | | | | | | | | |
| Participant Impression<br>of Change in COPD<br>Severity | | | | | X | X | X | X | X | X | X | X | |

| | | | | | | S | Study V | isits | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre-<br>Screening <sup>a</sup><br>(Visit 0) | Screening <sup>a</sup> (Visit 1) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Early<br>Withdrawal | Follow Up |
| Study Day | | | -7 | 1 | 14 | 28 | 56 | 84 | 112 | 140 | 168 | | (up to 28 days post last dose) |
| Assessment Window | -30 | d | ±<br>0d | +<br>3d | ±<br>3d | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | | |
| Participant Global<br>Impression of Activity<br>Limitation | | | X | | | | | | | | | | |
| Participant Impression of Change in Activity Limitation | | | | | X | X | X | X | X | X | X | X | |
| Genetic, Pharmacokine | rtic and Biomar | ker Blood Col | lections | ; | | | | | | | | | |
| Blood sample for<br>Genetics | | | | X | | | | | | | | | |
| Blood sample for pharmacokinetics (PK) <sup>m</sup> | | | | X | | | X | X | | | X | | |
| Blood sample for Fibrinogen | | | | X | | | | X | | | X | X | |
| Blood sample for CRP | | | | X | | | | X | | | X | X | |
| Blood Sample for<br>Exploratory<br>Biomarkers | | | | X | | | | X | | | X | X | |

| | | | | | | \$ | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre-<br>Screening <sup>a</sup><br>(Visit 0) | Screening <sup>a</sup> (Visit 1) | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Early<br>Withdrawal | Follow Up |
| Study Day | | | -7 | 1 | 14 | 28 | 56 | 84 | 112 | 140 | 168 | | (up to 28 days post last dose) |
| Assessment Window | -30 | d | ±<br>0d | +<br>3d | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | ± 3d | | |

- a. Pre-screening and screening visits may be completed on the same day.
- b. Agreeing to the genetic sample consent is not required for study participation.
- c. A pre-screening plasma fibringen measurement is only required for participants with 1 COPD exacerbation in the prior year.
- d. Smoking status /history assessed at screening: smoking status rechecked at Visit 2
- e. Includes substance usage, past and present medical conditions and family history of premature CV disease.
- f. See inclusion/exclusion criteria for CXR screening requirement
- g. Hepatitis B (HBsAg) and Hepatitis C (HepC antibody) testing is required. If testing otherwise performed within 3 months prior to the first dose of study treatment, testing at screening is not required. Hepatitis C RNA testing is optional; however a confirmatory negative Hepatitis C RNA test must be obtained, to be able to enrol participants with positive Hepatitis C antibody due to prior resolved disease.
- h. Participant's clinical status should be reviewed.
- i. Pregnancy testing only required for women of child bearing potential (WOCBP). A positive urine pregnancy test requires confirmation with a serum pregnancy test.
- j. E-RS: COPD is a subset of EXACT-PRO and is not a separate assessment.
- k. Rescue medication use will be assessed via e-diary and MDI sensor.
- 1. The Clinic Visit PROactive Physical Activity in COPD tool will be assessed in a subset of approximately 50% of study participants
- m. Pre-dose PK samples will be collected in all participants at Visits 3, 6, 7, and 10. In a subset of participants (approx. 50 participants at each dose level) at Visit 3, PK samples will be collected at pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12 hours post-dose. In a subset of participants (approx.. 50 participants at each dose level) at Visit 10, PK samples will be collected at pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12 hours post-dose.

# 14.3. Appendix 3: Assessment Windows

In general, data will be reported according to the nominal time of clinic visits and assessments as specified in the protocol. For example, if a participant recorded values for the Day 28 visit that were actually made on the 21st day of treatment, they will be presented as Day 28 values in the summary tables.

Participants that withdraw from the study at the time of a scheduled study visit will have data collected in the eCRF as part of the scheduled study visit. In order to collect all questionnaires that are scheduled to be performed at the Early Withdrawal (EW) Visit, eDiary data is reported as an EW Visit. If the date of the EW diary assessment is the same as the date of a scheduled visit date from the eCRF and there is no diary data present at the scheduled visit in question, the EW diary data will be listed, summarized and analysed as part of the scheduled visit (if the diary data was scheduled to be performed at the visit in question).

# 14.4. Appendix 4: Study Phases

# 14.4.1. Study Phases

Assessments and events collected outside scheduled study visits will be classified into study phases according to the time of occurrence relative to the start and/or stop date of study treatment. The 'worst case-post baseline' derivation for summaries will consider all scheduled and unscheduled measurements that have been assigned a treatment phase of 'On-treatment'.

#### 14.4.1.1. Study Phases for Diary Data

Diary data (including EXACT events) treatment states are specified in Section 14.6.3.

#### 14.4.1.2. Study Phases for Concomitant Medication

COPD medication combinations taken at screening will include all COPD medications that were taken on the day of the screening visit, excluding medications that stopped on the day of the screening visit.

Treatment phases for summaries of COPD and non-COPD concomitant medications will be assigned as follows:

| Study Phase | Definition |
|---|---|
| Prior | Medications taken on or before the day before treatment start date defined as: (conmed start date < treatment start date or 'Taken prior to study?' is 'Yes' or study treatment not started or conmed start date is missing) Note: prior concomitant medication data will only be summarized for COPD medications. All screening data will be listed. |
| On-treatment | If study treatment stop date > study treatment start date then this includes medications taken between the study treatment start date and study treatment stop date - 1 (inclusive) defined as follows: (conmed start date < study treatment stop date or conmed start date is missing) and (conmed stop date >= study treatment start date or (conmed stop date is completely missing and study treatment start date is non-missing)) If study treatment stop date = study treatment start date then this includes medications taken on the study treatment start date (which is equal to the study treatment stop date) defined as follows. (conmed start date <= study treatment stop date or conmed start date is missing) and (conmed stop date >= study treatment start date or (conmed stop date is completely missing and study treatment start date is non-missing)) |
| Post-treatment | If study treatment stop date > study treatment start date then this includes medications taken after the study treatment stop date defined as follows: (conmed stop date >= study treatment stop date or (conmed stop date is completely missing and study treatment stop date is non-missing)) If study treatment stop date = study treatment start date then this includes medications taken after the study treatment stop date + 1 defined as follows. (conmed stop date > study treatment stop date or (conmed stop date is completely missing and study treatment stop date is non-missing)) |

#### NOTES:

- A concomitant medication will be classed in every period of the study in which it was taken.
- See Section 14.7.2.1 for handling of partial dates.
- If the study treatment stop date is missing, it will be imputed as described in Section 14.6.1.

### 14.4.1.3. Study Phases for Event Data

Classification of a HCRU exacerbation/AE as having onset on-treatment will be made with reference to the study treatment start and stop dates and the event onset date. If the event onset date is missing, then the event will be considered on-treatment.

| Study Phase | Definition |
|---|---|
| Pre-treatment | If onset date is prior to treatment start date |
| | Start Date < Study Treatment Start Date |
| On-treatment | If onset date is on or after treatment start date & on or before treatment stop date + 3. |
| | Study Treatment Start Date ≤ Start Date ≤ Study Treatment Stop Date + 3 days |
| Post-treatment | If onset date is after treatment stop date + 3. |
| | Start Date > Study Treatment Stop Date + 3 days |

Note: assume on-treatment unless there is evidence to the contrary

#### 14.4.1.4. Study Phases for Other Data

All data collected at scheduled study visits after Day 1 will be considered on-treatment. Any data collected at unscheduled visits (ie, laboratory data, vital signs, ECGs, spirometry, CAT and SGRQ) will be classified as on-treatment based on the study treatment start date (and time, if available) and study treatment stop date and the date (and time, if available) of the visit/assessment. If the visit/assessment date is missing, then the event will be considered on-treatment.

| Study Phase | Definition |
|---|---|
| Pre-treatment | If assessment/visit date (and time) is on or prior to treatment start date (and time) |
| | Assessment/Visit Date (and time) ≤ Study Treatment Start Date (and time) |
| On-treatment | If assessment/visit date (and time) is after treatment start date (and time) & on or before treatment stop date + 3. Study Treatment Start Date (and time) < Assessment/Visit Date (and time) ≤ Study Treatment Stop Date + 3 days |
| Post-treatment | If assessment/visit date is after treatment stop date + 3. |
| 1 Ost-treatment | Assessment/Visit Date > Study Treatment Stop Date + 3 days |

Note: assume on-treatment unless there is evidence to the contrary

# 14.5. Appendix 5: Data Display Standards & Handling Conventions

# 14.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Compound | : GSK1325756 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to Legacy GSK A&amp;R dataset standards for the strategic<br/>interim and CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG Version 1.1].</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for strategic interim and final reporting efforts | |

# 14.5.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.24: General Principles
- 5.01 to 5.08: Principles Relating to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principle 4.24 for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - E-RS: COPD and SGRQ will have a min and max to 1 decimal places (dp) and then follow IDSL standards for reporting other summary statistics.
  - CAT will have a min and max to 0 dp and then follow IDSL standards for reporting other summary statistics.
- Categories will be based on rounded values to the precision collected on the eCRF, i.e., categories of % predicted FEV1 will be based on the rounded (to 1 dp) values of the variable FEV1PDPC
- Summaries of continuous data will include number of participants, mean, SD, median, minimum and maximum and for C-RP and fibrinogen outputs the 25th and 75th percentile.
- Percentages between 1% and 99%, inclusive, will be rounded to integers. Percentages greater than 0%, but less than 1%, will be reported as <1%, and percentages greater than 99%, but less than 100%, will be reported as >99%.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.

- Actual time will be used for calculation of times to events and Kaplan-Meier plots.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures except as part of a
  maximum/minimum/worst case post-baseline assessment or if they are assigned as the baseline
  assessment as detailed in Section 5.2.
- All unscheduled visits will be included in listings.

#### **Cardiovascular Event Reports**

 Laboratory results, ECG results/findings and vital signs measurements collected as part of cardiovascular event reports will not be included in any tables, listings or any minimum/maximum postbaseline assessments.

#### **Time to Event Results**

• For all time to event analyses, the first quartile and median time to event will be presented. If less than 25% of participants experienced the event within a treatment group then the first quartile will be displayed as NA (not applicable) for that treatment. If less than 50% of participants experienced the event within a treatment group then the median will be displayed as NA for that treatment.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |

#### **Graphical Displays**

• Refer to IDSL Statistical Principals 7.01 to 7.13.

#### **Seeds for Bayesian Analyses**

• The seeds used to for the Bayesian analyses were generated using the ranuni function in SAS. The same seeds should be applied for all endpoints and populations.

| Chain | Seed |
|-------|------|
| 1 | 2619 |
| 2 | 413 |
| 3 | 9243 |

# 14.5.3. Reporting Standards for Pharmacokinetic Data

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to GUI_51487 and PKOne documents. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. Additionally, include geometric mean and 90% CI for the summary of blood concentration data. |
| NONMEM/Pop PK<br>File | PopPK file (CSV format) for the PopPK analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Appendix 9. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | None |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | No. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

# 14.6. Appendix 6: Derived and Transformed Data

#### 14.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Potential Clinical Importance criteria at any postbaseline visit for safety parameters will be counted in both the High and Low categories of "Worst case post-baseline" row of related summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

# **Study Treatment Stop Date**

- If the study treatment stop date is missing, it will be imputed as follows:
  - If any of EW Visit date, Visit 10 (Day 168) date or date of death are non-missing then the study treatment stop date will be imputed as the minimum of (EW Visit date, Visit 10 (Day 168) date, date of death, date that all study treatment containers were returned).
  - For all other missing treatment stop dates, the last recorded exposure start or stop date will be used.
- For ongoing participants at the strategic interim, treatment stop date will be imputed as 5SEP2018

#### **Study Completion Definition**

 A participant is considered to have completed the study if they have not withdrawn and attended Visit 10.

# 14.6.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Age will be calculated based on the Pre-screening visit date.
- Age group categories are 18-64, 65-74, 75-84, >=85

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### **Baseline Characteristics**

#### % Predicted Normal FEV1 at Screening

• The following categories will be derived: <50%, >=50%

#### **Smoking Status**

- If the last smoked date (SUSMLSDT) is missing and a partial date (SUSMLSD) is not missing, then the following imputation should be applied to the partial smoking date for use in the reclassification of smoking status calculation:
  - '01' will be used for the day and 'Jan' will be used for the month.
- Former smokers will be reclassified as current smokers if screening date last smoked date < 183 days.

# **Chronic Mucus Hypersecretion**

- A participant is considered to have CMH (CMH+) if baseline SGRQ Q1(cough) = Most or several days a week AND baseline SGRQ Q2 (phlegm) = Most or several days a week.
- A participant is considered not to have CMH (CMH-) if baseline SGRQ Q1(cough) not equal to
  Most or several days a week OR baseline SGRQ Q2(phlegm) not equal to Most or several days a week
  and both questions are non-missing at baseline.
- Otherwise participants are considered to have a missing CMH status.

# **Baseline E-RS: COPD Total Score Categories**

- The following categories will be derived for baseline E-RS: COPD Total Score
  - o <8, >=8
  - o <10, >=10
    - <12, >=12

# **Exacerbation History Categories**

0

- Exacerbations (historical) will be classified as follows:
  - Mild: Managed without oral/systemic corticosteroids and/or antibiotics (not involving hospitalisation)
  - Moderate: Requiring oral/systemic corticosteroids and/or antibiotics (not involving hospitalisation)
  - Severe: Requiring hospitalisation
  - Moderate/severe: Requiring oral/systemic corticosteroids and/or antibiotics or hospitalisation.
- The total number of moderate/severe exacerbations will be categorized as ≤1, ≥2 for inclusion as a covariate in statistical models.

#### **GOLD Grade 1-4 at Screening**

- Participants will be classified into Global Initiative on Obstructive Lung Disease (GOLD) Grades
   1-4 using the post-bronchodilator percent predicted FEV1 assessment at Screening:
  - o GOLD Grade 1 (Mild): percent predicted FEV1 ≥80%
  - o GOLD Grade 2 (Moderate): 50%≤ percent predicted FEV1 <80%
  - o GOLD Grade 3 (Severe): 30%≤ percent predicted FEV1 <50%
    - GOLD Grade 4 (Very Severe): percent predicted FEV1 <30%

# ○ GOLD Grade A-D at Screening

- Participants will be classified into GOLD Grades A-D definitions as follows:
  - A. Low risk, less symptoms: baseline CAT < 10 AND GOLD Grade 1-2 AND  $\leq$ 1 exacerbation; (no hospitalizations for exacerbations), prior year.
  - B. Low risk, more symptoms: baseline CAT  $\geq$  10 AND GOLD Grade 1-2 AND  $\leq$ 1 exacerbation (no hospitalizations for exacerbations), prior year
  - C. High risk, less symptoms: baseline CAT < 10 AND either GOLD Grade 3-4 OR  $\geq$  2 exacerbations, prior year OR >=1 exacerbation leading to hospitalization, prior year
  - D. High risk, more symptoms: baseline CAT  $\geq$  10 AND either GOLD Grade 3-4 OR  $\geq$  2 exacerbations, prior year OR  $\geq$  1 exacerbation leading to hospitalization, prior year

#### **Baseline Characteristics**

#### **Participant Disposition**

- For Kaplan-Meier plots of study withdrawal over time, censoring will be performed as follows:
  - Participants are represented from their Day 1 date to the date of early withdrawal from the study (or date of death). Participants that completed the study are censored at the earliest of the date of completion and Day 168.

#### **Medical Conditions and Concomitant Medications**

#### **Respiratory Medication Class**

- COPD concomitant medications will be grouped into the following RMCs based on pre-defined code lists derived from ATC classifications:
  - Androgens and Estrogens
  - Anti-IgE, Anti-IL5
  - Anticholinergic
  - Antiinfectives (antibiotics, antiseptics only)
  - Antimycotics
  - Antivirals
  - Beta 2 Agonist
  - o Corticosteroid Inhaled
  - Corticosteroid Depot
  - O Corticosteroid Systemic, oral, parenteral and intra-articular
  - Corticosteroid Other
  - Leukotriene Receptor Antagonist
  - Long-acting anticholinergic
  - Long-acting beta-2 agonist
  - Mucolytics
  - Nedocromil or Cromolyn Sodium
  - Oxygen
  - PDE4 Inhibitors
  - Short-acting anticholinergic
  - Short-acting beta-2 agonist
  - Xanthine
  - Other medication given for exacerbation
  - Other COPD medication

#### **COPD Medication Combination**

- COPD medications will be summarized at the following time points:
  - At Screening: Taken on the day of the Screening visit excluding medications that stopped on the day of the Screening visit
  - O At Baseline: Taken on the day of start of treatment
  - At Month 6: Taken during Month 6 (Study Day 141 to earliest of (Study day 168 and day before study treatment stop date))
- Medication combinations of all RMC categories will be derived. Medications will be summarized based on individual and combinations of the following RMC categories, with or without other medications:
  - o ICS
  - o LABA
  - o LAMA
  - Xanthine
  - PDE4 inhibitor
  - Anti-IgE, Anti-IL5

#### **Medical Conditions and Concomitant Medications**

#### **Cardiovascular Risk Factors**

- Subjects with at least one of the following current or past medical conditions at Screening will be classed
  as having cardiovascular (CV) risk factor at screening. The number of CV risk factors at Screening (0, 1,
  or >=2) will be derived.
  - Coronary artery disease
  - Myocardial infarction
  - Arrithymia
  - Congestive heart failure
  - Hypertension
  - Cerebrovascular accident
  - Hypercholesterolemia
  - Diabetes mellitus

#### Compliance

#### **Treatment Compliance**

Compliance= (tablets issued-tablets returned) x 100 / 2 x (treatment stop date – treatment start date +1)

If any count of tablets returned is missing overall compliance will be set to missing.

- Compliance will be categorized as follows:
  - < 80 %
  - $\geq 80$  % to < 95 %
  - $\geq$  95 % to  $\leq$ 105 %
  - >105 % to ≤120 %
  - >120 %
- If a participant received a treatment other than the randomized treatment during the study, the compliance will still be calculated using data from all containers received and overall treatment start and stop dates.

#### **Daily Diary Compliance**

Overall compliance= (number of days with non-missing data between study treatment start and the earliest of (Study day 168 and day before study treatment stop)) x 100 / (Earliest of (Study day 168 and day before study treatment stop date) – treatment start date +1)

- Overall compliance will be categorized as follows:
  - < 50 %
  - $\geq$  50 % to < 60 %
  - $\geq$  60 % to < 70 %
  - $\geq$  70 % to < 80 %
  - $\geq$  80 % to < 90 %
  - $\geq$  90 % to  $\leq$ 100 %

Baseline and Monthly compliance= number of days with non-missing data between periods defined in Section 14.6.3

- Baseline compliance will be categorized as follows: Number of days completed <4, ≥4</li>
- Monthly compliance will be categorized as follows: Number of days completed <10, 10-20, >20

#### **Exposure**

#### **Exposure to Study Treatment**

Duration of exposure to study treatment is calculated as (treatment stop date – treatment start date +1).

The following exposure categories will be derived:

≥1 day, ≥4 weeks, ≥8 weeks, ≥12 weeks, ≥16 weeks, ≥20 weeks and ≥24 weeks. An additional category of 23-25 weeks will also be summarized.

## 14.6.3. **Efficacy**

#### Daily eDiary endpoints

#### General

Participants were instructed to complete the daily eDiary in the evening (typically at bedtime). The parameters collected include rescue use and EXACT-PRO scores.

The tables below show which daily eDiary records are used to calculate the daily eDiary parameters for each period. Any diary data collected after the minimum of (Day 168 and the day before study treatment stop date) will not be slotted.

To be used for rescue use endpoints and E-RS: COPD total and subscale scores:

| Period | First day | Last day |
|---|---|---|
| Baseline <sup>[1]</sup> | Latest of (7 days before Study | Day before Day 1 of study |
| | treatment start date (Day 1) and | treatment |
| | day of Visit 1 (Screening)) | |
| Month 1 <sup>[1]</sup> | Study day 1 | Study day 28 |
| Month 2 <sup>[1]</sup> | Study day 29 | Study day 56 |
| Month 3 <sup>[1]</sup> | Study day 57 | Study day 84 |
| Month 4 <sup>[1]</sup> | Study day 85 | Study day 112 |
| Month 5 <sup>[1]</sup> | Study day 113 | Study day 140 |
| Month 6 <sup>[1]</sup> | Study day 141 | Earliest of (Study day 168 and day |
| | | before study treatment stop date) |

[1] The denominator for baseline and monthly mean scores is the number of days with a non-missing score; this is also used to determine whether or not a baseline (>=4 days) or monthly mean (>=10 days) is calculated.

#### **EXACT PRO**

- The EXACT-PRO (Evidera, 2016a) is a 14-item daily diary (typically completed at bedtime)
- The daily E-RS: COPD total score (and subscales) will be computed according to the E-RS in COPD user manual (Evidera, 2016b).
- The monthly mean for E-RS: COPD total score, and the subscale scores RS-Breathlessness, RS-Cough and Sputum, and RS-Chest Symptoms will be calculated as the mean of the daily scores in the monthly intervals defined above.
- Mean monthly score = (sum of daily scores/# diary days completed).
- A participant must have at least 10 days of diary data in any month to contribute a non-missing monthly mean of daily values; otherwise the monthly mean for that month will be considered missing.
- A participant must have at least 4 days of diary data in the 7 days prior to treatment start date to contribute a non-missing mean of daily values for baseline; otherwise baseline will be considered missing.
- If missing values occur for individual items, the E-RS: COPD total score and E-RS: COPD subscale

#### Daily eDiary endpoints

score that contain the item will be set to missing on that day.

#### Responders according to E-RS: COPD Total and Subscale Scores

- A participant will be considered as a responder according to E-RS: COPD total score if their monthly mean change from baseline E-RS: COPD total score ≤ -2.0.
- A participant will be considered as a non-responder according to E-RS: COPD total score if their monthly mean change from baseline E-RS: COPD total score >-2.0.
- A participant will be considered as a responder according to E=RS: COPD breathlessness score if their month mean change from baseline E-RS: COPD breathlessness score ≤ -1.0.
- A participant will be considered as a non-responder according to E-RS: COPD breathlessness score if their monthly mean change from baseline E-RS: COPD breathlessness score >-1.0.
- A participant will be considered as a responder according to E-RS: COPD cough & sputum score if their monthly mean change from baseline E-RS: COPD cough & sputum score ≤ -0.70.
- A participant will be considered as a non-responder according to E-RS: COPD cough & sputum score if their monthly mean change from baseline E-RS: COPD cough & sputum score >-0.70.
- A participant will be considered as a responder according to E-RS: COPD chest symptoms score if their monthly mean change from baseline E-RS: COPD chest symptoms score ≤ -0.70.
- A participant will be considered as a non-responder according to E-RS: COPD chest symptoms score if their monthly mean change from baseline E-RS: COPD chest symptoms score >-0.70.
- If the monthly mean E-RS: COPD score is missing then response status will be missing.

#### Season

- For each participant and each month, season will be assigned based on the first date with a non-missing daily score in the monthly mean E-RS: COPD total score.
- Australia will add 6 months to the first day of the monthly mean E-RS: COPD total score before season is assigned.
- If the month of the first day of the monthly mean score period is:
  - Dec, Jan or Feb then season is Winter
  - Mar, Apr or May then season is Spring
  - Jun, Jul or Aug then season is Summer
  - Sep. Oct or Nov then season is Fall

#### Mean Number of Rescue Puffs per Day and Percentage Rescue Free Days

- If a participant has more than one daily diary record for any given day, the worst case response on that
  day for each endpoint will be used in the summaries and analyses. i.e. the maximum number of puffs of
  rescue use reported will be counted for the day in question and used to determine if it was a recue-free
  day.
- A rescue-free day is defined as a day where the total puffs is 0.
- For each summary period, the mean number of puffs per day and the percentage of rescue free days, will be calculated, using the number of days with non-missing values for the endpoint as denominator.
- Rescue use will be summarized over the periods defined above.

#### **HCRU Exacerbations**

#### Duration

 The duration of the exacerbation will be calculated as (exacerbation resolution date or date of death exacerbation onset date + 1).

#### Severity

- Each HCRU exacerbation will be categorized based on severity as follows:
  - Mild: no treatment with oral/systemic corticosteroids and/or antibiotics and not involving hospitalisation, an emergency room visit or resulting in death
  - Moderate: required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalisation, an emergency room visit or resulting in death).
  - O Severe: required in-patient hospitalization, an emergency room visit, or resulted in death

#### Time to First Exacerbation

- The time to first on-treatment Moderate/Severe HCRU exacerbation will be calculated as exacerbation onset date of first on-treatment moderate or severe on-treatment exacerbation – date of start of treatment +1
- Participants will be represented from their treatment start date to their first on-treatment moderate or severe exacerbation or date of censoring.
- For the strategic interim analysis, participants that have not experienced an on-treatment exacerbation are censored at the earliest of (treatment stop date + 3, date of death, or the interim cut-off date, 1AUG2018).
- For the final analysis, participants that have not experienced an on-treatment exacerbation are censored at the earliest of (treatment stop date + 3, date of death, date of exclusion from the per protocol population (if analysis is in Per Protocol population))

#### **Raw Annual Rate**

• Raw annual rate is the event rate per 1000 participant-years, calculated as the number of events x 1000, divided by the total duration at risk (minimum(treatment stop date + 1, date of death, date of exclusion from the per protocol population (if analysis is in Per Protocol population)) – treatment start date + 1).

#### Offset Variable

• For analyses of exacerbation rate, the offset variable will be defined as the logarithm of the ((minimum (date of end of study treatment + 3, date of death, date of exclusion from the per protocol population (if analysis is in Per Protocol population)) – date of start of treatment + 1)/365.25)

#### **EXACT Events**

#### General

- The daily EXACT-PRO scores will be computed according to the EXACT-PRO user manual (Evidera, 2016a) and used to identify EXACT-defined events, including the frequency, duration and severity of the events.
- Events will be categorized as recovered, censored, or persistent worsening (according to the manual).

#### Time to First Event

- The time to first on-treatment EXACT event will be calculated as the onset date of the first on-treatment EXACT event – date of start of treatment +1
- Participants will be represented from their treatment start date to their first EXACT event or date of censoring.
- For the final analysis, participants that have not experienced an EXACT event are censored at the
  earliest of (Day 168, treatment stop date 1, date of death, or date of final EXACT-PRO assessment,
  date of exclusion from the per protocol population (if analysis is in Per Protocol population))

#### **Raw Annual Rate**

Raw annual rate is the event rate per 1000 participant-years, calculated as the total number of EXACT-defined events x 1000, divided by the total duration at risk (minimum(Day 168, treatment stop date - 1, date of death, date of final EXACT-PRO assessment, date of exclusion from the per protocol population (if analysis is in Per Protocol population)) – treatment start date + 1).

#### Offset Variable

For analyses of EXACT event rate, the offset variable will be defined as the logarithm of the ((minimum (Day 168, treatment stop date - 1, date of death, date of final EXACT-PRO assessment, date of exclusion from the per protocol population (if analysis is in Per Protocol population)) – date of start of treatment + 1)/365.25)

#### CAT

#### **CAT Score**

- The CAT consists of eight items each formatted as a six-point differential scale: 0 (no impact) to 5 (high impact). A CAT score will be calculated by summing the non-missing scores on the eight items. The score can have values ranging from 0 to 40.
- If one item is missing, then the score for that item is set as the average of the non-missing items. If more than one item is missing, then the CAT score will be set to missing.
- If the language of the CAT conducted at a post-baseline visit is different to the language used at baseline, the CAT score for that visit and all subsequent visits will be set to missing.
- If there is more than one response to a question at a visit or duplicate questionnaires, the CAT score for that visit will be set to missing.

#### Responders according to CAT Score

- A participant will be considered as a responder according to CAT score if their change from baseline CAT score ≤ -2.0.
- A participant will be considered as a non-responder according to CAT score if their change from baseline CAT score >-2.0.
- If CAT score is missing at a visit, the response status will be missing at that visit.

#### Season

- For each participant and each visit, season will be assigned based on visit date.
- Australia will add 6 months to the visit date before season is assigned.
- If the month of the visit is:
  - Dec. Jan or Feb then season is Winter
  - Mar, Apr or May then season is Spring
  - Jun, Jul or Aug then season is Summer
  - Sep, Oct or Nov then season is Fall

#### **SGRQ**

#### **SGRQ Domain and Total Scores**

- The SGRQ-C contains 14 questions with a total of 40 items grouped into three domains (Symptoms, Activity and Impacts).
- Details for how to score the SGRQ-C, including handling of missing data or multiple responses to questions, are outlined in the SGRQ-C manual (Jones, 2016).
- SGRQ-C domains and total scores will be converted to SGRQ scores as described in the manual.
- Changes from baseline in domain and total score will be calculated for the converted scores.
- If the language of the SGRQ-C conducted at a post-baseline visit is different to the language used at baseline, all SGRQ scores at that visit and all subsequent visits will be set to missing.

#### Responders according to SGRQ Total Score

- A participant will be considered as a responder according to SGRQ total score if their change from baseline SGRQ total score ≤ -4.0.
- A participant will be considered as a non-responder according to SGRQ total score if their change from baseline SGRQ total score >-4.0.
- If SGRQ total score is missing at a visit, the response status will be missing at that visit.
- Change from baseline SGRQ total score will be rounded to 1dp prior to assigning responder status.

#### Rescue Use via Sensor

#### Mean Number of Occasions and Percentage Rescue Free Days via Sensor

- The mean number of occasions of rescue per day and the percentage of rescue-free days will be calculated over the same time periods and using the same assumptions as rescue use via diary.
- Rescue-free Days days within the diary data collection period with no recorded rescue inhaler usage by the sensor will be assigned a rescue inhaler usage of 0.

#### **PROactive**

#### General

- A PROactive Total Score and two domain scores (amount and difficulty) are derived using data from the C-PPAC questionnaire and a physical activity monitor worn for 7 days prior to the questionnaire.
- To derive the PROactive score at each visit the following is required:
  - Response to valid (i.e., no missing items) C-PPAC questionnaire
  - Median values of steps/day and VMU/min on at least 3 days of the 7 days prior to the C-PPAC questionnaire with >=8 hours wearing (the 3 days do not need to be consecutive).
- The C-PPAC questionnaire contains 14 items (12 questions and 2 scores from the activity monitor outputs) each scored from 0 to 4.
- The amount domain is calculated using 2 items from the C-PPAC questionnaire (amount of walking outside and chores outside) and 2 activity monitor outputs (vector magnitude units per minute (VMU/min) and steps/day).
- The difficulty domain is calculated using 10 items from the C-PPAC guestionnaire.
- Each domain score is based on the addition of items (0-15 for amount and 0-40 for difficulty) and then scaled from 0-100.
- The total score is calculated as (amount+difficulty)/2
- Further details for how to score and scale the domain and total scores are outlined in the IMI PROactive user guide (14JUN16).

#### 14.6.4. Safety

#### **Adverse Events**

# **AEs of Special Interest**

- AESI are defined as events in the 'Infective pneumonia' SMQ in the MedDRA version current at the time of reporting.
- Subjects receiving ICS (RMC Corticosteroid Inhaled) for at least 7 days at the time of Pneumonia onset.

| Maximum/Minimum Post-Baseline and Worst-Case Post-Baseline | |
|---|---|
| Definition | Reporting Details |
| Maximum post-baseline<br>(QTcF, QTc B, PR interval, ECG<br>heart rate, pulse rate, systolic BP,<br>diastolic BP and laboratory tests) | Change from baseline of maximum value over all time-points after Day 1 |
| Minimum post-baseline (Diastolic BP and laboratory tests that do not have a lower limit = 0) | Change from baseline of minimum value over all time-points after Day 1 |
| Worst case post-baseline (ECG findings) | <ul> <li>'Abnormal' if any on-treatment assessment is evaluated as 'Abnormal'</li> <li>'Unable to evaluate' if all on-treatment assessments are 'Unable to evaluate'</li> <li>'Normal' if any on-treatment assessment is evaluated as 'Normal' and there are no on-treatment assessments evaluated as 'Abnormal'</li> </ul> |

#### NOTES:

- The treatment phase definitions specified in Section 14.4.1.4 will be used and only assessments within the ontreatment period will be considered in assessment of minimum/maximum/worst-case post-baseline.
- Assessment of minimum/maximum/worst-case post-baseline will include on-treatment data from scheduled, unscheduled and study treatment discontinuation visits (if applicable)

#### **Laboratory Parameters**

#### General

- NQ laboratory results will be treated as missing in summary displays. However, the results will be listed as received (e.g. '<x' or '>x').
- If numeric laboratory results are missing but a character result has been recorded, ie. <X, (the numeric part of the character value)/2 will be used to assign the PCI ranges.
- A 'worst case post-baseline' change classification will be derived, in which participants will be counted in
  the 'to low' and 'to high' categories if they reported a change from an 'in range' baseline to a value
  below or above the PCI criteria (respectively) at any scheduled or unscheduled on-treatment visit.
  Participants who did not report a change to a value outside the PCI criteria at any visit after the start of
  study treatment will be counted in the 'to w/in range or no change' category.

#### Multiple Measurements for On-Treatment Visits for Safety

Participants having both high and low values relative to PCI criteria at post-baseline visits for safety
parameters will be counted in both the high and low categories of the "worst case post-baseline" row of
related summary tables.

#### **ECG**

#### General

- The QTc data was collected via machine derived values (QTCB/QTCF) or manually derived values (QTCBC/QTCFC). For the purposes of reporting the following variable should be combined:
  - Combine QTCF with QTCFC
- If both QTCF and QTCFC are missing (and QT and RR are non-missing then the QTcF interval will be derived as follows:
  - QTcF interval (msec) = QT/[(RR/1000)\*\*(1/3)]
  - If RR interval is not collected and the corrected QT interval by Bazett's method (QTcB) is collected, then RR interval (msec) will be derived prior to deriving QTcF as follows: RR interval (msec) = 1000\*[(QT/QTcB)\*\*2]
- If QTcF intervals are collected they will not be rederived.

### **ECG Categories**

Maximum and maximum increase in d QTcF values will be reported in categories as below. In subjects who have QTc above 450 at baseline, decreases that result in a QTc that remains above 450 will be considered No Change.

| ECG Parameter | Units | Category |
|---------------------------|-------|--------------------------------|
| Absolute | | |
| | msec | No Change or Decrease to <=450 |
| Abaduta OTaF Intarval | | Increase To >450 to <=480 |
| Absolute QTcF Interval | | Increase To >480 to <=500 |
| | | Increase To >500 |
| Change from Baseline | | |
| | | Increase of <=30 ms |
| Change from Baseline QTcF | msec | Increase of 31-60 msec |
| | | Increase of >60 msec |

Assessment of maximum post-baseline will include on-treatment data from scheduled, unscheduled and study treatment discontinuation visits (if applicable)

# 14.7. Appendix 7: Reporting Standards for Missing Data

# 14.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as<br/>completion of all phases of the study including the last study visit and the last<br/>scheduled procedure shown in the Schedule of Activities (Appendix 2).</li> </ul> |
| | • For the purposes of reporting, a participant is considered to have completed the study if they have not withdrawn and attended Visit 10. |
| | Withdrawn participants were not replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Data from the Early Withdrawal visit will not be included in any summaries or analyses except as part of a worst case post-baseline assessment. |

# 14.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | If outliers are identified, analyses may be repeated excluding the outlying data. |
| | Any participants/data excluded from summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 14.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied.</li> <li>Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 14.8. Appendix 8: Values of Potential Clinical Importance

# 14.8.1. Laboratory Values

The following table identifies a range of potential clinical importance (PCI) for each laboratory analyte. Limits with an 'x' are multipliers of the central laboratory normal range. Values above and below this range will be considered of PCI.

| Hematology Analyte (units) | Effect | COPD Patients | |
|---------------------------------|---------|---------------|-------|
| | | Low | High |
| Platelet Count (x109/L) | | 0.90x | 1.10x |
| Red Blood Cell Count (x1012/L) | | 0.93x | 1.07x |
| White Blood Cell Count (x109/L) | | 0.70x | 1.60x |
| Reticulocyte Count (%) | | | >4% |
| Homoglobin (g/L) | Males | 0.85x | 1.20x |
| Hemoglobin (g/L) | Females | 0.85x | 1.20x |
| Homotocrit (Datio of 1) | Males | 0.50x | 1.30x |
| Hematocrit (Ratio of 1) | Females | 0.50x | 1.30x |
| MCV (fL) | | 0.25x | 2.00x |
| MCH (pg) | | 0.85x | 1.20x |
| MCHC (g/dL) | | 0.85x | 1.10x |
| Neutrophils (%) | | 0.65x | 1.50x |
| Lymphocytes (%) | | 0.80x | 1.20x |
| Monocytes (%) | | 0.80x | 1.60x |
| Eosinophils (%) | | | 2.00x |
| Basophils (%) | | | 5.00x |

Note: Multipliers are identified by "x", otherwise actual comparison values are provided with units.

| Chemistry Analyte | Effect | COPD | COPD Patients |
|---|---|---|---|
| | | Low | High |
| BUN (mmol/L) | | 0.70x | 1.60x |
| | | | 1.30x |
| Creatinine (μmol/L) | | | (or >27 μmol/L increase from baseline) |
| Glucose fasting (mmol/L) | | <0.6x | >4x |
| Sodium (mmol/L) | | 0.80x | 1.15x |
| Potassium (mmol/L) | | 0.75x | 1.30x |
| Chloride (mmol/L) | | 0.90x | 1.10x |
| Bicarbonate (mmol/L) | | <18 mmol/L | >32 mmol/L |
| Calcium (mmol/L) | | 0.85x | 1.08x |
| GGT (U/L) | | 0.85x | 1.10x |
| Livia A aid (man/dl.) | Males | <2.1 mg/dL | >8.5 mg/dL |
| Uric Acid (mg/dL) | Females | <2.0 mg/dL | >7.0 mg/dL |
| Albumin (mmol/L) | | 0.90x | 1.50x |
| Total Protein (mg/dL) | | | 1.25x |

Note: Multipliers are identified by "x", otherwise actual comparison values are provided with units.

| Liver Function Test Analyte | Effect | PCI Range | Unit |
|-----------------------------|--------|---------------------------|--------|
| ALT/SGPT | High | ≥ 3x ULN | U/L |
| AST/SGOT | High | ≥ 3x ULN | U/L |
| Alkaline Phosphatase | High | ≥ 2x ULN | U/L |
| Total Bilirubin | High | ≥ 2x ULN | μmol/L |
| Direct Bilirubin | High | ≥ 2x ULN | μmol/L |
| | | ≥ 2x ULN Total Billirubin | μmol/L |
| Total Bilirubin + ALT | High | + | |
| | | ≥ 3x ULN ALT | U/L |

# 14.8.2. ECG

| ECG Parameter | PCI Range | Unit |
|------------------------------------|---------------|------|
| Absolute QTc Interval (QTcB, QTcF) | >530 | msec |
| Increase from Baseline QTc | >60 | msec |
| QT Interval | <300 or >500 | msec |
| PR Interval | <120 or >240 | msec |
| QRS Interval | <70 or >125 | msec |
| RR Interval | <375 or >1714 | msec |
| Heart Rate | <35 or >120 | bpm |

# 14.8.3. Vital Signs

| Vital Sign Parameter | PCI Range | Unit |
|----------------------|-------------|-----------------|
| Systolic BP | <90 or >160 | mmHg |
| Diastolic BP | <40 or >110 | mmHg |
| Heart Rate | <35 or >120 | bpm |
| Respiration Rate | <8 or >30 | breaths<br>/min |

# 14.9. Appendix 9: Population Pharmacokinetic Analyses

# 14.9.1. Population Pharmacokinetic Dataset Specification

#### 14.9.1.1. Handling Missing Demographic and Covariate Data

Missing demographic and covariate data will not be imputed.

# 14.9.1.2. Handling Missing Dose Times

Missing dose time information will be handled on a case by case basis by imputing this information based on prior dosing times or based on recorded PK collection times. The details of these imputations will be described in the report.

#### 14.9.1.3. Handling Missing Times of PK Samples

Missing times for PK will be handled on a case by case basis by imputing this information based on the dose time and/or times of other PK. The details of these imputations will be described in the report.

# 14.9.1.4. Handling of PK Data Below the Lower Limit of Quantification

Any PK data below the lower limit of quantification will be set to missing.

#### 14.9.1.5. Dataset Specification

General description and rules:

- Missing or unknown values in covariates, if not to be imputed, will be assigned -99.
- The dataset is sorted by STUD, SUBJID, DATE, RTFD, EVID descending.
- The data items (columns) in the analysis-ready data file will be provided in the same order as follows.
- NQ concentration values will be included as detailed for the CONC variable.
- Non-numerical concentration values (such as NS, NR, NA) will not be included.
- Placebo participants will not be included.
- The dataset will be a comma delimited ASCII text file and will be named:
  - o NM.compound.study.PK.v1.csv
  - o Where "compound" is the compound name (e.g. GSK1234567) and "study" is the study number (e.g. 205724).
| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing<br>value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| ID | NONMEM participant identifier | Integer | None | Never | Sequential participant identifier across study after data is sorted by STUD, SUBJID, DATE, RTFD, EVID. Numbering to start at 1. To be entered in all rows for each participant. |
| STUDYID | Unique identifier for a study | Char | None | Never | 205724 for all records |
| STUD | Study ID | Num | None | Never | 205724 for all records |
| SUBJID | Participant identifier for study | Num | None | Never | Participant identifier, which must be unique within the study. The identification number of the participant as recorded on the CRF. Exclude placebo participants. Include participants who have received IP and have at least one measurable drug concentration. To be entered in all rows for each participant. |
| COUNTRY | Country | Char | None | Never | Country of the investigational site in which the participant participated in the trial; e.g. USA. To be entered in all rows for each participant. |
| SITEID | Unique identifier for a study site | Char | None | Never | e.g. PPD any lead zero should not be included. To be entered in all rows for each participant. |
| CONC | Drug<br>Concentration | Num | ng/mL | Never | CONC=0 for DOSE_GSK1325756 records. No sample (NS), insufficient sample (IS) and no result (NR) records will be excluded from dataset. CONC='.' for PK_GSK1325756 records < LOQ (i.e. if drug conc is NQ). |
| LNCONC | Natural log of CONC column | Num | ng/mL | Never | Natural log of CONC column. If CONC=0, then LNCONC='.'. |
| LLQ | Lower Limit of quantification | Num | ng/mL | Never | LLQ=5 or from source data if different. To be entered in all rows for each participant. |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing<br>value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| LNLLQ | Natural log of LLQ column | Num | ng/mL | Never | Natural log of LLQ column. If LLQ=0, then LNLLQ='.'. |
| MATRIX | Sample matrix | Num | None | Never | MATRIX=1 (blood). |
| MATRTEXT | Sample matrix text | Char | None | Never | Text corresponding to code for MATRIX. Enter 'Blood' for all rows. |
| LABL | Label describing the record | Char | None | Never | LABL explains the type of measurement for CONC for the current record. LABL=DOSE_GSK1325756 for dose record. LABL=PK_GSK1325756 for blood concentration record. |
| DATE | Date of<br>Record | MM/DD/YYYY | None | Never | Date of record. |
| DATETIME | Date and time of record | MM/DD/YYYY<br>HH:MM:SS | None | Never | Date and time of record. |
| DAY | Study day<br>number of<br>record | Num | None | Never | Day of study relative to first IP dose. |
| NDAY | Nominal day | Num | day | Never | Schedule visit day of study relative to first IP dose. |
| NOMT | Nominal time<br>since FIRST<br>IP dose | Num | h | Never | Nominal time of study relative to first IP dose. NOMT=0 for first dosing record only. |
| NOMTLD | Nominal time since latest IP dose | Num | h | Never | Nominal time of study relative to last IP dose prior to sample. NOMTLD=0 for dosing records. |
| RTFD | Relative time<br>from FIRST IP<br>dose | Num | h | Never | Actual time from FIRST dose of IP. |
| RTLD | Relative time<br>from latest IP<br>dose | Num | h | Never | Actual time from last dose of IP prior to sample. When LABL=DOSE_GSK1325756, RTLD=0. For pre-dose PK sample Visit 6, 7 and 10, RTLD is relative to the previous dose. |
| DOSE | Dose amount | Num | mg | Never | DOSE=5, 10, 25, 35 or 50 per treatment administered. To be entered in all rows for each participant. |
| DRUG | Name of drug | Char | None | Never | DRUG=GSK1325756. To be entered in all rows for each participant. |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| REG | Dosing<br>Regimen | Integer | None | Never | REG=2 for BD. To be entered in all rows for each participant. |
| REGTEXT | Participant<br>dose regimen<br>text | Char | None | Never | REGTXT=BD, text corresponding to code for REG. To be entered in all rows for each participant. |
| ROUT | Route of administration | Integer | None | Never | ROUT=1 for PO. To be entered in all rows for each participant. |
| ROUTTEXT | Participant route of administration text | Char | None | Never | ROUTTEXT=PO, text corresponding to code for ROUT. To be entered in all rows for each participant. |
| CNC | NONMEM<br>Country code | Integer | None | Never | Australia, Canada, Germany,<br>Korea, Netherlands, Poland,<br>Romania, Spain, US.<br>Assign integer as appropriate for<br>each country. Eg. 1=US<br>To be entered in all rows for each<br>participant. |
| CMT | NONMEM<br>Compartment<br>code | Integer | None | Never | CMT=1 for DOSE_GSK1325756 records. CMT=2 for PK_GSK1325756 records. |
| EVID | NONMEM<br>Event ID | Integer | None | Never | EVID=1 for LABL=<br>DOSE_GSK1325756.<br>EVID=0 for LABL=<br>PK_GSK1325756. |
| AMT | NONMEM<br>Amount of<br>drug<br>administered | Num | mg | Never | AMT=0 for LABL= PK_GSK1325756 records. AMT=5, 10, 25, 35 or 50 (ass appropriate) for LABL= DOSE_GSK1325756 records. |
| II | NONMEM<br>Inter-dose<br>interval | Integer | h | Never | II=0 for LABL= PK_GSK1325756. II=12 for LABL= DOSE_GSK1325756, except II=0 for LABL= DOSE_GSK1325756 on Day 1 only. |
| SS | Steady-state<br>data item | Integer | None | Never | SS=0 for LABL= PK_GSK1325756 records. SS=1 for LABL= DOSE_GSK1325756 records, except SS=0 for LABL= DOSE_GSK1325756 records on Day 1 only. |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing<br>value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| RATE | NONMEM<br>Rate of drug<br>infusion | Integer | None | Never | RATE=0 for LABL= PK_GSK1325756 records. RATE=-2 for LABL= DOSE_GSK1325756 records. |
| MDV | NONMEM<br>Missing data<br>value | Integer | None | Never | MDV=1 for LABL= DOSE_GSK1325756 records. MDV=0 for LABL= PK_GSK1325756 records. MDV=1 for LABL= PK_GSK1325756 records < LOQ (NQ). |
| VIS | Visit number | Integer | None | Never | From source data. |
| POP | Population | Integer | None | Never | POP=1, for COPD. To be entered in all rows for each participant. |
| POPTEXT | Participant population text | Char | None | Never | POPTEXT=COPD, text corresponding to code for POP. To be entered in all rows for each participant. |
| COH | Cohort | Integer | None | Never | COH=1. To be entered in all rows for each participant. |
| AGE | Participant<br>Age | Integer | year | If missing impute with -99 | From source data. To be entered in all rows for each participant. |
| SEX | Participant gender | Integer | None | Never | 0=Male, 1=Female To be entered in all rows for each participant. |
| SEXTEXT | Participant gender text | Char | None | Never | Text corresponding to code for SEX, e.g. MALE or FEMALE). To be entered in all rows for each participant. |
| BMI | Baseline Body<br>Mass Index | Num | kg/m <sup>2</sup> | If missing impute with -99 | Ensure consistent with S&P formula. E.g. Formula: Weight(kg)/(height(m)**2) To be entered in all rows for each participant. |
| BSA | Baseline Body<br>Surface Area | Num | m <sup>2</sup> | If missing impute with -99 | Formula: BSA (m²) = 0.024265 • Height(cm) <sup>0.3964</sup> • Weight(kg) <sup>0.5378</sup> Ensure consistent to with S&P formula. To be entered in all rows for each participant. |
| WT | Baseline<br>Participant<br>weight | Num | kg | If missing impute with -99 | From source data. To be entered in all rows for each participant. |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing<br>value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| НТ | Baseline<br>Participant<br>height | Num | m | If missing impute with -99 | From source data. To be entered in all rows for each participant. |
| RACE1 | Participant race code1 | Integer | None | Never | From source data e.g. 1=African American / African Heritage 2=American Indian or Alaska Native 3=Asian – Central / South Asian Heritage 4=Asian – East Asian Heritage 5=Asian – Japanese Heritage 6=Asian – South East Asian Heritage 7=Asian – Mixed Race 8=Native Hawaiian or other Pacific Islander 9=White – Arabic / North African Heritage 10=White – White / Caucasian / European Heritage 11=White – Mixed Race 12=Mixed Race To be entered in all rows for each participant. |
| RACE1TXT | Participant race 1 text | Char | None | Never | Text corresponding to code for RACE1 To be entered in all rows for each participant. |
| RACE2 | Participant race code2 | Integer | None | Never | 1=East Asian: Asian – East Asian Heritage & Asian – Japanese Heritage 2=White: White – Arabic / North African Heritage White – White / Caucasian / European Heritage 3=African: African American / African Heritage; 4=Other: American Indian or Alaska Native; Asian – Central / South Asian Heritage; Asian – South East Asian Heritage; Asian – Mixed Race; Native Hawaiian or other Pacific Islander; White – Mixed Race & Mixed Race To be entered in all rows for each participant. |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| RACE2TXT | Participant race 2 text | Char | None | Never | Text corresponding to code for RACE2 To be entered in all rows for each participant. |
| ETHN | Participant ethnicity | Num | None | Never | From source data definition. E.g 1=Hispanic or Latino, 2=Non-Hispanic To be entered in all rows for each participant. |
| ETHNTEXT | Participant ethnicity text | Char | None | Never | Text corresponding to code for ETHN. To be entered in all rows for each participant. |
| REGN | Region for participant | Num | None | Never | 1 = East Asia (to include Japan,<br>South Korea and Taiwan)<br>2 = Rest of the World (to include<br>all other countries)<br>To be entered in all rows for each<br>participant. |
| SMOK | Participant<br>smoking<br>status | Integer | None | Never | 0=Non-smoker, 1=Smoker,<br>2=Former smoker<br>To be entered in all rows for each<br>participant. |
| SMOKTEXT | Participant<br>smoking<br>status text | Char | None | Never | Text corresponding to code for SMOK. To be entered in all rows for each participant. |
| CMED1 | COPD<br>conmeds<br>identifier | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each participant. |
| CMED1TXT | Participant<br>CMED1 text | Char | None | Never | Text corresponding to code for CMED1. To be entered in all rows for each participant. |
| CRCL | Baseline<br>Creatinine<br>Clearance | Num | mL/min | If missing impute with -99 | From source data. OR Specify appropriate formula e.g. Creatinine Clearance will be calculated based on the Cockcroft-Gault equation. • CrCL (ml/min) = [140 – AGE (in years)]*Weight(kg)*0.85 (for female particpants) / |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| | | | | | [72* Serum Creatinine (micromol/L) * 0.0113 • CrCL (mL/min) = (140 – Age (yr)) * IBW (kg) / (72 • SCr (μmol/L) * 0.0113) * [0.85 if female], where IBW (kg) = 50 (kg) [ - 4.5 (kg) if female]+ 2.3 (kg) * (HT (inch) - 60) • Delete one as appropriate and ensure consistency with S&P formula • To be entered in all rows for each participant. |
| CMED2 | Gastric acid reducing conmeds identifier | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each participant. |
| CMED2TXT | Participant<br>CMED2 text | Char | None | Never | Text corresponding to code for CMED2. To be entered in all rows for each participant. |
| CMED3 | Identifier for on-treatment gastric acid increasing concomitant medication | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each participant. |
| CMED3TXT | Participant concomitant medication text | Char | None | Never | Text corresponding to code for CMED3. To be entered in all rows for each participant. |
| CMED4 | P-gp inhibitor<br>conmeds<br>identifier | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each participant. |
| CMED4TXT | Participant<br>CMED4 text | Char | None | Never | Text corresponding to code for CMED4. To be entered in all rows for each participant. |
| CMED5 | Identifier for on-treatment p-gp inducer concomitant medication | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each participant. |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing<br>value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| CMED5TXT | Participant concomitant medication text | Char | None | Never | Text corresponding to code for CMED5. To be entered in all rows for each participant. |
| ALB | Baseline<br>Albumin | Num | Specify | If missing impute with -99 | Baseline defined in the source dataset To be entered in all rows for each participant. |
| TBIL | Baseline Total bilirubin | Num | Specify | If missing impute with -99 | Baseline defined in the source dataset To be entered in all rows for each participant. |
| TFIB | Baseline<br>Fibrinogen | Num | Specify | If missing impute with -99 | Baseline defined in the source dataset To be entered in all rows for each participant. |

#### **<u>Current Therapies for COPD:</u>** CMED1

| Therapy | Efficacy Claims | Main Safety Concerns |
|---|---|---|
| Long-acting β <sub>2</sub> -agonists (LAI | BAs) | |
| Formoterol<br>Indacaterol<br>Salmeterol<br>Olodaterol | Bronchodilator treatment to relieve symptoms in patients with COPD. Not used alone, generally in combination with inhaled corticosteroids and LAMAs. | Adverse reactions related to β receptor agonist pharmacology e.g. tremor, tachycardia, hypokalaemia, hyperglycaemia. Use of indacaterol has been associated with post-inhalation cough. Hypersensitivity reactions can occur with ICS, LAMA and LABAs, but are unlikely to affect the majority of patients. Cardiovascular effects have also been associated with use of muscarinic antagonists and β2 agonists in patients with COPD. |

| Therapy | Efficacy Claims | Main Safety Concerns |
|---|---|---|
| Long acting anti-muscarinic a | Long acting anti-muscarinic antagonists (LAMAs) | |
| Tiotropium<br>Aclidinium Bromide<br>Glycopyrronium bromide<br>Umeclidinium | Bronchodilator treatment to relieve symptoms in patients with COPD. Same as above. | Adverse reactions related to anti-<br>muscarinic pharmacology. The<br>most commonly reported adverse<br>effects include dry mouth, GI<br>effects and upper respiratory<br>system infection. |
| | | Hypersensitivity reactions can occur with ICS, LAMA and LABAs, but are unlikely to affect the majority of patients |
| | | Cardiovascular effects have also been associated with use of muscarinic antagonists and $\beta_2$ agonists in patients with COPD. |
| Long acting combination bro | nchodilators | |
| Albuterol/ipratropium bromide Vilanterol/umeclidinium Olodaterol/tiotropium Indacaterol/glycopyrrolate Formoterol/glycopyrrolate Formoterol/aclidinium | Bronchodilator treatment<br>superior to LABA or<br>LAMA alone relieving<br>symptoms in patients with<br>COPD. | Adverse reactions related to β receptor agonist and antimuscarinic pharmacology |
| Methylxanthines | | |
| Theophylline<br>Aminophylline | Bronchodilator effects and claimed anti-inflammatory effects. | Dose-related toxicity including the development of atrial and ventricular arrhythmias and grand mal seizures. |
| Inhaled glucocorticosteroids | | |
| Beclomethasone Budesonide Fluticasone propionate Fluticasone furoate Mometasone | Anti-inflammatory effects;<br>normally used in<br>combination with LAMAs<br>and LABAs | The class effects of inhaled corticosteroids can include oral candidiasis, hoarse voice, skin bruising and increased risk of pneumonia. Systemic corticosteroid class effects including hypothalamic-pituitary-adrenal (HPA) axis suppression, decrease in bone mineral density and ocular disorders (e.g. glaucoma and cataracts). Pneumonia is a recognized class |

| Therapy | Efficacy Claims | Main Safety Concerns |
|---|---|---|
| | | risk with the use of inhaled corticosteroid (ICS) in COPD [Spencer, 2011; Drummond, 2008], however, the benefit of ICS continue to outweigh the risks [EMA, 2016] Hypersensitivity reactions can occur with ICS, LAMA and LABAs, but are unlikely to affect the majority of patients. |
| Inhaled glucocorticosteroids | (ICS, in combination with inh | aled bronchodilators) |
| Formoterol/budesonide Salmeterol/Fluticasone propionate Vilanterol/Fluticasone Furoate | An inhaled corticosteroid combined with a LABA is more effective than the individual components in | As described for LABAs and inhaled glucocorticosteriods above. |
| Formoterol/mometasone Formoterol/mometasone | reducing exacerbations and improving lung function and health status. | Crim et al. (2015) pneumonia was shown to be more frequent in patients who received fluticasone/vilanterol than those who received vilanterol alone. |
| Inhaled glucocorticosteroids | (ICS, in combination with inh | aled LABA and LAMA) |
| Fluticasone<br>Furoate/Umeclidium/Vilanterol | Adding a LAMA to existing LABA/ICS improves lung function and patient reported outcomes in particular, exacerbation risk. | As described for LABAs, LAMAs and inhaled corticosteroids above. |
| Phospodiesterase-4 inhibitor | S | |
| Roflumilast | Reduction of exacerbations in patients with severe COPD. Modest improvement in FEV1 (versus placebo) and small improvements in SCRQ and COPD-related systems. No significant changes in exercise tolerance with PDE4 inhibitors. Unclear benefit on modifying FEV1 decline, hospitalization or mortality in COPD. [Chong J et al. 2013]. | Weight loss, abdominal pain, diarrhoea, nausea, headache and sleep disturbances. Caution for use is advised in patients with depression. |

| Therapy | Efficacy Claims | Main Safety Concerns |
|---|---|---|
| Antibiotics | | |
| Macrolides (e.g. azithromycin, erythromycin) | Regular use of may reduce exacerbation rate. Azithromycin or erythromycin for one year in patients prone to exacerbations reduced the risk of exacerbations compared to usual care. | Azithromycin use associated with increased incidence of bacterial resistance and impaired hearing. |

## **CMED2: Gastric acid reducing conmeds**

| 0bs | VAR1 | VAR2 |
|---|---|---|
| 1<br>2<br>3<br>4<br>5<br>6<br>7<br>8<br>9<br>10<br>11<br>12<br>13<br>14<br>15<br>16<br>17<br>18<br>19<br>20<br>21<br>22<br>23<br>24<br>25<br>26<br>27<br>28<br>29<br>30<br>31<br>32<br>33<br>34<br>35 | Term Name ESOMEPRAZOLE MAGNESIUM PEPTAZOL (NOS) DOMPERIDONE MALEATE + RABEPRAZOLE SODIUM CLARITHROMYCIN + LANSOPRAZOLE PANTOPRAZOLE ESOMEPRAZOLE ESOMEPRAZOLE DOMPERIDONE + PANTOPRAZOLE ZEGERID (NOS) LANSOPRAZOLE SODIUM ESOMEPRAZOLE STRONTIUM ESOGARD (NOS) OMEPRAZOLE MAGNESIUM ZOLTUM (NOS) TENATOPRAZOLE PRAZOL (NOS) DEXLANSOPRAZOLE DOMPERIDONE + RABEPRAZOLE DOMPERIDONE + RABEPRAZOLE CLARITHROMYCIN + LANSOPRAZOLE + TINIDAZOLE LEVOSULPIRIDE + RABEPRAZOLE SODIUM LEVOSULPIRIDE + RABEPRAZOLE PROTON PUMP INHIBITOR NOS IPP (NOS) OMEPRAZOLE SODIUM PANTOPRAZOLE SODIUM PANTOPRAZOLE SODIUM PANTOPRAZOLE SODIUM POMPERIDONE MALEATE + PANTOPRAZOLE SODIUM PROTONIX (NOS) GASTROZOL (NOS) OMEPRAZOLE + SODIUM BICARBONATE ALIMENTARY TRACT AND METABOLISM; DRUGS FOR LANSOPRAZOLE MOSAPRIDE CITRATE + RABEPRAZOLE SODIUM ESOMEPRAZOLE | 54543201<br>54411301<br>54724001<br>53827801 |

**NDAY**: For deriving the nominal day which is the planned day, DAY specific information is not available in EXPOSURE dataset. VISIT variable and the time and events table might have to be taken into account to find the exact plan of events.

**NOMT:** It is twice daily dosing with inter-dose interval given to be 12 hours. Therefore, to find the planned time of event since the first dose in hours, again the VISIT variable and time and events will have to be considered.

**NOMTLD**: In case of PK\_GSK1325756 records, the planned time point variable will give the value of this variable for all the post-dose records. For the pre-dose records, this variable will have missing values since there is no fixed time point since the previous dose for pre-dose records.

**RTFD**: The time difference between the first dose of the subject and the current dose (when LABL=DOSE\_GSK1325756) should be calculated in hours. The time difference between the first dose of the subject and the PK sample collection time (when LABL=PK\_GSK1325756) should be calculated in hours.

**RTLD**: The latest dose prior to the PK sample collection time will have to be found out and the time difference between that dose and the PK sample collection time will be calculated in hours.

## 14.10. Appendix 10: Abbreviations & Trade Marks

#### 14.10.1. Abbreviations

| Abbreviation | Description |
|--------------|----------------------------------------------------|
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALLSUB | |
| ALLSUB | All Subjects Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical Classification |
| BD | Bronchodilator |
| BP | Blood Pressure |
| BUN | Blood urea nitrogen |
| C-PPAC | Clinical Visit PROactive Physical Activity in COPD |
| CAT | COPD Assessment Test |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CID | Clinically Important Deterioration |
| CMH | Chronic Mucus Hypersecretion |
| Crl | Credible Interval |
| COPD | Chronic Obstructive Pulmonary Disease |
| CSR | Clinical Study Report |
| DBF | Database Freeze |
| DM | Data Management |
| DP | Decimal Places |
| E-RS: COPD | Evaluating Respiratory Symptoms in COPD |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| EW | Early Withdrawal |
| EXACT | Exacerbations of Chronic Pulmonary Disease Tool |
| FEV1 | Forced Expiratory Volume in 1 Second |
| FUP | Functional Uniform Prior |
| FVC | Forced Vital Capacity |
| GGT | Gamma-glutamyl transferase |
| GOLD | Global Initiative for Obstructive Lung Disease |
| GSK | GlaxoSmithKline |
| HCRU | Healthcare Resource Utilization |
| IDSL | Integrated Data Standards Library |
| LS | Least Squares |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCSE | Monte Carlo Standard Error |
| MCV | Microtic cell volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-treat |

| Abbreviation | Description |
|--------------|-----------------------------------------|
| MLE | Maximum likelihood estimate |
| MMRM | Mixed Model Repeated Measures |
| NQ | Non-quantifiable |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PopPK | Population PK |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| RMC | Respiratory Medication Class |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SE | Standard Error |
| SDL | Source Data Lock |
| SDTM | Study Data Tabulation Model |
| SGOT | Serum glutamic oxalocaetic transaminase |
| SGPT | Siamane glutamate pyruvate transaminase |
| SGRQ | St. George's Respiratory Questionnaire |
| SGRQ-C | SGRQ for COPD patients |
| SI | System Independent |
| SMQ | Standardized MedDRA Query |
| SRDP | Study Results Dissemination Plan |
| ULN | Upper limit of normal |

#### 14.10.2. Trademarks

| Trader | marks of the GlaxoSmithKline<br>Group of Companies |
|--------|----------------------------------------------------|
| NONE | |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

#### 14.11. Appendix 11: List of Data Displays

## 14.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Strategic Interim | Statistical Analysis Complet | te |
|---|---|---|
| Section | Tables | Figures |
| Study Population | 1.1 to 1.20 | |
| Efficacy | 2.1 to 2.52 | 2.1 to 2.35 |
| Conditional Efficacy | | 2.36 to 2.xx |
| Safety | 3.1 to 3.23 | 3.1 to 3.6 |
| Pharmacokinetic | | |
| Pharmacokinetic / Pharmacodynamic | | |
| Biomarker | 6.1 to 6.2 | 6.1 to 6.2 |
| Section | List | ings |
| ICH Listings | 1 t | o 1 |
| Other Listings | 2 t | o 2 |
| Final Statistical Analy | rsis Complete (Including Pos | t SAC) |
| Section | Tables | Figures |
| Study Population | 1.1 to 1.43 | 1.1 |
| Efficacy | 2.1 to 2.49 | 2.1 to 2.32 |
| Conditional Efficacy | | 2.33 to 2.xx |
| Safety | 3.1 to 3.37 | 3.1 to 3.11 |
| Pharmacokinetic | 4.1 to 4.8 | 4.1 to 4.13 |
| Pharmacokinetic / Pharmacodynamic | | 5.1 to 5.4 |
| Biomarker | 6.1 to 6.4 | 6.1 to 6.4 |
| Section | List | ings |
| ICH Listings | 1 to 36 | |
| Other Listings | 37 to 69 | |

#### 14.11.2. Deliverables

In all displays the term "Subjects" is used to refer to "Participants".

| Delivery [Priority] | Description |
|---------------------|-------------------------------------------------|
| StInt | Strategic Interim Statistical Analysis Complete |
| SAC | Final Statistical Analysis Complete |
| Post SAC | Additional outputs provided after SAC |

# 14.11.3. Study Population Tables

| Study | Popula | ation Tables | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Partic | ipant D | isposition | · | | · | |
| 1.1 | 1.1 | mITT | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT<br>Include number of ongoing<br>participants for strategic<br>interim | StInt, SAC |
| | 1.2 | All Subjects | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| | 1.3 | All Subjects | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical<br>Operations | SAC |
| 1.2 | 1.4 | mITT | NS1 | Summary of Number of Subjects by Country and Site ID | | StInt, SAC |
| 1.3 | 1.5 | PP | NS1 | Summary of Number of Subjects by Country and Site ID | | StInt, SAC |
| 1.4 | 1.6 | mITT | | Summary of Attendance at Each Clinic Visit | | StInt, SAC |
| Proto | col Dev | riation | | | | |
| | 1.7 | mITT | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| | 1.8 | All Subjects | IE2 | Summary of Inclusion/ Exclusion/ Randomization<br>Criteria Deviations for Screen or Run-in failures | Add a row "Number of<br>Screen Failures" above<br>"any criteria deviations".<br>Percentage will be based<br>on number of screen<br>failures | SAC |

| Study | Popula | ation Tables | | | | |
|---|---|---|---|---|---|---|
| Stint<br>No. | SAC<br>No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | 1.9 | mITT | IE1 | Summary of Inclusion/ Exclusion/ Randomization<br>Criteria Deviations for the Modified Intent-to-treat<br>Population | | SAC |
| Popul | lation A | nalysed | | | | |
| 1.5 | 1.10 | All Subjects | SP1 | Summary of Study Populations | IDSL Number of participants who were in the All Participants population, who were randomized, the number in the ITT population (Strategic interim only), the number in the mITT population. Of those in the mITT, the number and percentage of participants in the PP, Symptomatic (Strategic interim only), PK and PK2 populations | StInt, SAC |
| | 1.11 | mITT | SP2 | Summary of Exclusions from the Per Protocol Population | IDSL | SAC |
| Demo | graphi | c and Baseline Cha | aracteristics | | | |
| 1.6 | 1.12 | mITT | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | StInt, SAC |
| 1.7 | 1.13 | PP | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | StInt, SAC |
| | 1.14 | All Subjects | DM11 | Summary of Age Ranges | EudraCT | SAC |
| | 1.15 | mITT | DM6 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA,<br>EudraCT | SAC |

| Study | Popula | ation Tables | | | | |
|---|---|---|---|---|---|---|
| Stint<br>No. | SAC<br>No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | 1.16 | All Subjects | EMA Table 1 | Summary of Number of Subjects Enrolled by Country | EMA Reporting Package. Macro: EMA_COUNTRY | SAC |
| | 1.17 | All Subjects | EMA Table 2 | Summary of Number of Subjects Enrolled by Age Category | EMA Reporting Package.<br>Macro: EMA_AGEGRP | SAC |
| 1.8 | 1.18 | mITT | SU1 | Summary of Smoking History and Smoking Status at Screening | Include smoking status,<br>smoking pack years,<br>cigarettes smoked/day | StInt, SAC |
| 1.9 | 1.19 | PP | SU1 | Summary of Smoking History and Smoking Status at Screening | Include smoking status,<br>smoking pack years,<br>cigarettes smoked/day | StInt, SAC |
| 1.10 | | Symptomatic | SU1 | Summary of Smoking History and Smoking Status at Screening | Include smoking status,<br>smoking pack years,<br>cigarettes smoked/day | StInt |
| | 1.20 | mITT | SP_T12 | Summary of COPD History at Screening | | SAC |
| 1.11 | 1.21 | mITT | SP_T13 | Summary of HCRU Exacerbation History at Screening | See notes in Section 14.6.3 | StInt, SAC |
| 1.12 | 1.22 | PP | SP_T13 | Summary of HCRU Exacerbation History at Screening | See notes in Section 14.6.3 | StInt, SAC |
| 1.13 | 1.23 | mITT | | Summary of Screening Spirometry Measures | Pre-BD FEV1 (L), Post-BD FEV1 (L), Predicted normal FEV1 (L), Percent predicted normal post-BD FEV1 (%), Percent predicted normal post-BD FEV1: <50%, >=50%, Post-BD FVC (L), Post-BD FEV1/FVC | StInt, SAC |

| Study | Popula | tion Tables | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.14 | 1.24 | PP | | Summary of Screening Spirometry Measures | Pre-BD FEV1 (L), Post-BD FEV1 (L), Predicted normal FEV1 (L), Percent predicted normal post-BD FEV1 (%), Percent predicted normal post-BD FEV1: <50%, >=50%, Post-BD FVC (L), Post-BD FEV1/FVC | StInt, SAC |
| | 1.25 | mITT | | Summary of GOLD Stages at Screening | GOLD 1-4 and GOLD A-D | SAC |
| 1.15 | 1.26 | mlTT | | Summary of Baseline Symptomatic Characteristics | Proportion of participants with CMH ± according to SGRQ, with baseline E-RS: COPD total score =10, with baseline CAT Score =10, with ICS+LABA+LAMA vs. ICS+LABA vs. LABA+LAMA vs. Other COPD medication | StInt, SAC |

| Study | Popula | ation Tables | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.16 | 1.27 | PP | | Summary of Baseline Symptomatic Characteristics | Proportion of participants with CMH ± according to SGRQ, with baseline E-RS: COPD total score =10, with baseline CAT Score =10, with ICS+LABA+LAMA vs. ICS+LABA vs. LABA+LAMA vs. Other COPD medication | StInt, SAC |
| Prior | and Co | ncomitant Medication | ons | | | |
| | 1.28 | mITT | CM1 | Summary of COPD Concomitant Medications Taken Pre-treatment | Use RMC instead of ATC Level 1 | SAC |
| | 1.29 | mITT | CM1 | Summary of COPD Concomitant Medications Taken On-Treatment, Medications Given for Reasons Other than an Exacerbation | Use RMC instead of ATC Level 1 | SAC |
| | 1.30 | mITT | CM1 | Summary of COPD Concomitant Medications Taken Post-treatment | Use RMC instead of ATC Level 1 | SAC |
| | 1.31 | mITT | CM1 | Summary of On-treatment COPD Concomitant Medications Given for an Exacerbation | Use RMC instead of ATC Level 1 | SAC |
| 1.17 | 1.32 | mITT | | Summary of COPD Concomitant Medication<br>Combinations Taken at Screening | Number and percentage of participants taking each medication in the RMC combination defined in Section 14.6.2 | StInt, SAC |

| Study | Popula | ation Tables | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.18 | 1.33 | mITT | | Summary of COPD Concomitant Medication<br>Combinations Taken at Baseline | Number and percentage of participants taking each medication in the RMC combination defined in Section 14.6.2 | StInt, SAC |
| 1.19 | | Symptomatic | | Summary of COPD Concomitant Medication<br>Combinations Taken at Baseline | Number and percentage of participants taking each medication in the RMC combination defined in Section 14.6.2 | StInt |
| | 1.34 | PP | | Summary of COPD Concomitant Medication<br>Combinations Taken at Month 6 | Number and percentage of participants taking each medication in the RMC combination defined in Section 14.6.2 during Month 6 | Post SAC |
| | 1.35 | mITT | CM1 | Summary of On-treatment Non-COPD Concomitant Medications | Use ATC Level 1 | SAC |
| | 1.36 | mITT | CM1 | Summary of Post-treatment Non-COPD Concomitant Medications | Use ATC Level 1 | SAC |
| Past a | nd Cur | rent Medical Histor | у | | | |
| | 1.37 | mITT | MH4 | Summary of Past Medical Conditions | ICH E3 | SAC |
| | 1.38 | mITT | MH4 | Summary of Current Medical Conditions | | SAC |
| | 1.39 | mITT | Table 1.23<br>Study<br>GSK2834425/CTT116853 | Summary of Cardiovascular History/Risk Factors | | SAC |

| Study | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.20 | 1.40 | mITT | FH1 | Summary of Family History of Cardiovascular Risk Factors | | StInt, SAC |
| Expos | ure and | d Treatment Compli | ance | | | |
| | 1.41 | mITT | IP1 | Summary of Treatment Compliance | | SAC |
| | 1.42 | mITT | | Summary of Daily Diary Compliance | | SAC |
| | 1.43 | mITT | EX1 | Summary of Exposure to Study Treatment | ICH E3 | SAC |

## 14.11.4. Study Population Figures

| Study P | Study Population Figures | | | |
|---|---|---|---|---|
| SAC<br>No. | Population Example Litle | Title | Programming Notes | Deliverable<br>[Priority] |
| Disposi | Disposition of Subjects | | | |
| 1.1. | 1.1. mITT | Kaplan-Meier Plot of Time to Study Withdrawal | | SAC |

# 14.11.5. Efficacy Tables

| Efficac | y: Tables | <b>5</b> | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| E-RS: | COPD | | | | | |
| 2.1 | 2.1 | PP | PD4 | Summary of Baseline E-RS: COPD Scores | Endpoints: E-RS: COPD total and subscale scores Include total column | StInt, SAC |
| 2.2 | | Symptomatic | PD4 | Summary of Baseline E-RS: COPD Scores | Endpoints: E-RS: COPD total and subscale scores Include total column | StInt |
| 2.3 | 2.2 | PP | PD4 | Summary of Monthly Mean E-RS: COPD Scores | Endpoints: E-RS: COPD total and subscale scores Include raw and change from baseline scores for participants with non-missing E-RS data for each month | StInt, SAC |
| 2.4 | | Symptomatic | PD4 | Summary of Monthly Mean E-RS: COPD Scores | Endpoints: E-RS: COPD total and subscale scores Include raw and change from baseline scores for participants with non-missing E-RS data for each month | StInt |
| 2.5 | 2.3 | PP | | Bayesian Dose Response Analysis of Change from Baseline E-RS: COPD Scores at Month 6 | Endpoint: Month 6 E-RS: COPD total and subscale scores | StInt, SAC |
| 2.6 | | Symptomatic | | Bayesian Dose Response Analysis of Change from Baseline E-RS: COPD Total Score at Month 6 | Endpoint: Month 6 E-RS: COPD total score | StInt |

| Efficac | y: Tables | ; | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.7 | 2.4 | PP | | Bayesian Analysis of Change from Baseline<br>Monthly Mean E-RS: COPD Scores up to<br>Month 6 | Bayesian MMRM on Change from Baseline Endpoints: E-RS: COPD total and subscale scores | StInt, SAC |
| 2.8 | | Symptomatic | | Bayesian Analysis of Change from Baseline<br>Monthly Mean E-RS: COPD Scores up to<br>Month 6 | Bayesian MMRM on Change from Baseline Endpoints: E-RS: COPD total and subscale scores | StInt |
| 2.9 | | ITT | | Bayesian Analysis of Change from Baseline<br>Monthly Mean E-RS: COPD Scores up to<br>Month 6 | Bayesian MMRM on Change from Baseline Endpoints: E-RS: COPD total and subscale scores | StInt |
| 2.10 | 2.5 | PP | | Analysis of Change from Baseline Monthly<br>Mean E-RS: COPD Total Score up to Month 6 | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt, SAC |
| 2.11 | 2.6 | PP | | Type III Tests of Fixed Effects for Analysis of Change from Baseline Monthly Mean E-RS: COPD Total Score up to Month 6 | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt, SAC |
| 2.12 | 2.7 | PP | | Analysis of Proportion of Responders<br>According to Monthly Mean E-RS: COPD<br>Scores up to Month 6 | Responder Analysis Generalized linear model Endpoints: E-RS: COPD total and subscale scores | StInt, SAC |
| 2.13 | 2.8 | PP | | Analysis of Change from Baseline Monthly<br>Mean E-RS: COPD Total Score up to Month 6:<br>Interaction of Treatment with Other Factors | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt, SAC |

| Efficac | y: Table: | s | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.14 | | PP | | Analysis of Change from Baseline Monthly Mean E-RS: COPD Total Score up to Month 6 by Baseline E-RS: COPD Total Score (<10, >=10) | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt |
| 2.15 | 2.9 | PP | | Analysis of Change from Baseline Monthly<br>Mean E-RS: COPD Total Score up to Month 6<br>by Smoking Status at Screening (Current,<br>Former) | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt, SAC |
| 2.16 | | PP | | Analysis of Change from Baseline Monthly<br>Mean E-RS: COPD Total Score up to Month 6<br>by Country | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt |
| 2.17 | 2.10 | PP | | Analysis of Change from Baseline Monthly<br>Mean E-RS: COPD Total Score up to Month 6<br>by % Predicted FEV1 at Screening (<50, >=50) | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt, SAC |
| 2.18 | 2.11 | PP | | Analysis of Change from Baseline Monthly Mean E-RS: COPD Total Score up to Month 6 by Baseline CAT Score (<10, >=10) | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt, SAC |
| 2.19 | | PP | | Analysis of Change from Baseline Monthly Mean E-RS: COPD Total Score up to Month 6 by Exacerbation History (>=2 moderate/severe vs. 1 moderate/severe, prior year) | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt |
| 2.20 | | PP | | Analysis of Change from Baseline Monthly<br>Mean E-RS: COPD Total Score up to Month 6<br>by COPD Medication Grouping at Baseline<br>(ICS+LABA+LAMA, ICS+LABA, LABA+LAMA,<br>Other) | Frequentist MMRM<br>Endpoints: E-RS: COPD total score | StInt |

| Efficac | y: Tables | S | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.21 | | PP | | Analysis of Change from Baseline Monthly<br>Mean E-RS: COPD Total Score up to Month 6<br>by CMH Status at Baseline | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt |
| 2.22 | | PP | | Analysis of Change from Baseline Monthly<br>Mean E-RS: COPD Total Score up to Month 6<br>by Season | Frequentist MMRM Endpoints: E-RS: COPD total score | StInt |
| | 2.12 | | | Summary of Responders to E-RS: COPD Total Score, SGRQ and CAT at Month 6 | Include categories for E-RS, SGRQ,<br>CAT, E-RS+SGRQ, E-RS+CAT.<br>SGRQ+CAT, E-RS+SGRQ+CAT, None,<br>Missing | Post SAC |
| Exace | rbations | | | | | |
| 2.23 | 2.13 | PP | | Summary of On-treatment HCRU Exacerbations | | StInt, SAC |
| | 2.14 | PP | | Summary of On-treatment Details of Moderate/Severe HCRU Exacerbations | | SAC |
| | 2.15 | PP | | Summary of On-treatment HCRU<br>Exacerbations Treated with Antibiotics | Include row for how many subjects were receiving ICS for at least 7 days at the time of exacerbation | Post SAC |
| 2.24 | 2.16 | PP | | Bayesian Analysis of On-treatment<br>Moderate/Severe HCRU Exacerbations | Bayesian generalized linear model | StInt, SAC |
| 2.25 | | ITT | | Bayesian Analysis of On-treatment<br>Moderate/Severe HCRU Exacerbations | Bayesian generalized linear model | StInt, |
| 2.26 | 2.17 | PP | | Summary and Bayesian Analysis of Time to First On-treatment Moderate/Severe HCRU Exacerbation | Bayesian proportional hazards model | StInt, SAC |

| Efficac | y: Tables | • | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27 | 2.18 | PP | | Summary and Bayesian Analysis of Time to First On-treatment Severe HCRU Exacerbation | Bayesian proportional hazards model | StInt, SAC |
| EXACT | Events | | • | | | |
| | 2.19 | PP | | Summary of On-treatment EXACT Events | | SAC |
| | 2.20 | PP | | Bayesian Analysis of On-treatment EXACT Events | Bayesian generalized linear model | SAC |
| | 2.21 | PP | | Summary and Bayesian Analysis of Time to First On-treatment EXACT Events | Bayesian proportional hazards model | SAC |
| SGRQ | | | | | | |
| 2.28 | 2.22 | PP | PD4 | Summary of Baseline SGRQ Scores | Include total column Total and domain scores | StInt, SAC |
| 2.29 | 2.23 | PP | PD4 | Summary of SGRQ Scores | Include raw and change from baseline Total and domain scores | StInt, SAC |
| 2.30 | 2.24 | PP | | Bayesian Analysis of Change from Baseline SGRQ Total Score up to Month 6 | Bayesian MMRM on Change from Baseline Endpoints: SGRQ Total Score | StInt, SAC |
| 2.31 | 2.25 | PP | | Analysis of Proportion of Responders<br>According to SGRQ Total Scores up to Month 6 | Responder Analysis<br>Generalized linear model | StInt, SAC |
| CAT | | | | | | |
| 2.32 | 2.26 | PP | PD4 | Summary of Baseline CAT Score | Include total column | StInt, SAC |
| 2.33 | 2.27 | PP | PD4 | Summary of CAT Score | Include raw and change from baseline | StInt, SAC |

| Efficac | y: Table | s | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.34 | 2.28 | PP | | Bayesian Analysis of Change from Baseline CAT Score up to Month 6 | Bayesian MMRM on Change from Baseline Endpoints: CAT Score | StInt, SAC |
| 2.35 | 2.29 | PP | | Analysis of Proportion of Responders<br>According to CAT Score up to Month 6 | Responder Analysis<br>Generalized linear model | StInt, SAC |
| 2.36 | 2.30 | PP | | Analysis of Change from Baseline CAT Score up to Month 6: Interaction of Treatment with Other Factors | Frequentist MMRM Endpoints: CAT Score | StInt, SAC |
| 2.37 | | PP | | Analysis of Change from Baseline CAT Score up to Month 6 by Baseline E-RS: COPD Total Score (<10, >=10) | Frequentist MMRM Endpoints: CAT Score | StInt |
| 2.38 | 2.31 | PP | | Analysis of Change from Baseline CAT Score up to Month 6 by Smoking Status at Screening (Current, Former) | Frequentist MMRM Endpoints: CAT Score | StInt, SAC |
| 2.39 | | PP | | Analysis of Change from Baseline CAT Score up to Month 6 by Country | Frequentist MMRM Endpoints: CAT Score | StInt |
| 2.40 | 2.32 | PP | | Analysis of Change from Baseline CAT Score up to Month 6 by % Predicted FEV1 at Screening (<50, >=50) | Frequentist MMRM Endpoints: CAT Score | StInt, SAC |
| 2.41 | 2.33 | PP | | Analysis of Change from CAT Score up to<br>Month 6 by Baseline CAT Score (<10, >=10) | Frequentist MMRM Endpoints: CAT Score | StInt, SAC |
| 2.42 | | PP | | Analysis of Change from CAT Score up to<br>Month 6 by Exacerbation History (>=2<br>moderate/severe vs. 1 moderate/severe, prior<br>year) | Frequentist MMRM Endpoints: CAT Score | StInt |

| Efficac | Efficacy: Tables | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.43 | | PP | | Analysis of Change from Baseline CAT Score up to Month 6 by COPD Medication Grouping at Baseline (ICS+LABA+LAMA, ICS+LABA, LABA+LAMA, Other) | Frequentist MMRM Endpoints: CAT Score | StInt |
| 2.44 | | PP | | Analysis of Change from Baseline CAT Score up to Month 6 by CMH Status at Baseline | Frequentist MMRM Endpoints: CAT Score | StInt |
| 2.45 | | PP | | Analysis of Change from Baseline CAT Score up to Month 6 by Season | Frequentist MMRM Endpoints: CAT Score | StInt |
| Rescu | e Use | | | | | |
| 2.46 | 2.34 | PP | PD4 | Summary of Baseline Mean Number of Puffs of Rescue Medication per Day using Diary Data | Include total column | StInt, SAC |
| 2.47 | 2.35 | PP | PD4 | Summary of Monthly Mean Number of Puffs of Rescue Medication per Day using Diary Data up to Month 6 | Include raw and change from baseline | StInt, SAC |
| 2.48 | 2.36 | PP | | Analysis of Change from Baseline in Monthly<br>Mean Number of Puffs of Rescue Medication<br>per Day using Diary Data up to Month 6 | MMRM on Change from Baseline | StInt, SAC |
| 2.49 | 2.37 | PP | PD4 | Summary of Baseline Percentage Rescue-free Days using Diary Data | Include total column | StInt, SAC |
| 2.50 | 2.38 | PP | PD4 | Summary of Percentage Rescue-free Days using Diary Data up to Month 6 | Include raw and change from baseline | StInt, SAC |
| 2.51 | 2.39 | PP | | Analysis of Change from Baseline in<br>Percentage Rescue-free Days using Diary Data<br>up to Month 6 | MMRM on Change from Baseline | StInt, SAC |

| Efficac | y: Tables | 3 | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | 2.40 | PP | PD4 | Summary of Baseline Mean Number of<br>Occasions of Rescue Medication per Day using<br>Sensor Data | Include total column | SAC |
| | 2.41 | PP | PD4 | Summary of Monthly Mean Number of<br>Occasions of Rescue Medication per Day using<br>Sensor Data up to Month 6 | Include raw and change from baseline | SAC |
| | 2.42 | PP | | Analysis of Change from Baseline Monthly<br>Mean Number of Occasions of Rescue<br>Medication per Day using Sensor Data up to<br>Month 6 | MMRM on Change from Baseline | SAC |
| | 2.43 | PP | PD4 | Summary of Baseline Percentage Rescue-free Days using Sensor Data | Include total column | SAC |
| | 2.44 | PP | PD4 | Summary of Percentage Rescue-free Days using Sensor Data up to Month 6 | Include raw and change from baseline | SAC |
| | 2.45 | PP | | Analysis of Change from Baseline Percentage<br>Rescue-free Days using Sensor Data up to<br>Month 6 | MMRM on Change from Baseline | SAC |
| Physic | al Activit | ty | | | | |
| | 2.46 | PP | PD4 | Summary of Baseline PROactive Score | Include total column Endpoints: PROactive Total Score and domain scores | SAC |
| | 2.47 | PP | PD4 | Summary of PROactive Score up to Month 6 | Include raw and change from baseline Endpoints: PROactive Total Score and domain scores | SAC |

| Efficac | Efficacy: Tables | | | | | |
|---|---|---|---|---|---|---|
| Stint<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.52 | | PP | | Summary of Responses to C-PPAC Questionnaire at Each Visit | | StInt |
| Subjec | t Global A | Assessments | | | | |
| | 2.48 | PP | PD4 | Summary of Subject Global Assessments at Baseline | Include total column Endpoints: severity, activity limitation | SAC |
| | 2.49 | PP | PD4 | Summary of Subject Global Assessments | Endpoints: severity, change in severity, activity limitation and change in activity limitation | SAC |

## 14.11.6. Efficacy Figures

| Efficacy: | Efficacy: Figures | | | | | |
|---|---|---|---|---|---|---|
| Stint<br>No. | SAC No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| E-RS: CC | )PD | | | | | |
| | 2.1 | PP | | Daily Mean E-RS: COPD Scores over Time | Total and subscale scores Day -7 to Day 168 | Post SAC |
| | 2.2 | PP | | Daily Mean E-RS: COPD Scores over Time by Completion Status | Total and subscale scores Day -7 to Day 168 One page for completers and one page for subjects who withdrew | Post SAC |
| 2.1 | 2.3 | PP | | Daily Mean Change from Baseline in E-RS: COPD Scores over Time | Total and subscale scores | StInt, SAC |

| Efficacy: | Efficacy: Figures | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.2 | 2.4 | PP | | Daily Mean (± SE) Change from Baseline in E-RS: COPD over Time by Dose | Total and subscale scores; one panel for each DNX dose to include DNX and placebo data | StInt, SAC |
| 2.3 | | Symptomatic | | Daily Mean (± SE) Change from Baseline in E-RS: COPD over Time by Dose | Total and subscale scores; one panel for each DNX dose to include DNX and placebo data | StInt |
| | 2.5 | PP | | Daily Mean (± SE) E-RS: COPD over Time by Dose | Total and subscale scores Day -7 to Day 168 | Post SAC |
| 2.4 | 2.6 | PP | | Bayesian Dose Response Model for E-RS: COPD Scores at Month 6 | Total and subscale scores; overlaid with mean/CI from Bayesian longitudinal model | StInt, SAC |
| 2.5 | | Symptomatic | | Bayesian Dose Response Model for E-RS: COPD Total Score at Month 6 | Total score; overlaid with mean/CI from Bayesian longitudinal model | StInt |
| 2.6 | 2.7 | PP | | Posterior Mean (90% Crl) Change from Baseline in E-RS: COPD Scores over Time | Total and subscale scores | StInt, SAC |
| 2.7 | | Symptomatic | | Posterior Mean (90% Crl) Change from Baseline in E-RS: COPD Total Score over Time | Total score | StInt |
| 2.8 | | ITT | | Posterior Mean (90% Crl) Change from Baseline in E-RS: COPD Total Score over Time | Total score | StInt |
| 2.9 | 2.8 | PP | | Adjusted Mean (90% CI) Change from Baseline in E-RS: COPD Total Score over Time | Total score | StInt, SAC |
| | 2.9 | PP | | Adjusted Mean (90% CI) E-RS: COPD Total Score over Time | Total score | Post SAC |

| Efficacy: | Efficacy: Figures | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10 | | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS:COPD Total Score at Month 6 by Baseline E-RS: COPD Total Score (<10, >=10) | One panel for each factor on the same page | StInt |
| 2.11 | 2.10 | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score at Month 6 by Smoking Status at Screening (Current, Former) | One panel for each factor on the same page | StInt, SAC |
| 2.12 | | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score at Month 6 by Country | One panel for each factor, 4 panels per page | StInt |
| 2.13 | 2.11 | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score at Month 6 by % Predicted FEV1 at Screening (<50, >=50) | One panel for each factor on the same page | StInt, SAC |
| 2.14 | 2.12 | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score at Month 6 by Baseline CAT Score (<10, >=10) | One panel for each factor on the same page | StInt, SAC |
| 2.15 | | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score at Month 6 by Exacerbation History (>=2 moderate/severe vs. <2 moderate/severe, prior year) | One panel for each factor on the same page | StInt |
| 2.16 | | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score at Month 6 by COPD Medication Grouping at Baseline (ICS+LABA+LAMA, ICS+LABA, LABA+LAMA, Other) | One panel for each factor on the same page | StInt |
| 2.17 | | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score at Month 6 by CMH Status at Baseline | One panel for each factor on the same page | StInt |

| Efficacy: | Figures | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18 | | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score at Month 6 by Season | All factors on one plot | StInt |
| | 2.13 | PP | | Empirical Distribution Function Plot of E-RS: COPD Total Scores at Baseline | Total and subscale scores | Post SAC |
| | 2.14 | PP | | Empirical Distribution Function Plot of E-RS: COPD Total Scores at Month 6 | Total and subscale scores | Post SAC |
| Exacerba | ations | | | | | |
| 2.19 | 2.15 | PP | | Median Rate Ratio (90% CrI) of On-treatment Moderate/Severe HCRU Exacerbations | | StInt, SAC |
| 2.20 | | ITT | | Median Rate Ratio (90% CrI) of On-treatment Moderate/Severe HCRU Exacerbations | | StInt |
| 2.21 | 2.16 | PP | | Kaplan-Meier Plot of Time to First On-treatment Moderate/Severe HCRU Exacerbation | | StInt, SAC |
| 2.22 | 2.17 | PP | | Kaplan-Meier Plot of Time to First On-treatment Severe HCRU Exacerbation | | StInt, SAC |
| EXACT E | vents | | • | | | <u>.</u> |
| | 2.18 | PP | | Median Rate Ratio (90% CrI) of On-treatment EXACT Events | | SAC |
| | 2.19 | PP | | Kaplan-Meier Plot of Time to First On-treatment EXACT Event | | SAC |
| SGRQ | • | | | | ' | 1 |
| 2.23 | 2.20 | PP | | Posterior Mean (90% Crl) Change from Baseline in SGRQ Total Score over Time | | StInt, SAC |
| | 2.21 | PP | | Mean (90% CI) SGRQ Total Score over Time | Baseline, Day 84 and 168 | Post SAC |

| Efficacy: | Efficacy: Figures | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CAT | | | | | | <u>'</u> |
| 2.24 | 2.22 | PP | | Posterior Mean (90% Crl) Change from Baseline in CAT Score over Time | | StInt, SAC |
| | 2.23 | PP | | Mean (90% CI) CAT Score over Time | Baseline, Day 84 and 168 | Post SAC |
| 2.25 | | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by Baseline E-RS: COPD Total Score (<10, >=10) | One panel for each factor | StInt |
| 2.26 | 2.24 | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by Smoking Status at Screening (Current, Former) | One panel for each factor | StInt, SAC |
| 2.27 | | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by Country | One panel for each factor | StInt |
| 2.28 | 2.25 | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by % Predicted FEV1 at Screening (<50, >=50) | One panel for each factor | StInt, SAC |
| 2.29 | 2.26 | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by Baseline CAT Score (<10, >=10) | One panel for each factor | StInt, SAC |
| 2.30 | | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by Exacerbation History (>=2 moderate/severe vs. 1 moderate/severe, prior year) | One panel for each factor | StInt |

| StInt<br>No. | SAC No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|---|
| 2.31 | | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by COPD Medication Grouping at Baseline (ICS+LABA+LAMA, ICS+LABA, LABA+LAMA, Other) | One panel for each factor | StInt |
| 2.32 | | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by CMH Status at Baseline | One panel for each factor | StInt |
| 2.33 | | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score at Month 6 by Season | All factors on one plot | StInt |
| Rescue | Use | | | | | |
| | 2.27 | PP | | Daily Mean Number of Puffs of Rescue Medication per Day using Diary Data over Time | Day -7 to Day 168 | Post SAC |
| 2.34 | 2.28 | PP | | Least Squares Mean (90% CI) Change from Baseline in Mean Number of Puffs of Rescue Use per Day using Diary Data over Time | | StInt, SAC |
| 2.35 | 2.29 | PP | | Least Squares Mean (90% CI) Change from Baseline in Percentage of Rescue-free Days using Diary Data over Time | | StInt, SAC |
| | 2.30 | PP | | Daily Mean Number of Occasions of Rescue<br>Medication per Day using Sensor Data over Time | Day -7 to Day 168 | Post SAC |
| | 2.31 | PP | | Least Squares Mean (90% CI) Change from Baseline in Mean Number of Occasions of Rescue Use per Day using Sensor Data over Time | | SAC |
| | 2.32 | PP | | Least Squares Mean (90% CI) Change from Baseline in Percentage of Rescue-free Days using Sensor Data over Time | | SAC |
| Efficacy: | Figures | | | | | |
|---|---|---|---|---|---|---|
| Stint<br>No. | SAC No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Condition | nal E-RS: Co | OPD | | | | |
| 2.36-<br>2.43 | 2.33-<br>2.35 | PP | | Least Squares Mean (90% CI) Change from Baseline in E-RS: COPD Total Score over Time by Factor | Produced if an interaction between treatment and factor is significant at the 10% level Where <i>Factor</i> is defined in Section 7.3.1 One panel for each factor | Stlnt, SAC |
| Continue<br>from<br>above | Continue<br>from<br>above | PP | | Least Squares Mean (90% CI) Change from Baseline in CAT Score over Time by <i>Factor</i> | Produced if an interaction between treatment and factor is significant at the 10% level Where <i>Factor</i> is defined in Section 7.3.1 One panel for each factor | StInt, SAC |

## 14.11.7. Safety Tables

| Safety: | Safety: Tables | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | (AEs) | | | | |
| 3.1 | 3.1 | mITT | AE1 | Summary of On-treatment Adverse Events by System Organ Class and Preferred Term | ICH E3 | StInt, SAC |
| 3.2 | 3.2 | mITT | AE3 | Summary of Common (>=5%) On-treatment Adverse Events by Overall Frequency | ICH E3 | StInt, SAC |

| Safety: | Tables | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.3 | 3.3 | mITT | AE1/AE3 | Summary All On-treatment Drug-Related Adverse Events by [System Organ Class and] Preferred Term | ICH E3 Use AE1 for interim with text in [] in title Use AE3 for final reporting with text in [] omitted. | StInt, SAC |
| | 3.4 | mITT | AE15 | Summary of Common (>=5%) Non-serious On-treatment<br>Adverse Events by System Organ Class and Preferred<br>Term (Number of Subject and Occurrences) | FDAAA, EudraCT | SAC |
| | 3.5 | mITT | AE1 | Summary of Post-treatment Adverse Events | | SAC |
| | 3.6 | ALLSUB | AE2 | Relationship of Adverse Event System Organ Class,<br>Preferred Term and Verbatim Text | | SAC |
| | 3.7 | mITT | AE5A | Summary of All On-treatment Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | ICH E3 | SAC |
| | 3.8 | mITT | AE5A | Summary of On-treatment Drug-Related Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | ICH E3 | SAC |
| Serious | s and Oth | ner Significant | Adverse Ever | nts | | |
| | 3.9 | mITT | AE16 | Summary of On-treatment Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | SAC |
| | 3.10 | ALLSUB | AE1/AE3 | Summary of Pre-treatment Serious Adverse Events by [System Organ Class and] Preferred Term | | SAC |
| 3.4 | 3.11 | mITT | AE1/AE3 | Summary of On-treatment Serious Adverse Events by [System Organ Class and] Preferred Term | Use AE1 for interim with text in [] in title Use AE3 for final reporting with text in [] omitted. | StInt, SAC |

| Safety: | Tables | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.5 | 3.12 | mITT | AE1/AE3 | Summary of On-treatment Fatal Serious Adverse Events by [System Organ Class and] Preferred Term | Use AE1 for interim with text in [] in title Use AE3 for final reporting with text in [] omitted. | StInt, SAC |
| 3.6 | 3.13 | mITT | AE1/AE3 | Summary of On-treatment Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by [System Organ Class and] Preferred Term | IDSL Use AE1 for interim with text in [] in title Use AE3 for final reporting with text in [] omitted. | StInt, SAC |
| 3.7 | 3.14 | mITT | | Summary of On-treatment Adverse Events of Special Interest | | StInt, SAC |
| | 3.15 | mITT | | Summary of On-treatment Pneumonia (AE and SAE) by ICS | AE and SAE Subjects who have an event in the 'Infective pneumonia' SMQ By subjects receiving ICS for at least 7 days at the time on pneumonia onset. | Post SAC |
| Labora | tory: Che | emistry | | | | |
| 3.8 | 3.16 | mITT | LB1 | Summary of Chemistry Changes from Baseline | ICH E3, include change from baseline of min/max value | StInt, SAC |
| 3.9 | 3.17 | mITT | LB17 | Summary of Worst Case Chemistry Results by Potential Clinical Importance Criteria | ICH E3 | StInt, SAC |
| Labora | atory: He | matology | • | | | • |
| 3.10 | 3.18 | mITT | LB1 | Summary of Hematology Changes from Baseline | ICH E3, include change from baseline of min/max value | StInt, SAC |
| 3.11 | 3.19 | mITT | LB17 | Summary of Worst Case Hematology by Potential Clinical Importance Criteria | ICH E3 | StInt, SAC |

| Safety: | Tables | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Hep | patobiliary (Liv | ver) | | | |
| 3.12 | 3.20 | mITT | LIVER1 | Summary/Listing of Liver Monitoring/Stopping Event Reporting | IDSL – if there are very small number of events this summary will be replaced with a listing. Table title to be determined by content. | StInt, SAC |
| 3.13 | 3.21 | mITT | LIVER10 | Summary/Listing of Hepatobiliary Laboratory Abnormalities | IDSL – if there are very small number of events this summary will be replaced with a listing. Table title to be determined by content. | StInt, SAC |
| ECG | | | | | | |
| | 3.22 | mITT | EG1 | Summary of ECG Findings | IDSL, include min/max value | SAC |
| | 3.23 | mITT | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL include change from baseline of min/max value | SAC |
| 3.14 | 3.24 | mITT | EG10 | Summary of Maximum QTcF Values Post-Baseline Relative to Baseline by Category | IDSL | StInt, SAC |
| 3.15 | 3.25 | mITT | EG11 | Summary of Maximum Increase in QTcF Values Post-<br>Baseline Relative to Baseline by Category | IDSL | StInt, SAC |
| Vital Si | gns | | | | | |
| | 3.26 | mITT | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3, include change from baseline of min/max value | SAC |
| | 3.27 | mITT | VS7 | Summary of Worst Case Vital Signs Results by Potential Clinical Importance Criteria | IDSL | SAC |

| Safety | Tables | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Spiron | netry | | | | | |
| 3.16 | 3.28 | mITT | | Summary of Baseline Post-Bronchodilator FEV1 (L) | Post bronchodilator FEV1 Include total column | StInt, SAC |
| 3.17 | 3.29 | mITT | | Summary of Post-Bronchodilator FEV1 (L) | Post bronchodilator FEV1 Include raw and change from baseline | StInt, SAC |
| 3.18 | 3.30 | mITT | | Analysis of Change from Baseline Post-Bronchodilator FEV1 (L) up to Month 6 | Frequentist MMRM Endpoints: Post bronchodilator FEV1 | StInt, SAC |
| 3.19 | 3.31 | mITT | | Type III Tests of Fixed Effects for Analysis of Change from Baseline Post-Bronchodilator FEV1 (L) | Frequentist MMRM Endpoints: Post bronchodilator FEV1 | StInt, SAC |
| 3.20 | 3.32 | mITT | | Summary of Baseline Post-Bronchodilator FVC (L) | Post bronchodilator FVC Include total column | StInt, SAC |
| 3.21 | 3.33 | mITT | | Summary of Post-Bronchodilator FVC (L) | Post bronchodilator FVC Include raw and change from baseline | StInt, SAC |
| 3.22 | 3.34 | mITT | | Analysis of Change from Baseline Post-Bronchodilator FVC (L) up to Month 6 | Frequentist MMRM Endpoints: Post bronchodilator FVC | StInt, SAC |
| 3.23 | 3.35 | mITT | | Type III Tests of Fixed Effects for Analysis of Change from Baseline Post-Bronchodilator FVC (L) | Frequentist MMRM Endpoints: Post bronchodilator FVC | StInt, SAC |
| | 3.36 | mITT | | Summary of Baseline Post-Bronchodilator FEV1/FVC | Post bronchodilator FEV1/FVC Include total column | Post SAC |
| | 3.37 | mITT | | Summary of Post-Bronchodilator FEV1/FVC | Post bronchodilator FEV1 Include raw and change from baseline Day 84 and 168 | Post SAC |

# 14.11.8. Safety Figures

| Safety | : Figures | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adver | se Events | 3 | | | | |
| | 3.1 | mITT | AE10 | Plot of Common (>=5%) On-Treatment Adverse Events and Relative Risk | IDSL One page per active treatment compared to placebo Include AEs which have >=5% incidence in any treatment group | SAC |
| Labora | atory | | | | | |
| 3.1 | 3.2 | mITT | LIVER14 | Scatter Plot of Maximum Post-Baseline vs. Baseline for ALT | IDSL | StInt, SAC |
| 3.2 | 3.3 | mITT | LIVER9 | Scatter Plot of Maximum Post-Baseline ALT vs. Maximum Post-Baseline Total Bilirubin | IDSL | StInt, SAC |
| 3.3 | 3.4 | mITT | | Plot of Mean (95% CI) Neutrophil Counts over Time | | StInt, SAC |
| | 3.5 | mITT | | Plot of Mean (95% CI) Neutrophil Counts over Time for Subjects with Pneumonia | | Post SAC |
| Spiro | metry | | | | | |
| | 3.6 | mITT | | Mean (90% CI) Post-Bronchodilator FEV1 (L) over Time | Baseline, Day 84 and 168 | Post SAC |
| 3.4 | 3.7 | mITT | | Adjusted Mean (90% CI) Change from Baseline Post-<br>Bronchodilator FEV1 (L) over Time | | StInt, SAC |
| | 3.8 | mITT | | Mean (90% CI) Post-Bronchodilator FVC (L) over Time | Baseline, Day 84 and 168 | Post SAC |
| 3.5 | 3.9 | mITT | | Adjusted Mean (90% CI) Change from Baseline Post-<br>Bronchodilator FVC (L) over Time | | StInt, SAC |

| Safety: | Safety: Figures | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | 3.10 | mITT | | Mean (90% CI) Post-Bronchodilator FEV1/FVC Ratio over Time | Baseline, Day 84 and 168 | Post SAC |
| ECG | ECG | | | | | |
| 3.6 | 3.11 | mITT | | Boxplot of Change from Baseline in QTcF by Time and Treatment | | StInt, SAC |

#### 14.11.9. Pharmacokinetic Tables

| SAC<br>No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4.1 | PK | PKCT1 | Summary of Danirixin Whole Blood Pharmacokinetic Concentration-Time Data (Dry Blood Spot) | Include geometric mean and 90% CI for the summary of blood concentration data | SAC |
| 4.2 | PK | PKPT4 | Summary of Derived Danirixin Whole Blood Pharmacokinetic Parameters (Dry Blood Spot) | | SAC |
| 4.3 | PK2 | Table 3.10<br>Study 201037 | Summary of Statistical Analysis of Log-Transformed Danirixin<br>Concentration-Time Data<br>Dry Blood Spot vs Wet Whole Blood Samples - Bland Altman<br>Analysis | | SAC |
| 4.4 | PK2 | Table 3.12<br>Study 201037 | Summary of Statistical Analysis of Log-Transformed Danirixin Pharmacokinetic Parameters Dry Blood Spot vs Wet Whole Blood Samples - Bland Altman Analysis | | SAC |
| 4.5 | PK2 | Table 3.11<br>Study 201037 | Summary of Statistical Analysis of Log-Transformed Danirixin Pharmacokinetic Parameters Dry Blood Spot vs Wet Whole Blood Samples | | SAC |

| SAC<br>No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4.6 | PK2 | Table 3.10<br>Study 201037 | Summary of Statistical Analysis of Log-Transformed Danirixin<br>Concentration-Time Data<br>Sensitivity Analysis: Dry Blood Spot vs Wet Whole Blood<br>Samples - Bland Altman Analysis | excluding dry blood spot<br>concentrations above the assay<br>HLOQ of 1000 ng/mL | SAC |
| 4.7 | PK2 | Table 3.12<br>Study 201037 | Summary of Statistical Analysis of Log-Transformed Danirixin Pharmacokinetic Parameters Sensitivity Analysis: Dry Blood Spot vs Wet Whole Blood Samples - Bland Altman Analysis | excluding dry blood spot<br>concentrations above the assay<br>HLOQ of 1000 ng/mL | SAC |
| 4.8 | PK2 | Table 3.11<br>Study 201037 | Summary of Statistical Analysis of Log-Transformed Danirixin Pharmacokinetic Parameters Sensitivity Analysis: Dry Blood Spot vs Wet Whole Blood Samples | excluding dry blood spot<br>concentrations above the assay<br>HLOQ of 1000 ng/mL | SAC |

## 14.11.10. Pharmacokinetic Figures

| SAC<br>No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4.1 | PK | PKCF1p | Individual Whole Blood Danirixin Concentration-Time Plots by Subject (Linear and Semi-log) (Dry Blood Spot) | X-axis displays actual relative time Include line for LLQ along with footnote defining LLQ value Include values below LLQ Overlay Visit 3, 6, 7 and 10. | SAC |
| 4.2 | PK | PKCF6 | Individual Whole Blood Danirixin Concentration-Time Plots by Day (Linear and Semi-log) (Dry Blood Spot) | X-axis displays actual relative time Include line for LLQ along with footnote defining LLQ value Include values below LLQ | SAC |

| SAC<br>No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4.3 | PK | PKCF4 | Mean (±SD) Whole Blood Danirixin Concentration-Time Plots (Linear and Semi-log) (Dry Blood Spot) | 1. Include the full SD bars at each time point 2. X-axis displays planned relative time 3. Include line for LLQ along with footnote defining LLQ value 4. Overlay Visit 3, 6, 7 and 10. | SAC |
| 4.4 | PK | PKCF5 | Median (Range) Whole Blood Danirixin Concentration-Time Plots (Linear and Semi-log) (Dry Blood Spot) | 1. Include bars for range at each time point 2. X-axis displays planned relative time 3. Include like for LLQ along with footnote defining LLQ value 4. Overlay Visit 3, 6, 7 and 10. | SAC |
| 4.5 | PK | PK27 | Median (Range) Pre-Dose Whole Blood Danirixin<br>Concentration Versus Day (Linear and Semi-log) (Dry Blood<br>Spot) | <ol> <li>Include bars for range at each time point</li> <li>X-axis displays Visit</li> <li>Include like for LLQ along with footnote defining LLQ value</li> <li>Visit include 3, 6, 7 and 10.</li> </ol> | SAC |
| 4.6 | PK | Figure 11.206<br>Study 200163 | Individual Whole Blood Pharmacokinetic Parameters (+Geometric Mean and 95% CI) versus Demographics | Demographics: Age, Weight,<br>Gender.<br>By day. | SAC |
| 4.7 | PK | | Scatter Plot of Whole Blood Danirixin Concentration-by Day (Dry Blood Spot) | | Post SAC |
| 4.8 | PK2 | Figure 3.10<br>Study 201037 | Individual Subject Danirixin Blood Concentration-Time Plot (Linear and Semi-Log) by Subject Dry Blood Spot vs Wet Whole Blood Samples | | SAC |

| SAC<br>No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4.9 | PK2 | Figure 3.8<br>Study 2010137 | Comparative Plot of Individual Subject Danirixin Blood Concentrations Dry Blood Spot vs Wet Whole Blood Samples | | SAC |
| 4.10 | PK2 | Figure 3.9<br>Study 201037 | Bland-Altman Plot of Individual Subject Log-Transformed Danirixin Blood Concentrations Dry Blood Spot vs Wet Whole Blood Samples | | SAC |
| 4.11 | PK2 | Figure 3.10<br>Study 201037 | Individual Subject Danirixin Blood Concentration-Time Plot (Linear and Semi-Log) by Subject Sensitivity Analysis: Dry Blood Spot vs Wet Whole Blood Samples | excluding dry blood spot concentrations above the assay HLOQ of 1000 ng/mL | SAC |
| 4.12 | PK2 | Figure 3.8<br>Study 2010137 | Comparative Plot of Individual Subject Danirixin Blood Concentrations Sensitivity Analysis: Dry Blood Spot vs Wet Whole Blood Samples | excluding dry blood spot<br>concentrations above the assay<br>HLOQ of 1000 ng/mL | SAC |
| 4.13 | PK2 | Figure 3.9<br>Study 201037 | Bland-Altman Plot of Individual Subject Log-Transformed Danirixin Blood Concentrations Sensitivity Analysis: Dry Blood Spot vs Wet Whole Blood Samples | excluding dry blood spot concentrations above the assay HLOQ of 1000 ng/mL | SAC |

## 14.11.11. Pharmacokinetic / Pharmacodynamic Figure

| Pharmacokinetic / Pharmacodynamic: Figures | | | | | |
|---|---|---|---|---|---|
| SAC<br>No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.1 | PK | | Scatter plot of PD endpoint versus Danirixin Concentration (Trough) | CAT Total Score Include Placebo imputed as DNX conc=0ng/mL, include DNX conc=NQ imputed as LLOQ/2, where LLOQ=5ng/mL By Day Different symbol for each treatment | Post SAC |
| 5.2 | PK | | Scatter plot of Safety versus Danirixin Concentration (Trough) | Blood Neutrophil Count and Creactive Protein (CRP) Highlight subjects with an ontreatment event in the 'Infective pneumonia' SMQ. Add footnote 'Note: Pneumonia may have occurred at any time during the study' Include Placebo imputed as DNX conc=0ng/mL, include DNX conc=NQ imputed as LLOQ/2, where LLOQ=5ng/mL By Day Different symbol for each treatment | Post SAC |
| 5.3 | PK | | Quartile plot of Danirixin Concentration versus PD endpoint | CAT Total Score | Post SAC |
| 5.4 | PK | | Quartile plot of Danirixin Concentration versus Safety endpoint | Blood Neutrophil Count and C-<br>reactive Protein (CRP) | Post SAC |

#### 14.11.12. Biomarker Tables

| Bioma | Biomarker: Tables | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Bioma | rkers | | | | | |
| 6.1 | 6.1 | mITT | LB1 | Summary of C-reactive Protein (CRP) Changes from Baseline | ICH E3 | StInt, SAC |
| 6.2 | 6.2 | mITT | LB1 | Summary of Fibrinogen Changes from Baseline | ICH E3 | StInt, SAC |
| | 6.3 | mITT | | Summary of C-reactive Protein (CRP) for Subjects with Pneumonia | Screening, Baseline, Day 84 and 168 Subjects who have an event in the 'Infective pneumonia' SMQ | Post SAC |
| | 6.4 | mITT | | Summary of Fibrinogen for Subjects with Pneumonia | Screening, Baseline, Day 84 and 168 Subjects who have an event in the 'Infective pneumonia' SMQ | Post SAC |

## 14.11.13. Biomarker Figures

| Bioma | rker: Fig | gures | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Bioma | rkers | | | | | |
| 6.1 | 6.1 | mITT | | Boxplot of C-reactive Protein (CRP) by Time and Treatment | Screening, Baseline, Day 84 and 168 | Stint, SAC |
| 6.2 | 6.2 | mITT | | Boxplot of Fibrinogen by Time and Treatment | Screening, Baseline, Day 84 and 168 | Stint, SAC |
| | 6.2 | mITT | | Boxplot of C-reactive Protein (CRP) over Time for Subjects with Pneumonia | Screening, Baseline, Day 84 and 168 Subjects who have an event in the 'Infective pneumonia' SMQ | Post SAC |
| | 6.4 | mITT | | Boxplot of Fibrinogen over Time for Subjects with Pneumonia | Screening, Baseline, Day 84<br>and 168<br>Subjects who have an event in<br>the 'Infective pneumonia' SMQ | Post SAC |

## 14.11.14. ICH Listings

| ICH: Li | stings | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposit | ion | | | | |
| | 1 | ALLSUB | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| | 2 | mITT | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| | 3 | mITT | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| | 4 | mITT | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| | 5 | mITT | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviation | ons | • | | | 1 |
| | 6 | mITT | DV2 | Listing of Important Protocol Deviations | ICH E3 Listing also includes analysis population exclusions. | SAC |
| | 7 | ALLSUB | IE3 | Listing of Screen Failure Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| | 8 | mITT | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |

| ICH: Li | istings | | | | | |
|---|---|---|---|---|---|---|
| Stint<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | ations Ana | lysed | | | | |
| | 9 | mITT | SP3 | Listing of Subjects Excluded from Any Population | ICH E3 ITT (Strategic interim only), mITT, PP, Symptomatic (Strategic interim only), PK and PK2 population | SAC |
| Demog | graphic and | d Baseline Chara | cteristics | | | |
| | 10 | mITT | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| | 11 | miTT | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | nd Concor | mitant Medication | ns | | | |
| | 12 | mITT | CP_CM3 | Listing of Non-COPD Concomitant Medications | IDSL | SAC |
| | 13 | mITT | CP_CM3 | Listing of COPD Concomitant Medications | | SAC |
| Expos | ure and Tr | eatment Complia | nce | | • | |
| | 14 | mITT | EX3 | Listing of Exposure Data | ICH E3 | SAC |
| EXAC1 | Scores | | | | | |
| | 15 | mITT | | Listing of E-RS: COPD Daily Scores | Total and subscale scores | SAC |
| Advers | se Events | | | | | |
| 1 | 16 | mITT | AE8 | Listing of All Adverse Events | ICH E3 | StInt, SAC |
| | 17 | mITT | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| | 18 | mITT | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |

| ICH: Li | istings | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Seriou | s and Oth | er Significant Ad | verse Events | | | |
| | 19 | mITT | AE8 /<br>AE8CPa | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| | 20 | mITT | AE8 /<br>AE8CPa | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| | 21 | mITT | AE14 | Listing of Reasons for Considering as a Serious Adverse<br>Event | ICH E3 | SAC |
| | 22 | mITT | AE8 / AECP8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| | 23 | mITT | AE8 / AECP8 | Listing of Drug-Related Adverse Events | ICH E3 | SAC |
| | 24 | mITT | AE8 / AECP8 | Listing of Adverse Events of Special Interest | ICH E3 | SAC |
| Hepato | biliary (Li | ver) | | | | |
| | 25 | mITT | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | IDSL | SAC |
| | 26 | mITT | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | IDSL | SAC |
| All Lab | oratory | | | | | |
| | 27 | mITT | LB5 | Listing of Chemistry Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| | 28 | mITT | LB5 | Listing of Haematology Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| | 29 | mITT | LB5 | Listing of Chemistry Values of Potential Clinical Importance | | SAC |

| ICH: Li | stings | | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | 30 | mITT | LB5 | Listing of Haematology Values of Potential Clinical Importance | | SAC |
| | 31 | mITT | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| ECG | | | | | | |
| | 32 | mITT | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC |
| | 33 | mITT | EG3 | Listing of ECG Values of Potential Clinical Importance | | SAC |
| | 34 | mITT | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | | SAC |
| | 35 | mITT | EG5 | Listing of Abnormal ECG Findings | | SAC |
| Vital Si | Vital Signs | | | | | |
| | 36 | mITT | VS4 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |

## 14.11.15. Non-ICH Listings

| Non-IC | H: Listings | 3 | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Dispositi | on | | | | |
| | 37. | ALLSUB | ES9 | Listing of Subjects Who Were Rescreened | Include Inclusion/ Exclusion/<br>Randomization Criteria<br>Deviations | SAC |
| | 38. | ALLSUB | | Listing of Study Treatment Misallocations | | SAC |
| Demog | raphic and | d Baseline Chara | cteristics | | | |
| | 39. | mITT | | Listing of Smoking History and Smoking Status | | SAC |
| | 40. | mITT | | Listing of COPD History and Exacerbation History | | SAC |
| | 41. | mITT | | Listing of Screening Spirometry Measures and GOLD Stages at Screening | Include % predicted category (=50%) | SAC |
| | 42. | mITT | | Listing of Baseline Symptomatic Characteristics | Contents as for table | SAC |
| Past ar | nd Current | <b>Medical History</b> | | | | |
| | 43. | mITT | | Listing of Medical Conditions | | SAC |
| | 44. | mITT | | Listing of Family History of Cardiovascular Risk Factors | | SAC |
| | 45. | mITT | | Listing of Percent Oxygen in Blood | | SAC |
| Treatm | ent Comp | liance | | | • | |
| | 46. | mITT | | Listing of Treatment Compliance | | SAC |

| Non-IC | H: Listings | 3 | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| E-RS: ( | COPD | | | | | |
| | 47. | mITT | | Listing of E-RS: COPD Baseline and Monthly Mean Scores | Include baseline and baseline category (=10) Total and subscale scores Include change from baseline and season | SAC |
| Exacer | bations | | | | | |
| | 48. | mITT | | Listing of HCRU Exacerbation Data | | SAC |
| EXACT | Events | | | | | |
| | 49. | mITT | | Listing of EXACT Event Data | | SAC |
| SGRQ | | | | | | |
| | 50. | mITT | | Listing of SGRQ Scores | Total and domain scores Baseline, absolute and change from baseline | SAC |
| CAT | | | | | | |
| | 51. | mITT | | Listing of CAT Scores | Total score Baseline, absolute and change from baseline and season | SAC |
| Rescue | Use | | | | • | |
| | 52. | mITT | | Listing of Derived Rescue Use from Diary | Monthly means Absolute, baseline and change from baseline | SAC |

| Non-IC | H: Listings | 3 | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | 53. | mITT | | Listing of Derived Rescue Use from Sensor | Monthly means Baseline, absolute and change from baseline | SAC |
| Physic | al Activity | | | | | |
| | 54. | mITT | | Listing of C-PPAC Questionnaire Responses | | SAC |
| | 55. | mITT | | Listing of Activity Monitor Data | | SAC |
| | 56. | mITT | | Listing of PROactive Scores | Total and domain scores Baseline, absolute and change from baseline | SAC |
| Subjec | t Global A | ssessments | | | | |
| | 57. | mITT | | Listing of Subject Global Assessments | | SAC |
| Bioma | rkers | | | | | |
| | 58. | mITT | | Listing of Biomarkers | | SAC |
| ECG | | | | | | |
| 2. | 59. | mITT | | Listing of Subjects with Maximum Post-Baseline QTcF increasing to over 500 msec or by 60 msec from Baseline | | StInt, SAC |
| PK | | | | | | |
| | 60. | PK | PKCL1P | Listing of Danirixin Blood Concentration-Time Data – Dry Blood Spot Samples | | SAC |
| | 61. | PK | PKPL1P | Listing of Danirixin Blood Pharmacokinetic Parameter – Dry Blood Spot Samples | | SAC |
| | 62. | PK2 | PKCL1P | Listing of Danirixin Blood Concentration-Time Data – Wet Whole Blood Samples | | SAC |

| Non-IC | H: Listing | S | | | | |
|---|---|---|---|---|---|---|
| StInt<br>No. | SAC<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | 63. | PK2 | PKPL1P | Listing of Danirixin Blood Pharmacokinetic Parameter – Wet Whole Blood Samples | | SAC |
| | 64. | PK2 | Listing 40<br>Study<br>201037 | Supportive SAS Output from Statistical Analysis of Log-<br>Transformed Danirixin Blood Pharmacokinetic<br>Concentration Data - Bland Altman Analysis | | SAC |
| | 65. | PK2 | Listing 42<br>Study<br>2101037 | Supportive SAS Output from Statistical Analysis of Log-<br>Transformed Danirixin Pharmacokinetic Parameters -<br>Bland Altman Analysis | | SAC |
| | 66. | PK2 | Listing 41<br>Study<br>201037 | Supportive SAS Output from Statistical Analysis of Log-<br>Transformed Danirixin Pharmacokinetic Parameters | | SAC |
| | 67. | PK2 | Listing 40<br>Study<br>201037 | Supportive SAS Output from Statistical Analysis of Log-<br>Transformed Sensitivity Analysis: Danirixin Blood<br>Pharmacokinetic Concentration Data - Bland Altman<br>Analysis | excluding dry blood spot<br>concentrations above the assay<br>HLOQ of 1000 ng/mL | SAC |
| | 68. | PK2 | Listing 42<br>Study<br>2101037 | Supportive SAS Output from Statistical Analysis of Log-<br>Transformed Sensitivity Analysis: Danirixin<br>Pharmacokinetic Parameters - Bland Altman Analysis | excluding dry blood spot<br>concentrations above the assay<br>HLOQ of 1000 ng/mL | SAC |
| | 69. | PK2 | Listing 41<br>Study<br>201037 | Supportive SAS Output from Statistical Analysis of Log-<br>Transformed Sensitivity Analysis: Danirixin<br>Pharmacokinetic Parameters | excluding dry blood spot<br>concentrations above the assay<br>HLOQ of 1000 ng/mL | SAC |

## 14.12. Appendix 12: Example Mock Shells for Data Displays

Mock shells will be created in a separate document.